# STATISTICAL ANALYSIS PLAN

Final Version 1.1, dated 28-Jan 2020

A Phase IV Interventional Safety Study of ELIGARD® in Prostate Cancer Patients in Asia (ELIGANT)

ISN: 7015-MA-3072

NCT03035032

Astellas Pharma Singapore Pte Ltd

This confidential document is the property of the sponsor. No unpublished information contained in this document may be disclosed without prior written approval of the sponsor.

# **Table of Contents**

| I. | LIS | T OF ABBREVIATIONS AND KEY TERMS | 5 |
|---|---|---|---|
| 1 | INTRODUCTION····· | | |
| 2 | FLOW CHART AND VISIT SCHEDULE | | |
| 3 | STUDY OBJECTIVE(S) AND DESIGN | | |
| | 3.1 | Study Objective(s) | 10 |
| | 3.1.1 | Primary Objective: | 10 |
| | 3.1.2 | Secondary Objectives: | 10 |
| | 3.2 | Study Design | 10 |
| | 3.3 | Randomization | 10 |
| 4 | СН | ANGES TO ANALYSIS FROM PROTOCOL | 11 |
| 5 | SAI | MPLE SIZE ····· | 11 |
| 6 | AN | ALYSIS SETS ····· | 11 |
| | 6.1 | All Subjects Enrolled Set (ENR) | 11 |
| | 6.2 | Full Analysis Set (FAS) | 11 |
| | 6.3 | Per Protocol Set (PPS)···· | 11 |
| | 6.3.1 | Reasons for Exclusion From PPS | 12 |
| | 6.4 | Safety Analysis Set (SAF) | 12 |
| | 6.5 | Pharmacokinetics Analysis Set (PKAS) | 12 |
| | 6.6 | Pharmacodynamic Analysis Set (PDAS)····· | 12 |
| 7 | AN | ALYSIS VARIABLES | 12 |
| | 7.1 | Efficacy Endpoints | 12 |
| | 7.1.1 | Primary Efficacy Endpoint(s) | 12 |
| | 7.1.2 | Secondary Efficacy Endpoints | 13 |
| | 7.1.3 | Exploratory Efficacy Endpoints · | 13 |
| | 7.1.4 | Other Efficacy Variables · | 13 |
| | 7.2 | Safety Variables · | 13 |
| | 7.3 | Pharmacokinetic Variables | 14 |
| | 7.4 | Pharmacodynamic Variables · | 14 |
| | 7.5 | Other Variables | 14 |
| 8 | STA | ATISTICAL METHODOLOGY | 15 |
| | 8.1 | General Considerations | 15 |

| | 8.2 | Study Population | 16 |
|---|---|---|---|
| | 8.2.1 | Disposition of Subjects | 16 |
| | 8.2.2 | Protocol Deviations | 16 |
| | 8.2.3 | Demographic and Other Baseline Characteristics · | 16 |
| | 8.2.4 | Previous and Concomitant Medications · | 17 |
| | 8.3 | Study Drugs ···· | 18 |
| | 8.3.1 | Exposure | 18 |
| | 8.3.2 | Treatment Compliance | 18 |
| | 8.4 | Analysis of Efficacy | 18 |
| | 8.4.1 | Analysis of Primary Endpoint(s) | 18 |
| | 8.4.2 | Analysis of Secondary Endpoints · | 18 |
| | 8.4.3 | Analysis of Exploratory Endpoints | 20 |
| | 8.4.4 | Analysis of Other Variables · | 20 |
| | 8.5 | Analysis of Safety · | 20 |
| | 8.5.1 | Adverse Events | 20 |
| | 8.5.2 | Clinical Laboratory Evaluation · | 22 |
| | 8.5.3 | Vital Signs····· | 22 |
| | 8.5.4 | ECOG Performance Status · | 23 |
| | 8.5.5 | Pregnancies | 23 |
| | 8.5.6 | Other Safety-Related Observations | 23 |
| | 8.6 | Analysis of PK···· | 23 |
| | 8.7 | Analysis of PD | 23 |
| | 8.8 | Subgroups of Interest | 23 |
| | 8.9 | Other Analyses · | 23 |
| | 8.10 | Interim Analysis (and Early Discontinuation of the Clinical Study) · | 23 |
| | 8.11 | Handling of Missing Data, Outliers, Visit Windows, and Other Information $\cdots$ | 23 |
| | 8.11. | l Missing Data · | 23 |
| | 8.11.2 | 2 Outliers ····· | 24 |
| | 8.11.3 | 3 Visit Windows · | 24 |
| | 8.11.4 | 4 Multicenter | 24 |
| | 8.11. | Retests, Unscheduled Visits and Early Termination Data | 24 |
| 9 | DO | CUMENT REVISION HISTORY | 25 |
| 10 | RE | FERENCES ····· | 25 |
| 11 | API | PENDICES | 26 |

| 11.1 | Appendix 1: Key Contributors and Approvers26 |
|---|---|
| 11.2 | Appendix 2: Programming Conventions for Outputs · · · · · 28 |
| 11.3 | Appendix 3: Algorithm for Treatment Emergence of Adverse Events · · · · · · 29 |
| 11.4 | Appendix 4: Algorithm for Prior / Concomitant Medications:30 |
| 11.5 | Appendix 5: EQ-5D-5L Value Sets · · · · 31 |
| 11.6 | Appendix 6: Lab Reference Ranges96 |

# I. LIST OF ABBREVIATIONS AND KEY TERMS

# List of Abbreviations

| Abbreviations | Description of abbreviations |
|---|---|
| AE | Adverse Event |
| ВМІ | Body Mass Index |
| CI | Confidence Intervals |
| CRF | Case Report Form |
| CS | Classification Specifications |
| CSR | Clinical Study Report |
| DBP | Diastolic Blood Pressure |
| DMC | Data Monitoring Committee |
| FAS | Full Analysis Set |
| GD | Global Development |
| H | High |
| ICH | International Conference on Harmonization |
| L | Low |
| LLN | Lower Limit of Normal |
| LOCF | Last Observation Carried Forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| N | Normal |
| PD | Pharmacodynamic |
| PD | Pharmacodynamic Protocol Deviation 1-x Pharmacodynamic Analysis Set |
| PD<br>PD1-x | Pharmacodynamic Protocol Deviation 1-x Pharmacodynamic Analysis Set Pharmacokinetic |
| PD<br>PD1-x<br>PDAS | Pharmacodynamic Protocol Deviation 1-x Pharmacodynamic Analysis Set |
| PD PD1-x PDAS PK PKAS PPS | Pharmacodynamic Protocol Deviation 1-x Pharmacodynamic Analysis Set Pharmacokinetic Pharmacokinetics Analysis Set Per-Protocol Analysis Set |
| PD PD1-x PDAS PK PKAS | Pharmacodynamic Protocol Deviation 1-x Pharmacodynamic Analysis Set Pharmacokinetic Pharmacokinetics Analysis Set |
| PD PD1-x PDAS PK PKAS PPS | Pharmacodynamic Protocol Deviation 1-x Pharmacodynamic Analysis Set Pharmacokinetic Pharmacokinetics Analysis Set Per-Protocol Analysis Set |
| PD PD1-x PDAS PK PKAS PFS PT SAF SAP | Pharmacodynamic Protocol Deviation 1-x Pharmacodynamic Analysis Set Pharmacokinetic Pharmacokinetics Analysis Set Per-Protocol Analysis Set Preferred Term Safety Analysis Set Statistical Analysis Plan |
| PD PD1-x PDAS PK PKAS PFS PT SAF SAP SAS | Pharmacodynamic Protocol Deviation 1-x Pharmacodynamic Analysis Set Pharmacokinetic Pharmacokinetics Analysis Set Per-Protocol Analysis Set Preferred Term Safety Analysis Set Statistical Analysis Plan Statistical Analysis Software |
| PD PD1-x PDAS PK PKAS PFS PT SAF SAP SAS SBP | Pharmacodynamic Protocol Deviation 1-x Pharmacodynamic Analysis Set Pharmacokinetic Pharmacokinetics Analysis Set Per-Protocol Analysis Set Preferred Term Safety Analysis Set Statistical Analysis Plan Statistical Analysis Software Systolic Blood Pressure |
| PD PD1-x PDAS PK PKAS PKAS PPS PT SAF SAF SAP SAS | Pharmacodynamic Protocol Deviation 1-x Pharmacodynamic Analysis Set Pharmacokinetic Pharmacokinetics Analysis Set Per-Protocol Analysis Set Perferred Term Safety Analysis Set Statistical Analysis Plan Statistical Analysis Software System Organ Class |
| PD PD1-x PDAS PK PKAS PKAS PPS PT SAF SAP SAS SBP SOC TEAE | Pharmacodynamic Protocol Deviation 1-x Pharmacodynamic Analysis Set Pharmacokinetic Pharmacokinetics Analysis Set Per-Protocol Analysis Set Preferred Term Safety Analysis Set Statistical Analysis Plan Statistical Analysis Software System Organ Class Treatment Emergent Adverse Event |
| PD PD1-x PDAS PK PKAS PKAS PPS PT SAF SAF SAP SAS | Pharmacodynamic Protocol Deviation 1-x Pharmacodynamic Analysis Set Pharmacokinetic Pharmacokinetics Analysis Set Per-Protocol Analysis Set Preferred Term Safety Analysis Set Statistical Analysis Plan Statistical Analysis Software Systolic Blood Pressure System Organ Class Treatment Emergent Adverse Event Tables, Listings and Figures |
| PD PD1-x PDAS PK PKAS PKAS PPS PT SAF SAP SAS SBP SOC TEAE | Pharmacodynamic Protocol Deviation 1-x Pharmacodynamic Analysis Set Pharmacokinetic Pharmacokinetics Analysis Set Per-Protocol Analysis Set Preferred Term Safety Analysis Set Statistical Analysis Plan Statistical Analysis Software System Organ Class Treatment Emergent Adverse Event |

# List of Key Terms

| Dist of the free free free free free free free fr | |
|---|---|
| Terms | Definition of terms |
| Adverse Event (AE) | An adverse event is as any untoward medical occurrence in a patient administered a study drug and which does not necessarily have a causal relationship with this treatment (see also Eligard-related AE). |
| Baseline | <ol> <li>Observed values/findings which are regarded as starting points for<br/>comparison.</li> </ol> |
| | 2. Time when 'Baseline' is observed. |

| Case Report Form<br>(CRF) | A printed, optical, or electronic document designed to record all of the protocol required information to be reported to the sponsor for each trial patient. |
|---|---|
| Castrate Resistant<br>Prostate Cancer (CRPC) | The European Association of Urology (EAU) Prostate Cancer Guidelines 2016 defines CRPC as: |
| | Castrate serum testosterone < 50ng/dL or 1.7 nmol/L plus either; |
| | Biochemical progression: 3 consecutive rises in prostate specific antigen (PSA) at least 1 week apart resulting in two 50% increases over the nadir, and a PSA > 2 ng/mL or |
| | Radiological progression: the appearance of two or more new bone lesions on bone scan or enlargement of a soft tissue lesion using RECIST (Response Evaluation Criteria in Solid Tumors). |
| | Symptomatic progression alone must be questioned and is not sufficient to diagnose CRPC. |
| Causality Assessment | An evaluation performed by a medical professional concerning the likelihood that a therapy or product caused or contributed to an AE. A positive causality assessment made by either reporter and/or company makes an AE into an ADR. |
| Clinical Study | Any investigation in relation to humans intended: |
| | a) to discover or verify the clinical, pharmacological or other pharmacodynamic effects of 1 or more medicinal products; |
| | b) to identify any adverse reactions to 1 or more medicinal products; or |
| | c) to study the absorption, distribution, metabolism and excretion of 1 or more medicinal products; with the objective of ascertaining their safety or efficacy. |
| Confidence Interval (CI) | A measure of the precision of an estimated value. The interval represents the range of values, consistent with the data that is believed to encompass the "true" value with high probability (usually 95%) upon repeated sampling according to frequentist theory. The confidence interval (CI) is expressed in the same units as the estimate. Wider intervals indicate lower precision; narrow intervals, greater precision. |
| Confidentiality | Prevention of disclosure to other than authorized individuals of proprietary information or of a patient's identity. |
| Consent Form | Document used during the informed consent process that is the basis for explaining to potential patients the risks and potential benefits of a study and the rights and responsibilities of the parties involved. The informed consent document provides a summary of a clinical trial (including its purpose, the treatment procedures and schedule, potential risks and benefits, alternatives to participation, etc.) and explains an individual's rights as a patient. It is designed to begin the informed consent process, which consists of conversations between the patient and the research team. |

| | If the individual then decides to enter the trial, s/he gives her/his official |
|---|---|
| | consent by signing the document. Synonym: informed consent form (ICF) |
| Contract Research<br>Organization (CRO) | A person or an organization (commercial, academic, or other) contracted<br>by the sponsor to perform 1 or more of a sponsor's trial-related duties<br>and functions. |
| Data Monitoring | Process by which data are examined for completeness, consistency, and accuracy. |
| Demographic data | Characteristics of patients or study populations, which include such information as age, sex, family history of the disease or condition for which they are being treated, and other characteristics relevant to the study in which they are participating. |
| Discontinuation | The act of concluding participation, prior to completion of all protocol-<br>required elements, in a study by an enrolled patient. |
| Effectiveness | The capability of an intervention in producing a desired result under circumstances that more closely approach real-world practice, with more heterogeneous populations, less-standardized treatment protocols, and delivery in routine clinical settings. |
| Electronic Case Report<br>Form (eCRF) | Auditable electronic record designed to capture information required by<br>the clinical trial protocol to be reported to the sponsor on each trial<br>patient. |
| Eligard-related Adverse<br>Event | An adverse event in a patient administered Eligard where a causal relationship is at least a reasonable possibility (drug event with either a possible or probable causal relationship), as determined by the opinion of the investigator. |
| | Adverse events listed in the local label should be used by the investigator as reference safety information to understand whether an adverse event is expected with the use of Eligard. This understanding should inform causality assessments by the investigator. |
| Ethnic Asian | Any of the following races - Chinese, Filipino, Indonesian, Malay, Thai, Vietnamese, Indian, Japanese or Korean. |
| Final Visit | The final visit will be the same as the last follow-up visit for each patient. It will occur at the 18 <sup>th</sup> month after enrollment into the study, provided that none of discontinuation criteria (see Section Error! Reference source n ot found, in protocol) are met. |
| Protocol | A document that describes the objective(s), design, methodology, statistical considerations, and organization of a trial. The protocol usually also gives the background and rationale for the trial, but these could be provided in other protocol referenced documents. Throughout the International Conference on Harmonisation – Good Clinical Practice (ICH GCP) Guideline the term protocol refers to protocol and protocol amendments. |
| Quality of Life (QoL) | A broad ranging concept that incorporates an individual's physical health, psychological state, level of independence, social relationships, |

| | personal beliefs, and their relationships to salient features of the environment. |
|---|---|
| | Note: Quality of Life is one way to measure the benefits or negative impacts of an "improvement" measured in terms of a physiological or psychological symptom. QoL research seeks to quantify what an intervention means to a patient's sense that their life has changed. |
| Safety | Relative freedom from harm. In clinical trials, this refers to an absence of harmful side effects resulting from use of the product and may be assessed by laboratory testing of biological samples, special tests and procedures, psychiatric evaluation, and/or physical examination of patients. |
| Sample Size | A subset of a larger population, selected for investigation to draw conclusions or make estimates about the larger population. |
| Serious Adverse Event<br>(SAE) | An SAE is any experience that suggests a significant hazard, contraindication, side effect or precaution. An SAE must fulfill at least 1 of the following criteria at any dose level: results in death; is life threatening, results in persistent or significant disability/ incapacity or substantial disruption of the ability to conduct normal life functions; results in congenital anomaly, or birth defect; requires inpatient hospitalization or leads to prolongation of hospitalization; or a medically important event. |
| Serious Eligard-related<br>Adverse Event | An Eligard-related AE which results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/ incapacity, is a congenital anomaly/ birth defect, or results in other medically important events. |
| | Adverse events listed in the local label should be used by the investigator as reference safety information to understand whether a serious adverse event is expected with the use of Eligard. This understanding should inform causality assessments by the investigator |
| Statistical Analysis Plan<br>(SAP) | A document that contains a more technical and detailed elaboration of<br>the principal features of the analysis described in the protocol, and<br>includes detailed procedures for executing the statistical analysis of the<br>primary and secondary variables and other data. |
| Statistical Method | The particular mathematical tests and techniques that are to be used to evaluate the clinical data in a trial. |
| Study Period | Period of time from the initiation date to the completion date of the study. |
| Study Population | Defined by protocol inclusion/exclusion criteria. |
| Visit | A clinical encounter that encompasses planned and unplanned trial interventions, procedures, and assessments that may be performed on a patient. A visit has a start and an end, each described with a rule. |
| Withdrawal | The act of discontinuing participation in a clinical study. See also discontinuation. |

# 1 INTRODUCTION

This Statistical Analysis Plan (SAP) contains a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and includes detailed procedures for executing the statistical analysis of the primary and secondary endpoints and other data.

# 2 FLOW CHART AND VISIT SCHEDULE

#### Flow Chart

Decision has been made by clinician to initiate treatment of the patient with LHRH agonist (3 month formulation) before patient is consented for entering this study. Anti-androgen for at least 3 days to 4 weeks prior to the first ELIGARD® injection and continuing for the first two to three weeks of treatment should be considered.

Pre-screening/Consent / Baseline visit Mandatory collection of testosterone & PSA; AE and SAE assessment; Other data collection at time of administration of ELIGARD® Treatment, visit window +/- 14 days

Follow-up visit at 18 months: AE, PSA, Testosterone, and QoL.



### Legend:



Administration of ELIGARD®, details are listed in #.



Data Collection Points

#### Notes:

#: ELIGARD® will be administered at baseline, 3 months, 6 months, 9 months, 12 months, and 15 months. PSA and Testosterone levels to be measured in all the visits. Visit window is +/-14 days. QoL to be measured at baseline, 6 months, 12 months and 18 months. Any other assessments including imaging tests are not mandatory and will be performed according to routine standard of care and physician's discretion. One month = 30 days.

# Schedule of Assessment

The table of scheduled assessments can be found in Section V of protocol.

# 3 STUDY OBJECTIVE(S) AND DESIGN

# 3.1 Study Objective(s)

The objectives of this Phase IV, prospective, interventional study are to evaluate the safety, efficacy, and QoL of ELIGARD® in hormone-dependent prostate cancer patients in Asia.

# 3.1.1 Primary Objective:

To establish the safety profile of ELIGARD® in ethnic Asian prostate cancer patients.

#### 3.1.2 Secondary Objectives:

- To describe the efficacy of ELIGARD® 22.5 mg (3-monthly formulation) in controlling PSA and testosterone levels
- 2) To assess HRQoL through QoL questionnaires EORTC QLQ-PR25 and EQ5D-5L

# 3.2 Study Design

This is a multicenter, prospective, single-arm, interventional study to assess the safety, efficacy, and QoL of ELIGARD® 22.5 mg (3-monthly formulation) in male patients with prostate adenocarcinoma who fulfill the eligibility criteria in Asia. The sample size planned for this study is approximately 107 enrolled prostate cancer patients. The inclusion/exclusion criteria are listed in Section 3.1 and 3.2 in the study protocol. This study will be conducted in approximately 20 centers in 8 countries (Hong Kong, Indonesia, Malaysia, Philippines, Singapore, Taiwan, Thailand and Vietnam).

The enrollment period will be up to 12 months. Patients will be prescreened to confirm access to Androgen Deprivation Therapy (ADT) prior to informed consent. Following written informed consent by the patient and confirmation of eligibility, patients will be treated for 1.5 years (18 months), with ELIGARD® 22.5 mg being administered at baseline, 3rd month, 6th month, 9th month, 12th month and 15th month. AE and SAE collection will start at baseline until the follow-up visit at 18 months (see protocol Section Error! Reference source not f ound. for AE collection and SAE reporting). QoL will be measured at baseline, 6th month, 12th month and 18th month. The PSA and testosterone levels will be assessed at all scheduled visits and during the follow-up visit. Patients will be followed up at 18th month in the physician's office. The time window for each visit following baseline is +/- 14 days.

A minimum of 1 interim analysis will be conducted when 50 patients complete 1 year of follow-up.

### 3.3 Randomization

Not Applicable.

#### 4 CHANGES TO ANALYSIS FROM PROTOCOL

- Patients who are less than 80% compliant with the dosage regimen for any two visit
  periods during the study should be withdrawn. The two visits are not necessarily
  consecutive.
- Added Protocol Deviation rule 5 of windowing convention.
- Added analyses of PSA reduction in categorical summarization.
- Included Kaplan-Meier curve for deterioration of quality of life variables (EQ5D02-EQ VAS score, EQ-5D-5L score and QLQ-PR25 score)
- KM estimates for incidence rate at each scheduled time points will not be provided, as incidence rate is not a time to event variable.

#### 5 SAMPLE SIZE

This study targets to enroll approximately 107 prostate cancer patients meeting all inclusion criteria and none of the exclusion criteria. The sample size calculation is based on assumptions that percentage of ELIGARD®-related AEs will be 50%, a drop-out rate of 10%, and a Wald 95% CI of width 20%, based on a finite population correction, with factor N =10,000.

#### 6 ANALYSIS SETS

In accordance with International Conference on Harmonization (ICH) recommendations in guidelines E3 and E9, the following analysis sets will be used for the analyses.

# 6.1 All Subjects Enrolled Set (ENR)

The all subjects enrolled (ENR) set will contain all subjects who provide informed consent for this study. Subject disposition will be presented using ENR.

# 6.2 Full Analysis Set (FAS)

The full analysis set (FAS) will consist of all patients who are enrolled and receive at least one dose of study drug and have at least one post baseline measurement of PSA and testosterone level.

Specifically, the following will lead to a subject's exclusion from the FAS:

- No study drug taken
- No post baseline measurement of PSA and testosterone.

The FAS will be used for summaries and primary analyses of efficacy data.

# 6.3 Per Protocol Set (PPS)

The Per-Protocol Set (PPS) includes all subjects of the FAS who do not meet criteria for exclusion from PPS listed in section 6.3.1 of this SAP.

The PPS will be used for secondary analyses of efficacy data. Also, selected demographic and baseline characteristics will be summarized for the PPS.

#### 6.3.1 Reasons for Exclusion From PPS

The following criteria are to capture relevant non-adherence to the protocol and the following reasons may lead to subject's exclusion from PPS:

- Entered into the study even though they did not satisfy entry criteria
- Developed withdrawal criteria during the study and was not withdrawn (Patients who
  discontinued the study for efficacy-related reasons, such as insufficient therapeutic effect,
  will be included in the PPS.)
- Full dose was not administered or drug reconstitution was not performed as prescribed
- Patients with treatment compliance <80%</li>
- Patients who used prohibited concomitant medications as defined in the protocol sections 5.1.6 and 12.2.

# 6.4 Safety Analysis Set (SAF)

The Safety Analysis Set (SAF) consists of all subjects who received at least one ELIGARD® injection and any follow-up safety information is available.

The SAF will be used for statistical summaries of safety data. Demographic and baseline characteristics and all safety and tolerability related variables will be summarized using SAF as well.

# 6.5 Pharmacokinetics Analysis Set (PKAS)

Not Applicable.

# 6.6 Pharmacodynamic Analysis Set (PDAS)

Not Applicable.

#### 7 ANALYSIS VARIABLES

The primary endpoint for this study is ELIGARD®-related AEs throughout the entire observation period, as determined by the opinion of the investigator.

Secondary endpoints include:

- Efficacy outcomes of clinical response based on testosterone and PSA levels (Testosterone level and PSA will be assessed for all patients at each scheduled visit, prior to administering ELIGARD<sup>®</sup>, and at the follow-up visit.)
- HRQoL assessment through QoL questionnaires EORTC QLQ-PR25 (prostate cancer disease specific PRO) and EQ5D-5L (generic PRO) measured at 0, 6, 12, and 18 months.

# 7.1 Efficacy Endpoints

#### 7.1.1 Primary Efficacy Endpoint(s)

As the primary analysis of this study is the safety outcomes, primary efficacy variable is not applicable.

# 7.1.2 Secondary Efficacy Endpoints

The following secondary efficacy endpoints, as derived, are:

- Percentage of patients with Testosterone <20 ng/dL, 20-50ng/dL and >50 ng/dL at 1 and 1.5 years
- Time to PSA progression
- PSA percent reduction to reach ≥30%, ≥50 and ≥90%
- Scores and change from baseline for EORTC, QLQ-PR25 and EQ-5D-5L

Relevant derivations are as below:

General

Change from baseline = Test value at visit X – baseline value.

Percentage of patients with Testosterone <20 ng/dL, 20-50ng/dL and >50 ng/dL at 1 and 1.5 years

Percentage = (number of patients with corresponding Testosterone level) / (total number of patients in FAS/PPS for that follow-up time).

Time to PSA progression

Time to PSA progression (months) = ((date of 25% or greater increase and an absolute increase of 2ng/mL) - (date of first administration of ELIGARD® 22.5 mg) + 1)/30.

PSA response percentage = number of patients with PSA response (at each visit)/ total number of patients in FAS/PPS.

PSA percent reduction to reach  $\geq$ 30%,  $\geq$ 50 and  $\geq$ 90%

PSA response percent reduction (%) = ((PSA tested–baseline PSA) / baseline PSA)\*100%.

Scores and change from baseline for EORTC, QLQ-PR25 and EQ-5D-5L

For each respective scale, Raw score (RS) =  $(I1+I2+\cdots+In)/n$ ,

with I<sub>n</sub> being the score for each question and n for total number of questions included.

For functional scale (SAC, SFU), Scale score (S) = (1 - (RS-1)/range) \* 100, for symptom scales (URI, AID, BOW, HTR), S = ((RS-1)/range) \* 100,

with range defined as the difference between the maximum and minimum possible value of RS, which is 3 for QLQ-PR25.

#### 7.1.3 Exploratory Efficacy Endpoints

Not Applicable.

# 7.1.4 Other Efficacy Variables

Not Applicable.

# 7.2 Safety Variables

All outputs for safety outcomes will be based on the Safety Analysis Set. There will be no

statistical comparisons as there is no comparative drug.

Safety will be assessed by evaluation of the following variables:

- Adverse events (AEs), serious adverse events (SAEs), and treatment-emergent adverse
  events (TEAEs; frequency, severity, seriousness, and relationship to study drug)
- Treatments including any intervention (e.g. medication(s), procedure(s), radiography, surgical treatment, visits to Accident & Emergency department and/or ambulatory clinic, hospitalization) to treat AEs and SAEs
- Clinical laboratory variables (hematology, biochemistry including liver enzymes and total bilirubin, and urinalysis)
- Vital signs (systolic and diastolic blood pressure, respiratory rate and pulse rate)

Treatment emergent adverse events (TEAEs) are defined as AEs with onset dates occurring within the treatment periods, i.e., starts on or after the earliest dosing date of any study treatment and prior to the latest dosing date of any treatment. If the patient early terminates, then AEs happen within early terminate date plus 90 days will be still counted as TEAEs, and after that, AEs occurred will not be seen as TEAEs. TEAEs will be captured and determined on "Adverse Events" page of CRF, with "Onset date of adverse event occurred after first dose of study drug" marked "yes".

For this study, an ELIGARD®-related AE is defined as an adverse event in a patient administered ELIGARD® where a causal relationship is at least a reasonable possibility (drug event with either a possible or probable causal relationship), as determined by the investigator.

Incidence of ELIGARD®-related AE(SAE) is defined as the new ELIGARD®-related AE(SAE) cases happen in study population within the specified period of time. Incidence rate is defined as the number of new cases per population at risk in a given time period.

#### 7.3 Pharmacokinetic Variables

Not Applicable.

# 7.4 Pharmacodynamic Variables

Not Applicable.

#### 7.5 Other Variables

# The duration of exposure

Duration of exposure months = (date of last study medication administration – date of first study medication administration + 1) / 30.

Duration of exposure years = (date of last study medication administration – date of first study medication administration + 1) / 365.25.

#### Cumulative dose

Cumulative dose (mg) = number of injections \* 22.5.

Cumulative dose will be calculated in the cases where response to 'drug administered?' and 'reconstituted and mixed as per instructions?' should be 'YES'.

# Study drug compliance

Overall compliance to the dosing schedule will be examined for subjects in the safety population.

Compliance with ELIGARD®—based on the injection given or not—will be calculated as the number of injections taken divided by the prescribed number of injections as a percentage, see calculations below.

Compliance for each patient = ((Number of Injections Given provided study drug reconstituted and mixed as per instructions) / Number of Injections Prescribed) \* 100%;

While considering number of injections given, study drug must be reconstituted and mixed according to the instructions provided. In case study drug administered but not reconstituted and mixed as per instructions provided, study drug will not be counted in numerator.

#### Duration of Prostate Cancer

Duration of Prostate Cancer = (Cutoff date of Data – Baseline Assessment Date of Prostate Cancer History+1)/30.

# Time Since Biopsy

Time Since Biopsy – (Cutoff Date of Data – Date of Biopsy+1)/30.

Date of biopsy will be taken from prostate cancer history form.

#### 8 STATISTICAL METHODOLOGY

#### 8.1 General Considerations

Unless otherwise specified, baseline is defined as the last non-missing measurement taken prior to reference start date (including unscheduled assessments). In the case where the last non-missing measurement and the reference start date coincide, that measurement will be considered pre-baseline, but Adverse Events (AEs) and medications commencing on the reference start date will be considered post-baseline.

For continuous variables, descriptive statistics will include the number of subjects (n), mean, standard deviation, median, minimum and maximum. When needed, the use of other percentiles (e.g. 25% and 75%) will be mentioned in the relevant section. Frequencies and percentages will be displayed for categorical data. If missing option is not included in summaries, percentages by categories will be based on the number of subjects with missing data, i.e. might not add up to 100%.

Summaries based on FAS and PPS (efficacy data), safety analysis and other summaries based on SAF will be presented by planned region, unless specifically stated otherwise.

No statistical tests will be conducted in this study. Confidence intervals will be 95% for analyses unless specified in the description.

All data processing, summarization, and analyses will be performed using SAS® Version 9.4 or higher on Windows. Sample size is calculated using PASS 14 Power Analysis and Sample

Size Software (2015) version 14.0.2 and validated using nQueries v4.0. Specifications for table, figures, and data listing formats can be found in the TLF specifications for this study.

For the definition of regions, please refer to section 8.11.4.

# 8.2 Study Population

#### 8.2.1 Disposition of Subjects

All subjects who provide informed consent will be accounted for in this study. ENR will be applied for screened, screen failure, and analysis sets disposition. Summary table will be provided in total, and by region defined in Section 8.11.4.

The following subject data will be presented:

- Number of subjects with informed consent, received study medication and screen failure;
- Number and percentage of subjects allocated to each analysis sets;
- Number and percentage of subjects completed and discontinued the study, and primary reasons for discontinuation and
- Number and percentage of subjects excluded from each analysis sets for each reason defined in Section 5.

#### 8.2.2 Protocol Deviations

Protocol deviations as defined in Section , in protocol will be summarized for all patients. Visiting window deviation is added as the 5<sup>th</sup> protocol deviation. A data listing will be provided by site and patient.

The protocol deviation criteria will be uniquely identified in the summary table and listing. The unique identifiers will be as follows:

- PD1 Entered into the study even though they did not satisfy entry criteria
- PD2 Developed withdrawal criteria during the study and was not withdrawn
- PD3 Full dose was not administered or drug reconstitution was not performed as prescribed
- PD4 Received excluded concomitant treatment
- PD5 Window deviation.

#### 8.2.3 Demographic and Other Baseline Characteristics

Demographic data and other baseline characteristics will be presented for the SAF and PPS. Descriptive statistics will include number of patients, mean, SD, median, minimum, maximum, 25<sup>th</sup> percentile (Q1) and 75<sup>th</sup> percentile (Q3) for continuous variables, and frequency and percentage for categorical variables. No statistical testing will be carried out for demographic or other baseline characteristics. The following demographic and other baseline characteristics will be reported for this study:

- Age (years) calculated relative to date of consent
- Sex
- Race
- Country of the investigational site

- Highest education level
- Medical history
- Vital Signs
- Weight(kg)
- Height(cm)
- BMI (kg/m<sup>2</sup>)
- ECOG performance status
- Laboratory tests

Surgical and Medical History (diabetes, hypertension and cardiac disorders) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) (Version 20.0 or higher). Numbers and percentages of patients will be presented for each System Organ Class (SOC) and Preferred Term (PT) and will be sorted by incidence rate (high to low) and then alphabetic order. The following variables will be summarized to describe the history/status of the disease being studied:

- Prostate cancer history
- Family history for prostate cancer
- Disease characteristics for prostate cancer
- Most important factors for selection of treatment

Disease characteristics include time since diagnosis, Gleason score at initial diagnosis, Tumor, Nodes, Metastasis (TNM) classification, staging, surgical history, biopsy results, dates and types of anti-neoplastic therapy including radiation therapy prior to study inclusion (including number of cycles, treatment duration, time interval since previous treatments), Eastern Cooperative Oncology Group (ECOG) status, bone lesions, soft tissue disease, visceral disease, and pain (using the Visual Analogue Scale [VAS] 0-10).

#### 8.2.4 Previous and Concomitant Medications

Previous medications are medications which started and stopped prior to the first dose of study medication.

Concomitant medications are medications which:

- Started prior to, on or after the first dose of study medication
- AND ended on or after the date of first dose of study medication or were ongoing at the end of the study.

As with previous medication, concomitant medication will be summarized for each regional group using SAF and coded using World Health Organization (WHO) Drug Dictionary Enhanced Version 01Jun2015 or higher. Prior and concomitant medication data will be captured from "Concomitant Medication" page on eCRF. Subjects taking the same medication multiple times will be counted once per medication and investigational period.

Bicalutamide 50 mg O.D. or a similar anti-androgen is an allowed concomitant medication for flare prevention only. Additional administration of an appropriate anti-androgen should be considered beginning three days prior to ELIGARD® treatment and continuing for the first two

to three weeks of treatment to avoid any flare reaction. Use of bicalutamide or similar antiandrogen beyond 3 weeks after starting ELIGARD® therapy and for reasons other than flare prevention is not allowed.

See Appendix 4 for handling of partial dates for medications, in the case where it is not possible to define a medication as prior, or concomitant treatment, the medication will be classified by the worst case; i.e. concomitant.

# 8.3 Study Drugs

#### 8.3.1 Exposure

Exposure to study medication in months and dose in mg will be presented for the SAF. The dose of each administration is fixed to 22.5mg and can be referenced to "ELIGARD® Use" page from CRF.

The following will be reported:

- Duration of therapy in months, using descriptive statistics
- Number of injections in categorical form and with descriptive statistics
- Cumulative dose with descriptive statistics
- Treatment compliance

The date of first study medication administration will be taken from the eCRF "Date of Visit" form in Baseline folder. The date of last study medication will be taken from the eCRF "End of Treatment" form. In case of missing data, see Appendix 3 for reference to determine the first and last date of study medication. Interruptions and incompliance are not taken into account for duration of exposure.

#### 8.3.2 Treatment Compliance

Overall compliance to study medication will be presented for the SAF. Summary statistics for compliance including mean, SD, median, Q1 and Q3 will be reported. As the study is a fixed-dose injection study, the compliance for each patient through the study is calculated by number of injections divided by total injections administered. Dose injected outside the visit periods will be considered as incompliant. In case dose injected but not reconstituted and mixed as per instructions, it will be considered as incompliant. Patients who are less than 80% compliant with the dosage regimen for any two visit periods (window  $\pm$  14 days) during the study should be withdrawn.

# 8.4 Analysis of Efficacy

#### 8.4.1 Analysis of Primary Endpoint(s)

Not applicable as the primary endpoint of this study is safety outcomes.

#### 8.4.2 Analysis of Secondary Endpoints

The secondary efficacy analyses will be performed for the FAS and PPS will be used to assess the robustness of the results.

#### 8.4.2.1 Testosterone Level

Testosterone levels are captured on "Serum Testosterone Level" page in CRF. Numbers and percentage of patients with following Testosterone level at 1 and 1.5 years will be summarized:

- <20 ng/dL,</p>
- 20-50 ng/dL,
- >50 ng/dL.

#### 8.4.2.2 PSA Progression and Reduction

PSA progression is defined as a 25% or greater increase and an absolute increase of 2 ng/mL, and confirmed by a second value obtained three or more weeks later (captured on "Unscheduled" page in CRF).

Number and percentage of patients to reach following PSA percent reduction will be summarized:

- >30%,
- >50%,
- ≥90%.

Time to PSA progression (months) = (date of 25% or greater increase and an absolute increase of 2ng/mL) - (date of first administration of ELIGARD® 22.5 mg)/30.

If confirmed by a second value obtained later, the date of first value obtained will be used for calculation.

PSA percent reduction (%) = ((PSA tested-baseline PSA) / baseline PSA)\*100%

#### 8.4.2.3 Health-related Quality of Life (HRQoL)

EORTC QLQ-PR25 and EQ-5D-5L (captured on "EORTC QLQ-PR25" and "EQ-5D-5L" page correspondingly in CRF) are used to examine health-related quality of life.

### EQ-5D-5L

Number and frequencies for each summary scale, including mobility, self-care, usual activities, pain/discomfort and anxiety/depression will be presented for EQ-5D-5L. Index scores will be generated using Japan, UK and USA value sets (see Appendix 5 for EQ-5D-5L value sets). Absolute index scores, changes from baseline and Kaplan-Meier curves for score deterioration will be presented.

EQ5D02-EQ VAS Score (also captured on "EQ-5D-5L" page) will be presented separately with absolute index score, change from baseline, Kaplan-Meier curves for score deterioration.

# EORTC QLQ-PR25

The rule of scoring for QLQ-PR25 follows instruction of EORTC QLQ-PR25 Scoring Manual 2.0. Scale scores after linear transformation (in a 0-100 scale) for each dimension, including urinary symptoms, incontinence aid, bowel symptoms, hormonal treatment related symptoms, sexual activities and sexual function will be presented for QLQ-PR25. Absolute scores of dimensions, changes from baseline and Kaplan-Meier curves for score deterioration will be presented.

# 8.4.2.4 Tumor Response

Tumors will be evaluated according to the standard of Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. Tumor responses are collected and will be summarized for each follow-up visits. FAS and PPS will be used for the analysis of tumor response. Best overall response will also be presented for both datasets.

# 8.4.3 Analysis of Exploratory Endpoints

Not Applicable.

# 8.4.4 Analysis of Other Variables

Not Applicable.

# 8.5 Analysis of Safety

All analysis of safety will be presented by region for SAF, unless specified otherwise.

#### 8.5.1 Adverse Events

# 7.5.1.1 Adverse events

An Adverse Event (AE) is defined as any untoward medical occurrence in a patient administered a study drug or has undergone study procedures and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. AEs will be captured on CRF page "Adverse Events", and collected after the first administration of study drug.

Severity is classed using the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Event (CTCAE) guidelines (Version 4.03). The items that are not stipulated in the NCI-CTCAE Version 4.03 will be assessed according to the criteria described in Section 5.6.4 in protocol.

Relationship, as indicated by the Investigator, is classed as "not related", "possible", "probable" (increasing severity of relationship). Detailed criteria for causal relationship are listed in Section 5.6.3 in protocol.

All AEs (including TEAEs, ELIGARD®-related AEs) will be coded using Medical Dictionary for Regulatory Activities (MedDRA) Version 20.0 or higher. It will be used to summarize AEs by SOC and PT.

See Appendix 2 for handling of partial dates for AEs. In the case where it is not possible to define an AE as treatment emergent or not, the AE will be classified by the worst case; i.e. ELIGARD®-related / treatment emergent.

An overview table will include the following details:

- Number of AEs, SAEs, TEAEs, and serious TEAEs,
- Number and percentage of subjects with AEs, SAEs, TEAEs, and serious TEAEs,
- Number of ELIGARD®-related AEs, SAEs,

- Number and percentage of subjects with ELIGARD®-related AEs, SAEs,
- Number of TEAEs leading to drug withdrawal and drug interrupted,
- Number and percentage of subjects with TEAEs leading to drug withdrawal and drug interrupted,
- Number of special adverse events and
- Number of death.

#### 7.5.1.2 Adverse events by SOC and/or PT

The number and percentage of subjects with TEAEs, as classified by SOC and PT will be summarized for each region. Summaries will be provided for:

- TEAEs
- drug related TEAEs,
- TEAEs by relationship to study drug,
- TEAEs and drug related TEAEs by severity,
- Drug related AEs and SAEs after CRPC managing,
- TEAEs and drug related TEAEs leading to treatment discontinuation.
- TEAEs and drug related TEAEs leading to drug interruption and,
- TEAEs and drug related TEAEs leading to death

The number of TEAEs and the number and percentage of subjects with TEAEs, as classified by SOC and PT will also be summarized by severity and by relationship to study drug. In the subject count, if a subject has multiple TEAEs with the same SOC or PT, but with differing severity or relationship, then the subject will be counted only once with the worst severity and highest degree of relationship. In the adverse event count, the adverse events will be presented in each category they were classified to. Drug related TEAEs will be presented in a similar way by severity only.

#### 7.5.1.3 Drug Related Adverse Events

The ELIGARD®-related AEs will be summarized according to their severity, NCI CTCAE Grade, outcome, course of event, seriousness, action taken with ELIGARD® and treatment required to manage the AE for SAF set.

The incidence of ELIGARD®-related AEs and SAEs will be analyzed based on SAF. Twosided 95% symmetric confidence intervals of incidence rates will be calculated based on normal approximation and adjusting for a finite sample size of 10000.

If applicable, estimated median time to first event together with a 95% CI will be prepared. In addition, incidence rates of ELIGARD® -related AEs and SAEs will be summarized at each scheduled visit time-point, together with a 95% CI. AEs that happen on the scheduled visit date will be counted in the visit, and AEs occur after scheduled visit will be counted into next visit.

Time to first occurrence, in months, of ELIGARD® -related AEs and SAEs will be presented graphically using Kaplan-Meier (KM) plots for three regions and all.

# 8.5.2 Clinical Laboratory Evaluation

The baseline visit is the last measurement taken prior to initial study drug administration.

Quantitative clinical laboratory variables, i.e. hematology, biochemistry, and coagulation will be summarized using mean, standard deviation, minimum, maximum, and median for each region at each visit. Additionally, a within-subject change will be calculated as the post-baseline measurement minus the baseline measurement and summarized in the same way. Each laboratory result will be classified as low (L), normal (N), or high (H) at each visit according to the laboratory supplied reference ranges, if applicable. Values including a comparator will be imputed by rounding 0.01 up or down, i.e., <x will be imputed to x-0.01 and >x will be imputed to x+0.01.

The number and percentage of subjects within, below and above reference range will be summarized for each region at each visit and last on-treatment.

Frequency tabulations of qualitative clinical laboratory variables (urinalysis and serology) will be presented for each region at each visit.

Laboratory abnormalities will be evaluated on their clinical significance and decided by investigator. Shift tables of change from baseline to each treatment visit, last on-treatment and worst finding during the treatment period will be presented for each region and all.

# 8.5.3 Vital Signs

The baseline visit is the last measurement taken prior to initial study drug administration. Baseline measurements of systolic and diastolic blood pressure should come from the same measurement and not from different dates.

Vital signs data will be captured on CRF page "Adverse Events" and will be summarized in tables and listings using mean, standard deviation, minimum, maximum, median, Q1 and Q3 by region and visit. The following Vital Signs measurements for both baseline and follow up visits will be reported for this study:

- Systolic Blood Pressure (mmHg)
- Diastolic Blood Pressure (mmHg)
- Respiratory Rate (breaths/min)
- Pulse Rate (bpm)
- Weight (kg)
- Height (m) at baseline only

Additionally, a within-subject change will be calculated per visit as the post-baseline measurement minus the baseline measurement and summarized by region and visit.

Tables for potentially clinically significant vital signs will be presented for SBP, DBP and pulse rate. Summaries will be generated using baseline value and highest value obtained during treatment for each subject for each region.

The following potentially clinically significant criteria are defined for the following parameters:

| Vital Sign Variable | Criteria |
|---------------------|---------------------------------------------|
| SBP | ≥180 mmHg AND ≥20 mmHg change from baseline |
| DBP | ≥105 mmHg AND ≥15 mmHg change from baseline |
| Pulse Rate | ≥120 bpm AND ≥15 bpm change from baseline |

#### 8.5.4 ECOG Performance Status

ECOG performance status data will be captured on CRF page "ECOG Performance Status at Present" and will be summarized by listing number and percentage to relevant analysis set selecting each score scale for each region at each treatment visit and time point, including changes from baseline.

#### 8.5.5 Pregnancies

A detailed listing of all pregnancies will be provided.

## 8.5.6 Other Safety-Related Observations

Not Applicable.

# 8.6 Analysis of PK

Not Applicable.

# 8.7 Analysis of PD

Not Applicable.

#### 8.8 Subgroups of Interest

Not Applicable.

# 8.9 Other Analyses

Not Applicable.

# 8.10 Interim Analysis (and Early Discontinuation of the Clinical Study)

A minimum of one interim analysis will be conducted at 20 months when 50 patients will complete 1 year of treatment after the first patient is enrolled. The 20 months timepoint is determined as 50 patients are expected to be recruited at 8 months after the first patient is enrolled. A full analysis will be conducted for interim analysis and will be using this Statistical Analysis Plan. As there are no statistical hypothesis tests in the planned analysis, the conduct of interim analyses will not have any statistical implications on the final study outcome.

# 8.11 Handling of Missing Data, Outliers, Visit Windows, and Other Information

#### 8.11.1 Missing Data

In general, missing data will not be imputed and the data will be analyzed as they are recorded in the study eCRF. See Appendix 3 for missing value handling of partial dates and treatment - emergent adverse events, and Appendix 4 for determination of prior or concomitant medications. Specifically, missing severity of AEs will be imputed to greatest severity for tabular summarization, and displayed as originally in listings. Missing relationship will be

imputed to "related" for tabular summarization, and displayed as originally in listings. This imputation rule will be applied when summarizing AEs in tables, and missing data will be displayed directly as they are from raw data in listings. For categorical endpoints, the percentage will be calculated based on total number of patients in relevant analysis sets, regardless of whether missing values are present or not. However, if more than 10% of data is missing for one or more key variables, i.e., the safety data, the impact of missing data on the analysis will be discussed, and the pattern of missing data will be explored. If there is evidence of bias in the missing data, and variables that are considered good predictors of the missing data are available, the multiple imputation method at the study level may be used to replace missing values as secondary exploratory analyses. If the multiple imputation method is used, a sensitivity analysis will be carried out comparing results from the complete case analysis (where records with missing data will be dropped) and the full set analysis (with imputed data).

#### 8.11.2 Outliers

All values will be included in the analyses.

#### 8.11.3 Visit Windows

The study protocol gives the overall study schedule and the permissible intervals for these visits as  $\pm$  14 days. Subject's failure to comply with the visit schedule will be regarded as protocol deviation.

#### 8.11.4 Multicenter

This study will be conducted by multiple investigators at 20 centers in 8 countries (Hong Kong, Indonesia, Malaysia, Philippines, Singapore, Taiwan, Thailand and Vietnam).

Data from all centers will be pooled prior to analysis. The analyses will be presented with both pooled data and by region. Hong Kong and Taiwan are considered as greater China region, Indonesia, Malaysia, and Philippines are considered as Asia-Pacific island region, and Singapore, Thailand and Vietnam are considered Indochina Peninsula region. The rule applies to tables, figures and listings.

#### 8.11.5 Retests, Unscheduled Visits and Early Termination Data

In general, for by-visit summaries, data recorded at the scheduled (nominal) visit will be presented. Unscheduled measurements will not be included in by-visit summaries.

In the case of a retest (same visit number assigned), the latest available safety measurement, nearest available efficacy measurement, and lab results closest to that visit will be used for by-visit summaries.

Early termination data will be mapped to the next available visit number for by-visit summaries.

Listings will include scheduled, unscheduled, retest and early discontinuation data.

# 9 DOCUMENT REVISION HISTORY

| Version | <u>Date</u> | <u>Changes</u> | Comment/rationale for change |
|---|---|---|---|
| 0.1 | 24-NOV-2017 | NA | Not applicable – 1 <sup>st</sup> version |
| 0.1 | 02-APR-2018 | 1.Updated to Astellas' template; 2.Added deterioration of HRQoL scores; 3.Added PSA reduction analysis; 4. Updated analyses performed for HRQoL; 5. Revised interim analysis time point to 50 patients followed 1 year; 6. Modified sample | 1, 2, 3, 4 Updated per request from Astellas' team; 5,6 Updated to incorporate protocol amendment 2.0; |
| | | size calculation. | |

# 10 REFERENCES

7015-MA-3072 ELIGANT Protocol Amendment Version 2.0 Dated 16Jan2018.

7015-MA-3072 ELIGANT Protocol Version 1.0 Dated 30May2016.

Case Report Forms Version 2.0 Dated 29May2017.

EORTC QLQ-PR25 Scoring Manual 2.0

# 11 APPENDICES

# 11.1 Appendix 1: Key Contributors and Approvers

# List of Key Contributors and Approvers

# **Key Contributors**

The following contributed to or reviewed this Statistical Analysis Plan as relevant to their indicated discipline or role.

| Primary author (s) | |
|----------------------------|----------|
| PPD | IQVIA |
| Contributors and Reviewers | |
| PPD | IQVIA |
| PPD | IQVIA |
| PPD | Astellas |
| PPD | Astellas |
| PPD | Astellas |
| PPD | Astellas |
| PPD | Astellas |

# **Author and Approver Signatories**

| PPD | IQVIA, was the study statistician for this study. |
|---|---|
| | - |
| PPD | , IQVIA was the biostatistics reviewer of this |
| Statistical Analysis Plan. | |
| This Statistical Analysis Plan wa | as approved by: |
| PPD | , Astellas Pharma Global Development Inc. |
| FFD | , ristellas i hailia Giotai Developineni inc. |
| This Statistical Analysis Plan wa | as approved by: |
| PPD | , Astellas Pharma Singapore Pte Ltd. |
| FFD | , Asicias i latita singapote i e Dio. |

# 11.2 Appendix 2: Programming Conventions for Outputs

# Dates & Times

Depending on data available, dates and times will take the form yyyy-mm-ddThh:mm:ss.

# Spelling Format

English US.

# Presentation of Regions

For outputs, regions will be represented as follows and in that order:

| Region | For Tables and Graphs | For Listings (include if different to tables) |
|---|---|---|
| Region A: Greater China | Region = Greater China | Same as tables |
| Region B: Asia-Pacific<br>Islands | Region = Asia-Pacific<br>Islands | Same as tables |
| Region C: Indochina<br>Peninsula | Region = Indochina<br>Peninsula | Same as tables |
| Total | | |

#### Presentation of Visits

For outputs, visits will be represented as follows and in that order:

| Long Name (default) | Short Name |
|---------------------|------------|
| Screening (Visit 0) | Scr (V0) |
| Baseline (Visit 1) | BL (V1) |
| 3 Month (Visit 2) | M3 (V2) |
| 18 Month (Visit X) | M18 (Vx) |
| Early Withdrawal | WD |

#### Listings

A listings will be ordered by the following (unless otherwise indicated in the template):

- center-subject ID,
- date (where applicable)

# 11.3 Appendix 3: Algorithm for Treatment Emergence of Adverse Events

| START DATE | STOP<br>DATE | ACTION |
|---|---|---|
| Known | Known | If start date < study med start date, then not TEAE |
| | | If start date >= study med start date, then TEAE |
| | Partial | If start date < study med start date, then not TEAE |
| | | If start date >= study med start date, then TEAE |
| | Missing | If start date < study med start date, then not TEAE |
| | | If start date >= study med start date, then TEAE |
| Partial, but known<br>components show that<br>it cannot be on or after<br>study med start date | Known | Not TEAE |
| | Partial | Not TEAE |
| | Missing | Not TEAE |
| Partial, could be on or | Known | If stop date < study med start date, then not TEAE |
| after study med start<br>date | | If stop date >= study med start date, then TEAE |
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: |
| | | If stop date < study med start date, then not TEAE |
| | | If stop date >= study med start date, then TEAE |
| | Missing | Assumed TEAE |
| Missing | Known | If stop date < study med start date, then not TEAE |
| | | If stop date >= study med start date, then TEAE |
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: |
| | | If stop date < study med start date, then not TEAE |

| START DATE | STOP<br>DATE | ACTION |
|------------|--------------|-------------------------------------------------|
| | | If stop date >= study med start date, then TEAE |
| | Missing | Assumed TEAE |

# 11.4 Appendix 4: Algorithm for Prior / Concomitant Medications:

| START<br>DATE | STOP<br>DATE | ACTION |
|---|---|---|
| Known | Known | If stop date < study med start date, assign as prior If stop date >= study med start date and start date <= end of treatment, assign as concomitant If stop date >= study med start date and start date > end of treatment, assign as post study |
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date and start date <= end of treatment, assign as concomitant If stop date >= study med start date and start date > end of treatment, assign as post treatment |
| | Missing | If stop date is missing could never be assumed a prior medication If start date <= end of treatment, assign as concomitant If start date > end of treatment, assign as post treatment |
| Partial | Known | Impute start date as earliest possible date (i.e. first day of month if day unknown or 1st January if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date and start date <= end of treatment, assign as concomitant If stop date >= study med start date and start date > end of treatment, assign as post treatment |

| START<br>DATE | STOP<br>DATE | ACTION |
|---|---|---|
| | Partial | Impute start date as earliest possible date (i.e. first day of month if day unknown or 1st January if day and month are unknown) and impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date and start date <= end of treatment, assign as concomitant If stop date >= study med start date and start date > end of treatment, assign as post treatment |
| | Missing | Impute start date as earliest possible date (i.e. first day of month if day unknown or 1st January if day and month are unknown), then: If stop date is missing could never be assumed a prior medication If start date <= end of treatment, assign as concomitant If start date > end of treatment, assign as post treatment |
| Missing | Known | If stop date < study med start date, assign as prior If stop date >= study med start date, assign as concomitant Cannot be assigned as 'post treatment' |
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date, assign as concomitant Cannot be assigned as 'post treatment' |
| | Missing | Assign as concomitant |

# 11.5 Appendix 5: EQ-5D-5L Value Sets

| 5L profile | Japan | UK | US |
|------------|-------|-------|-------|
| 11111 | 1.000 | 1.000 | 1.000 |
| 11112 | 0.829 | 0.879 | 0.876 |
| 11113 | 0.785 | 0.848 | 0.844 |
| 11114 | 0.761 | 0.635 | 0.700 |
| 11115 | 0.736 | 0.414 | 0.550 |
| 11121 | 0.814 | 0.837 | 0.861 |
| 11122 | 0.740 | 0.768 | 0.820 |
| 11123 | 0.721 | 0.750 | 0.809 |

| 11124 | 0.697 | 0.537 | 0.669 |
|-------|-------|--------|-------|
| 11125 | 0.672 | 0.316 | 0.524 |
| 11131 | 0.768 | 0.796 | 0.827 |
| 11132 | 0.718 | 0.740 | 0.806 |
| 11133 | 0.705 | 0.725 | 0.800 |
| 11134 | 0.681 | 0.512 | 0.661 |
| 11135 | 0.656 | 0.291 | 0.517 |
| 11141 | 0.723 | 0.584 | 0.682 |
| 11142 | 0.673 | 0.527 | 0.663 |
| 11143 | 0.660 | 0.513 | 0.659 |
| 11144 | 0.635 | 0.352 | 0.544 |
| 11145 | 0.611 | 0.186 | 0.426 |
| 11151 | 0.654 | 0.264 | 0.463 |
| 11152 | 0.604 | 0.208 | 0.450 |
| 11153 | 0.591 | 0.193 | 0.446 |
| 11154 | 0.567 | 0.112 | 0.369 |
| 11155 | 0.542 | 0.028 | 0.289 |
| 11211 | 0.843 | 0.906 | 0.888 |
| 11212 | 0.769 | 0.837 | 0.846 |
| 11213 | 0.750 | 0.819 | 0.835 |
| 11214 | 0.726 | 0.606 | 0.695 |
| 11215 | 0.701 | 0.385 | 0.550 |
| 11221 | 0.755 | 0.795 | 0.832 |
| 11222 | 0.700 | 0.736 | 0.796 |
| 11223 | 0.686 | 0.721 | 0.786 |
| 11224 | 0.662 | 0.508 | 0.654 |
| 11225 | 0.637 | 0.287 | 0.517 |
| 11231 | 0.733 | 0.767 | 0.818 |
| 11232 | 0.683 | 0.711 | 0.783 |
| 11233 | 0.670 | 0.696 | 0.774 |
| 11234 | 0.646 | 0.483 | 0.644 |
| 11235 | 0.621 | 0.262 | 0.508 |
| 11241 | 0.687 | 0.555 | 0.676 |
| 11242 | 0.637 | 0.498 | 0.647 |
| 11243 | 0.624 | 0.484 | 0.640 |
| 11244 | 0.600 | 0.323 | 0.532 |
| 11245 | 0.575 | 0.157 | 0.421 |
| 11251 | 0.619 | 0.235 | 0.463 |
| 11252 | 0.569 | 0.179 | 0.443 |
| 11253 | 0.556 | 0.164 | 0.437 |
| 11254 | 0.532 | 0.083 | 0.365 |
| 11255 | 0.507 | -0.001 | 0.289 |
| 11311 | 0.804 | 0.883 | 0.860 |
| 11312 | 0.754 | 0.827 | 0.839 |
| 11313 | 0.741 | 0.812 | 0.833 |
| 11314 | 0.717 | 0.599 | 0.694 |
| 11315 | 0.692 | 0.378 | 0.550 |
| 11321 | 0.740 | 0.785 | 0.825 |
| 11322 | 0.690 | 0.728 | 0.790 |

| 11323 | 0.677 | 0.714 | 0.781 |
|-------|-------|--------|-------|
| 11324 | 0.653 | 0.501 | 0.650 |
| 11325 | 0.628 | 0.280 | 0.515 |
| 11331 | 0.724 | 0.760 | 0.816 |
| 11332 | 0.674 | 0.704 | 0.778 |
| 11333 | 0.661 | 0.689 | 0.768 |
| 11334 | 0.637 | 0.476 | 0.639 |
| 11335 | 0.612 | 0.255 | 0.506 |
| 11341 | 0.679 | 0.548 | 0.675 |
| 11342 | 0.629 | 0.491 | 0.643 |
| 11343 | 0.616 | 0.477 | 0.635 |
| 11344 | 0.591 | 0.316 | 0.529 |
| 11345 | 0.567 | 0.150 | 0.419 |
| 11351 | 0.610 | 0.228 | 0.463 |
| 11352 | 0.560 | 0.172 | 0.441 |
| 11353 | 0.547 | 0.157 | 0.435 |
| 11354 | 0.523 | 0.076 | 0.363 |
| 11355 | 0.498 | -0.008 | 0.289 |
| 11411 | 0.775 | 0.776 | 0.783 |
| 11412 | 0.725 | 0.719 | 0.764 |
| 11413 | 0.712 | 0.705 | 0.759 |
| 11414 | 0.688 | 0.535 | 0.641 |
| 11415 | 0.663 | 0.359 | 0.518 |
| 11421 | 0.711 | 0.677 | 0.751 |
| 11422 | 0.661 | 0.621 | 0.721 |
| 11423 | 0.648 | 0.606 | 0.713 |
| 11424 | 0.624 | 0.437 | 0.601 |
| 11425 | 0.599 | 0.260 | 0.485 |
| 11431 | 0.695 | 0.653 | 0.742 |
| 11432 | 0.645 | 0.596 | 0.710 |
| 11433 | 0.632 | 0.582 | 0.701 |
| 11434 | 0.608 | 0.412 | 0.591 |
| 11435 | 0.583 | 0.236 | 0.477 |
| 11441 | 0.649 | 0.475 | 0.618 |
| 11442 | 0.599 | 0.419 | 0.591 |
| 11443 | 0.586 | 0.404 | 0.584 |
| 11444 | 0.562 | 0.270 | 0.490 |
| 11445 | 0.537 | 0.131 | 0.393 |
| 11451 | 0.581 | 0.209 | 0.431 |
| 11452 | 0.531 | 0.153 | 0.412 |
| 11453 | 0.518 | 0.138 | 0.406 |
| 11454 | 0.494 | 0.057 | 0.338 |
| 11455 | 0.469 | -0.027 | 0.266 |
| 11511 | 0.715 | 0.556 | 0.626 |
| 11512 | 0.665 | 0.500 | 0.613 |
| 11513 | 0.652 | 0.485 | 0.609 |
| 11514 | 0.628 | 0.404 | 0.532 |
| 11515 | 0.603 | 0.320 | 0.452 |
| 11521 | 0.651 | 0.458 | 0.599 |

| 11522 | 0.601 | 0.401 | 0.579 |
|-------|-------|--------|-------|
| 11523 | 0.588 | 0.387 | 0.574 |
| 11524 | 0.564 | 0.306 | 0.501 |
| 11525 | 0.539 | 0.222 | 0.425 |
| 11531 | 0.635 | 0.433 | 0.592 |
| 11532 | 0.585 | 0.377 | 0.571 |
| 11533 | 0.572 | 0.362 | 0.565 |
| 11534 | 0.548 | 0.281 | 0.493 |
| 11535 | 0.523 | 0.197 | 0.418 |
| 11541 | 0.590 | 0.328 | 0.501 |
| 11542 | 0.540 | 0.272 | 0.483 |
| 11543 | 0.527 | 0.257 | 0.478 |
| 11544 | 0.502 | 0.176 | 0.410 |
| 11545 | 0.478 | 0.092 | 0.339 |
| 11551 | 0.521 | 0.170 | 0.365 |
| 11552 | 0.471 | 0.114 | 0.352 |
| 11553 | 0.458 | 0.099 | 0.348 |
| 11554 | 0.434 | 0.018 | 0.285 |
| 11555 | 0.409 | -0.066 | 0.220 |
| 12111 | 0.829 | 0.846 | 0.854 |
| 12112 | 0.758 | 0.779 | 0.815 |
| 12113 | 0.740 | 0.761 | 0.805 |
| 12114 | 0.716 | 0.548 | 0.665 |
| 12115 | 0.691 | 0.327 | 0.520 |
| 12121 | 0.744 | 0.737 | 0.802 |
| 12122 | 0.690 | 0.678 | 0.765 |
| 12123 | 0.676 | 0.663 | 0.756 |
| 12124 | 0.652 | 0.450 | 0.623 |
| 12125 | 0.627 | 0.229 | 0.486 |
| 12131 | 0.723 | 0.709 | 0.789 |
| 12132 | 0.673 | 0.653 | 0.753 |
| 12133 | 0.660 | 0.638 | 0.743 |
| 12134 | 0.636 | 0.425 | 0.613 |
| 12135 | 0.611 | 0.204 | 0.478 |
| 12141 | 0.678 | 0.497 | 0.647 |
| 12142 | 0.628 | 0.441 | 0.617 |
| 12143 | 0.615 | 0.426 | 0.609 |
| 12144 | 0.591 | 0.266 | 0.502 |
| 12145 | 0.566 | 0.099 | 0.390 |
| 12151 | 0.609 | 0.177 | 0.433 |
| 12152 | 0.559 | 0.121 | 0.413 |
| 12153 | 0.546 | 0.106 | 0.408 |
| 12154 | 0.522 | 0.025 | 0.335 |
| 12155 | 0.497 | -0.059 | 0.259 |
| 12211 | 0.773 | 0.806 | 0.828 |
| 12212 | 0.719 | 0.748 | 0.792 |
| 12213 | 0.705 | 0.733 | 0.782 |
| 12214 | 0.681 | 0.520 | 0.650 |
| 12215 | 0.656 | 0.299 | 0.513 |
| | | | 2.2.0 |

| 12221 | 0.705 | 0.706 | 0.778 |
|-------|-------|--------|-------|
| 12222 | 0.654 | 0.649 | 0.731 |
| 12223 | 0.641 | 0.634 | 0.719 |
| 12224 | 0.617 | 0.421 | 0.595 |
| 12225 | 0.592 | 0.200 | 0.467 |
| 12231 | 0.688 | 0.681 | 0.765 |
| 12232 | 0.638 | 0.624 | 0.716 |
| 12233 | 0.625 | 0.610 | 0.703 |
| 12234 | 0.601 | 0.397 | 0.581 |
| 12235 | 0.576 | 0.176 | 0.455 |
| 12241 | 0.642 | 0.468 | 0.630 |
| 12242 | 0.592 | 0.412 | 0.587 |
| 12243 | 0.579 | 0.397 | 0.576 |
| 12244 | 0.555 | 0.237 | 0.477 |
| 12245 | 0.530 | 0.071 | 0.374 |
| 12251 | 0.574 | 0.149 | 0.426 |
| 12252 | 0.524 | 0.092 | 0.393 |
| 12253 | 0.511 | 0.078 | 0.385 |
| 12254 | 0.487 | -0.003 | 0.320 |
| 12255 | 0.462 | -0.088 | 0.252 |
| 12311 | 0.759 | 0.796 | 0.822 |
| 12312 | 0.709 | 0.740 | 0.786 |
| 12313 | 0.696 | 0.725 | 0.776 |
| 12314 | 0.672 | 0.512 | 0.646 |
| 12315 | 0.647 | 0.291 | 0.511 |
| 12321 | 0.695 | 0.698 | 0.772 |
| 12322 | 0.645 | 0.642 | 0.723 |
| 12323 | 0.632 | 0.627 | 0.710 |
| 12324 | 0.608 | 0.414 | 0.588 |
| 12325 | 0.583 | 0.193 | 0.462 |
| 12331 | 0.679 | 0.673 | 0.759 |
| 12332 | 0.629 | 0.617 | 0.707 |
| 12333 | 0.616 | 0.602 | 0.693 |
| 12334 | 0.592 | 0.389 | 0.574 |
| 12335 | 0.567 | 0.168 | 0.449 |
| 12341 | 0.634 | 0.461 | 0.625 |
| 12342 | 0.584 | 0.405 | 0.580 |
| 12343 | 0.571 | 0.390 | 0.568 |
| 12344 | 0.547 | 0.230 | 0.471 |
| 12345 | 0.522 | 0.063 | 0.370 |
| 12351 | 0.565 | 0.141 | 0.424 |
| 12352 | 0.515 | 0.085 | 0.388 |
| 12353 | 0.502 | 0.070 | 0.379 |
| 12354 | 0.478 | -0.011 | 0.316 |
| 12355 | 0.453 | -0.095 | 0.250 |
| 12411 | 0.730 | 0.689 | 0.748 |
| 12412 | 0.680 | 0.633 | 0.717 |
| 12413 | 0.667 | 0.618 | 0.709 |
| 12414 | 0.643 | 0.448 | 0.597 |

| 12415 | 0.618 | 0.272 | 0.482 |
|-------|-------|--------|-------|
| 12421 | 0.666 | 0.591 | 0.703 |
| 12422 | 0.616 | 0.534 | 0.659 |
| 12423 | 0.603 | 0.520 | 0.648 |
| 12424 | 0.579 | 0.350 | 0.545 |
| 12425 | 0.554 | 0.174 | 0.438 |
| 12431 | 0.650 | 0.566 | 0.692 |
| 12432 | 0.600 | 0.510 | 0.645 |
| 12433 | 0.587 | 0.495 | 0.632 |
| 12434 | 0.563 | 0.325 | 0.531 |
| 12435 | 0.538 | 0.149 | 0.427 |
| 12441 | 0.604 | 0.389 | 0.573 |
| 12442 | 0.554 | 0.332 | 0.533 |
| 12443 | 0.541 | 0.318 | 0.522 |
| 12444 | 0.517 | 0.184 | 0.437 |
| 12445 | 0.492 | 0.044 | 0.348 |
| 12451 | 0.536 | 0.122 | 0.395 |
| 12452 | 0.486 | 0.066 | 0.364 |
| 12453 | 0.473 | 0.051 | 0.356 |
| 12454 | 0.449 | -0.030 | 0.295 |
| 12455 | 0.424 | -0.114 | 0.230 |
| 12511 | 0.670 | 0.469 | 0.596 |
| 12512 | 0.620 | 0.413 | 0.576 |
| 12513 | 0.607 | 0.398 | 0.571 |
| 12514 | 0.583 | 0.317 | 0.498 |
| 12515 | 0.558 | 0.233 | 0.422 |
| 12521 | 0.606 | 0.371 | 0.562 |
| 12522 | 0.556 | 0.315 | 0.529 |
| 12523 | 0.543 | 0.300 | 0.521 |
| 12524 | 0.519 | 0.219 | 0.456 |
| 12525 | 0.494 | 0.135 | 0.388 |
| 12531 | 0.590 | 0.346 | 0.554 |
| 12532 | 0.540 | 0.290 | 0.518 |
| 12533 | 0.527 | 0.275 | 0.508 |
| 12534 | 0.503 | 0.194 | 0.445 |
| 12535 | 0.478 | 0.110 | 0.380 |
| 12541 | 0.545 | 0.241 | 0.466 |
| 12542 | 0.495 | 0.185 | 0.437 |
| 12543 | 0.482 | 0.170 | 0.429 |
| 12544 | 0.458 | 0.089 | 0.368 |
| 12545 | 0.433 | 0.005 | 0.304 |
| 12551 | 0.476 | 0.083 | 0.335 |
| 12552 | 0.426 | 0.027 | 0.315 |
| 12553 | 0.413 | 0.012 | 0.310 |
| 12554 | 0.389 | -0.069 | 0.251 |
| 12555 | 0.364 | -0.153 | 0.190 |
| 13111 | 0.794 | 0.815 | 0.825 |
| 13112 | 0.744 | 0.759 | 0.803 |
| 13113 | 0.731 | 0.744 | 0.797 |
| 13114 | 0.707 | 0.531 | 0.658 |
|-------|-------|--------|-------|
| 13115 | 0.682 | 0.310 | 0.514 |
| 13121 | 0.730 | 0.717 | 0.790 |
| 13122 | 0.680 | 0.660 | 0.754 |
| 13123 | 0.667 | 0.646 | 0.745 |
| 13124 | 0.643 | 0.433 | 0.614 |
| 13125 | 0.618 | 0.212 | 0.479 |
| 13131 | 0.714 | 0.692 | 0.781 |
| 13132 | 0.664 | 0.636 | 0.742 |
| 13133 | 0.651 | 0.621 | 0.732 |
| 13134 | 0.627 | 0.408 | 0.603 |
| 13135 | 0.602 | 0.187 | 0.470 |
| 13141 | 0.669 | 0.480 | 0.640 |
| 13142 | 0.619 | 0.423 | 0.608 |
| 13143 | 0.606 | 0.409 | 0.599 |
| 13144 | 0.581 | 0.248 | 0.493 |
| 13145 | 0.557 | 0.082 | 0.383 |
| 13151 | 0.600 | 0.160 | 0.427 |
| 13152 | 0.550 | 0.104 | 0.406 |
| 13153 | 0.537 | 0.089 | 0.400 |
| 13154 | 0.513 | 0.008 | 0.328 |
| 13155 | 0.488 | -0.076 | 0.253 |
| 13211 | 0.759 | 0.786 | 0.816 |
| 13212 | 0.709 | 0.730 | 0.781 |
| 13213 | 0.696 | 0.715 | 0.771 |
| 13214 | 0.672 | 0.502 | 0.641 |
| 13215 | 0.647 | 0.281 | 0.505 |
| 13221 | 0.695 | 0.688 | 0.767 |
| 13222 | 0.645 | 0.631 | 0.718 |
| 13223 | 0.632 | 0.617 | 0.705 |
| 13224 | 0.608 | 0.404 | 0.583 |
| 13225 | 0.583 | 0.183 | 0.456 |
| 13231 | 0.679 | 0.663 | 0.755 |
| 13232 | 0.629 | 0.607 | 0.702 |
| 13233 | 0.616 | 0.592 | 0.689 |
| 13234 | 0.592 | 0.379 | 0.569 |
| 13235 | 0.567 | 0.158 | 0.444 |
| 13241 | 0.633 | 0.451 | 0.620 |
| 13242 | 0.583 | 0.394 | 0.575 |
| 13243 | 0.570 | 0.380 | 0.563 |
| 13244 | 0.546 | 0.219 | 0.466 |
| 13245 | 0.521 | 0.053 | 0.364 |
| 13251 | 0.565 | 0.131 | 0.418 |
| 13252 | 0.515 | 0.075 | 0.383 |
| 13253 | 0.502 | 0.060 | 0.374 |
| 13254 | 0.478 | -0.021 | 0.311 |
| 13255 | 0.453 | -0.105 | 0.244 |
| 13311 | 0.750 | 0.779 | 0.814 |
| 13312 | 0.700 | 0.723 | 0.775 |

| 13313 | 0.687 | 0.708 | 0.765 |
|-------|-------|--------|-------|
| 13314 | 0.663 | 0.495 | 0.636 |
| 13315 | 0.638 | 0.274 | 0.503 |
| 13321 | 0.686 | 0.681 | 0.761 |
| 13322 | 0.636 | 0.624 | 0.709 |
| 13323 | 0.623 | 0.610 | 0.695 |
| 13324 | 0.599 | 0.397 | 0.575 |
| 13325 | 0.574 | 0.176 | 0.451 |
| 13331 | 0.670 | 0.656 | 0.748 |
| 13332 | 0.620 | 0.600 | 0.693 |
| 13333 | 0.607 | 0.585 | 0.678 |
| 13334 | 0.583 | 0.372 | 0.560 |
| 13335 | 0.558 | 0.151 | 0.438 |
| 13341 | 0.625 | 0.444 | 0.615 |
| 13342 | 0.575 | 0.387 | 0.567 |
| 13343 | 0.562 | 0.373 | 0.554 |
| 13344 | 0.537 | 0.212 | 0.459 |
| 13345 | 0.513 | 0.046 | 0.360 |
| 13351 | 0.556 | 0.124 | 0.416 |
| 13352 | 0.506 | 0.068 | 0.378 |
| 13353 | 0.493 | 0.053 | 0.368 |
| 13354 | 0.469 | -0.028 | 0.306 |
| 13355 | 0.444 | -0.112 | 0.242 |
| 13411 | 0.721 | 0.672 | 0.740 |
| 13412 | 0.671 | 0.615 | 0.707 |
| 13413 | 0.658 | 0.601 | 0.699 |
| 13414 | 0.634 | 0.431 | 0.589 |
| 13415 | 0.609 | 0.255 | 0.474 |
| 13421 | 0.657 | 0.573 | 0.693 |
| 13422 | 0.607 | 0.517 | 0.647 |
| 13423 | 0.594 | 0.502 | 0.635 |
| 13424 | 0.570 | 0.333 | 0.533 |
| 13425 | 0.545 | 0.156 | 0.428 |
| 13431 | 0.641 | 0.549 | 0.682 |
| 13432 | 0.591 | 0.492 | 0.632 |
| 13433 | 0.578 | 0.478 | 0.619 |
| 13434 | 0.554 | 0.308 | 0.519 |
| 13435 | 0.529 | 0.132 | 0.416 |
| 13441 | 0.595 | 0.371 | 0.564 |
| 13442 | 0.545 | 0.315 | 0.521 |
| 13443 | 0.532 | 0.300 | 0.510 |
| 13444 | 0.508 | 0.166 | 0.426 |
| 13445 | 0.483 | 0.027 | 0.339 |
| 13451 | 0.527 | 0.105 | 0.387 |
| 13452 | 0.477 | 0.049 | 0.355 |
| 13453 | 0.464 | 0.034 | 0.346 |
| 13454 | 0.440 | -0.047 | 0.286 |
| 13455 | 0.415 | -0.131 | 0.223 |
| 13511 | 0.661 | 0.452 | 0.590 |

| 13512 | 0.611 | 0.396 | 0.569 |
|-------|-------|--------|-------|
| 13513 | 0.598 | 0.381 | 0.563 |
| 13514 | 0.574 | 0.300 | 0.491 |
| 13515 | 0.549 | 0.216 | 0.416 |
| 13521 | 0.597 | 0.354 | 0.555 |
| 13522 | 0.547 | 0.297 | 0.519 |
| 13523 | 0.534 | 0.283 | 0.510 |
| 13524 | 0.510 | 0.202 | 0.447 |
| 13525 | 0.485 | 0.118 | 0.381 |
| 13531 | 0.581 | 0.329 | 0.546 |
| 13532 | 0.531 | 0.273 | 0.507 |
| 13533 | 0.518 | 0.258 | 0.497 |
| 13534 | 0.494 | 0.177 | 0.436 |
| 13535 | 0.469 | 0.093 | 0.372 |
| 13541 | 0.536 | 0.224 | 0.459 |
| 13542 | 0.486 | 0.168 | 0.427 |
| 13543 | 0.473 | 0.153 | 0.419 |
| 13544 | 0.448 | 0.072 | 0.359 |
| 13545 | 0.424 | -0.012 | 0.297 |
| 13551 | 0.467 | 0.066 | 0.329 |
| 13552 | 0.417 | 0.010 | 0.308 |
| 13553 | 0.404 | -0.005 | 0.302 |
| 13554 | 0.380 | -0.086 | 0.244 |
| 13555 | 0.355 | -0.170 | 0.184 |
| 14111 | 0.782 | 0.723 | 0.753 |
| 14112 | 0.732 | 0.667 | 0.733 |
| 14113 | 0.719 | 0.652 | 0.728 |
| 14114 | 0.695 | 0.471 | 0.604 |
| 14115 | 0.670 | 0.283 | 0.475 |
| 14121 | 0.718 | 0.624 | 0.720 |
| 14122 | 0.668 | 0.568 | 0.688 |
| 14123 | 0.655 | 0.553 | 0.680 |
| 14124 | 0.631 | 0.373 | 0.563 |
| 14125 | 0.606 | 0.185 | 0.442 |
| 14131 | 0.702 | 0.600 | 0.712 |
| 14132 | 0.652 | 0.544 | 0.677 |
| 14133 | 0.639 | 0.529 | 0.668 |
| 14134 | 0.615 | 0.348 | 0.553 |
| 14135 | 0.590 | 0.160 | 0.434 |
| 14141 | 0.657 | 0.414 | 0.583 |
| 14142 | 0.607 | 0.357 | 0.554 |
| 14143 | 0.594 | 0.343 | 0.546 |
| 14144 | 0.570 | 0.202 | 0.450 |
| 14145 | 0.545 | 0.055 | 0.349 |
| 14151 | 0.588 | 0.133 | 0.388 |
| 14152 | 0.538 | 0.077 | 0.369 |
| 14153 | 0.525 | 0.062 | 0.364 |
| 14154 | 0.501 | -0.019 | 0.294 |
| 14155 | 0.476 | -0.103 | 0.221 |

| 14211 | 0.747 | 0.694 | 0.746 |
|-------|-------|--------|-------|
| 14212 | 0.697 | 0.638 | 0.715 |
| 14213 | 0.684 | 0.623 | 0.706 |
| 14214 | 0.660 | 0.442 | 0.590 |
| 14215 | 0.635 | 0.254 | 0.469 |
| 14221 | 0.683 | 0.596 | 0.701 |
| 14222 | 0.633 | 0.539 | 0.656 |
| 14223 | 0.620 | 0.525 | 0.644 |
| 14224 | 0.596 | 0.344 | 0.536 |
| 14225 | 0.571 | 0.156 | 0.423 |
| 14231 | 0.667 | 0.571 | 0.690 |
| 14232 | 0.617 | 0.515 | 0.641 |
| 14233 | 0.604 | 0.500 | 0.629 |
| 14234 | 0.580 | 0.319 | 0.523 |
| 14235 | 0.555 | 0.131 | 0.412 |
| 14241 | 0.622 | 0.385 | 0.567 |
| 14242 | 0.572 | 0.328 | 0.525 |
| 14243 | 0.559 | 0.314 | 0.514 |
| 14244 | 0.535 | 0.173 | 0.426 |
| 14245 | 0.510 | 0.026 | 0.333 |
| 14251 | 0.553 | 0.104 | 0.382 |
| 14252 | 0.503 | 0.048 | 0.350 |
| 14253 | 0.490 | 0.033 | 0.342 |
| 14254 | 0.466 | -0.048 | 0.280 |
| 14255 | 0.441 | -0.132 | 0.215 |
| 14311 | 0.738 | 0.687 | 0.745 |
| 14312 | 0.688 | 0.631 | 0.710 |
| 14313 | 0.675 | 0.616 | 0.701 |
| 14314 | 0.651 | 0.435 | 0.586 |
| 14315 | 0.626 | 0.247 | 0.467 |
| 14321 | 0.674 | 0.588 | 0.696 |
| 14322 | 0.624 | 0.532 | 0.648 |
| 14323 | 0.611 | 0.517 | 0.635 |
| 14324 | 0.587 | 0.337 | 0.529 |
| 14325 | 0.562 | 0.149 | 0.419 |
| 14331 | 0.658 | 0.564 | 0.684 |
| 14332 | 0.608 | 0.508 | 0.633 |
| 14333 | 0.595 | 0.493 | 0.619 |
| 14334 | 0.571 | 0.312 | 0.515 |
| 14335 | 0.546 | 0.124 | 0.407 |
| 14341 | 0.613 | 0.378 | 0.563 |
| 14342 | 0.563 | 0.321 | 0.518 |
| 14343 | 0.550 | 0.307 | 0.506 |
| 14344 | 0.526 | 0.166 | 0.420 |
| 14345 | 0.501 | 0.019 | 0.330 |
| 14351 | 0.544 | 0.097 | 0.380 |
| 14352 | 0.494 | 0.041 | 0.346 |
| 14353 | 0.481 | 0.026 | 0.337 |
| 14354 | 0.457 | -0.055 | 0.276 |

| 14355 | 0.432 | -0.139 | 0.213 |
|-------|-------|--------|-------|
| 14411 | 0.709 | 0.601 | 0.681 |
| 14412 | 0.659 | 0.545 | 0.651 |
| 14413 | 0.646 | 0.530 | 0.644 |
| 14414 | 0.622 | 0.382 | 0.544 |
| 14415 | 0.597 | 0.228 | 0.440 |
| 14421 | 0.645 | 0.502 | 0.638 |
| 14422 | 0.595 | 0.446 | 0.595 |
| 14423 | 0.582 | 0.431 | 0.584 |
| 14424 | 0.558 | 0.283 | 0.492 |
| 14425 | 0.533 | 0.130 | 0.397 |
| 14431 | 0.629 | 0.478 | 0.627 |
| 14432 | 0.579 | 0.422 | 0.581 |
| 14433 | 0.566 | 0.407 | 0.569 |
| 14434 | 0.542 | 0.259 | 0.479 |
| 14435 | 0.517 | 0.105 | 0.386 |
| 14441 | 0.584 | 0.318 | 0.517 |
| 14442 | 0.534 | 0.262 | 0.478 |
| 14443 | 0.521 | 0.247 | 0.468 |
| 14444 | 0.497 | 0.126 | 0.390 |
| 14445 | 0.472 | 0.000 | 0.310 |
| 14451 | 0.515 | 0.078 | 0.353 |
| 14452 | 0.465 | 0.022 | 0.324 |
| 14453 | 0.452 | 0.007 | 0.316 |
| 14454 | 0.428 | -0.074 | 0.257 |
| 14455 | 0.403 | -0.158 | 0.196 |
| 14511 | 0.649 | 0.425 | 0.551 |
| 14512 | 0.599 | 0.369 | 0.532 |
| 14513 | 0.586 | 0.354 | 0.527 |
| 14514 | 0.562 | 0.273 | 0.457 |
| 14515 | 0.537 | 0.189 | 0.384 |
| 14521 | 0.585 | 0.327 | 0.518 |
| 14522 | 0.535 | 0.270 | 0.486 |
| 14523 | 0.522 | 0.256 | 0.478 |
| 14524 | 0.498 | 0.175 | 0.416 |
| 14525 | 0.473 | 0.091 | 0.351 |
| 14531 | 0.569 | 0.302 | 0.510 |
| 14532 | 0.519 | 0.246 | 0.475 |
| 14533 | 0.506 | 0.231 | 0.466 |
| 14534 | 0.482 | 0.150 | 0.406 |
| 14535 | 0.457 | 0.066 | 0.343 |
| 14541 | 0.524 | 0.197 | 0.425 |
| 14542 | 0.474 | 0.141 | 0.396 |
| 14543 | 0.461 | 0.126 | 0.389 |
| 14544 | 0.437 | 0.045 | 0.331 |
| 14545 | 0.412 | -0.039 | 0.270 |
| 14551 | 0.455 | 0.039 | 0.297 |
| 14552 | 0.405 | -0.017 | 0.278 |
| 14553 | 0.392 | -0.032 | 0.273 |

| 14554 | 0.368 | -0.113 | 0.217 |
|-------|-------|--------|-------|
| 14555 | 0.343 | -0.197 | 0.160 |
| 15111 | 0.746 | 0.436 | 0.529 |
| 15112 | 0.696 | 0.380 | 0.516 |
| 15113 | 0.683 | 0.365 | 0.512 |
| 15114 | 0.659 | 0.284 | 0.435 |
| 15115 | 0.634 | 0.200 | 0.355 |
| 15121 | 0.682 | 0.338 | 0.503 |
| 15122 | 0.632 | 0.281 | 0.482 |
| 15123 | 0.619 | 0.267 | 0.477 |
| 15124 | 0.595 | 0.186 | 0.404 |
| 15125 | 0.570 | 0.102 | 0.328 |
| 15131 | 0.666 | 0.313 | 0.496 |
| 15132 | 0.616 | 0.257 | 0.474 |
| 15133 | 0.603 | 0.242 | 0.468 |
| 15134 | 0.579 | 0.161 | 0.396 |
| 15135 | 0.554 | 0.077 | 0.321 |
| 15141 | 0.621 | 0.208 | 0.405 |
| 15142 | 0.571 | 0.152 | 0.386 |
| 15143 | 0.558 | 0.137 | 0.381 |
| 15144 | 0.533 | 0.056 | 0.313 |
| 15145 | 0.509 | -0.028 | 0.242 |
| 15151 | 0.552 | 0.050 | 0.268 |
| 15152 | 0.502 | -0.006 | 0.255 |
| 15153 | 0.489 | -0.021 | 0.251 |
| 15154 | 0.465 | -0.102 | 0.188 |
| 15155 | 0.440 | -0.186 | 0.123 |
| 15211 | 0.711 | 0.407 | 0.529 |
| 15212 | 0.661 | 0.351 | 0.509 |
| 15213 | 0.648 | 0.336 | 0.503 |
| 15214 | 0.624 | 0.255 | 0.430 |
| 15215 | 0.599 | 0.171 | 0.354 |
| 15221 | 0.647 | 0.309 | 0.496 |
| 15222 | 0.597 | 0.252 | 0.463 |
| 15223 | 0.584 | 0.238 | 0.454 |
| 15224 | 0.560 | 0.157 | 0.389 |
| 15225 | 0.535 | 0.073 | 0.321 |
| 15231 | 0.631 | 0.284 | 0.487 |
| 15232 | 0.581 | 0.228 | 0.452 |
| 15233 | 0.568 | 0.213 | 0.442 |
| 15234 | 0.544 | 0.132 | 0.379 |
| 15235 | 0.519 | 0.048 | 0.312 |
| 15241 | 0.585 | 0.179 | 0.400 |
| 15242 | 0.535 | 0.123 | 0.370 |
| 15243 | 0.522 | 0.108 | 0.362 |
| 15244 | 0.498 | 0.027 | 0.301 |
| 15245 | 0.473 | -0.057 | 0.237 |
| 15251 | 0.517 | 0.021 | 0.268 |
| 15252 | 0.467 | -0.035 | 0.248 |

| 15253 | 0.454 | -0.050 | 0.242 |
|-------|-------|--------|-------|
| 15254 | 0.430 | -0.131 | 0.184 |
| 15255 | 0.405 | -0.215 | 0.123 |
| 15311 | 0.702 | 0.400 | 0.529 |
| 15312 | 0.652 | 0.344 | 0.507 |
| 15313 | 0.639 | 0.329 | 0.501 |
| 15314 | 0.615 | 0.248 | 0.429 |
| 15315 | 0.590 | 0.164 | 0.354 |
| 15321 | 0.638 | 0.302 | 0.494 |
| 15322 | 0.588 | 0.245 | 0.458 |
| 15323 | 0.575 | 0.231 | 0.449 |
| 15324 | 0.551 | 0.150 | 0.385 |
| 15325 | 0.526 | 0.066 | 0.319 |
| 15331 | 0.622 | 0.277 | 0.485 |
| 15332 | 0.572 | 0.221 | 0.446 |
| 15333 | 0.559 | 0.206 | 0.436 |
| 15334 | 0.535 | 0.125 | 0.374 |
| 15335 | 0.510 | 0.041 | 0.310 |
| 15341 | 0.577 | 0.172 | 0.398 |
| 15342 | 0.527 | 0.116 | 0.366 |
| 15343 | 0.514 | 0.101 | 0.358 |
| 15344 | 0.489 | 0.020 | 0.298 |
| 15345 | 0.465 | -0.064 | 0.235 |
| 15351 | 0.508 | 0.014 | 0.268 |
| 15352 | 0.458 | -0.042 | 0.246 |
| 15353 | 0.445 | -0.057 | 0.240 |
| 15354 | 0.421 | -0.138 | 0.183 |
| 15355 | 0.396 | -0.222 | 0.123 |
| 15411 | 0.673 | 0.381 | 0.497 |
| 15412 | 0.623 | 0.325 | 0.478 |
| 15413 | 0.610 | 0.310 | 0.472 |
| 15414 | 0.586 | 0.229 | 0.403 |
| 15415 | 0.561 | 0.145 | 0.332 |
| 15421 | 0.609 | 0.282 | 0.464 |
| 15422 | 0.559 | 0.226 | 0.434 |
| 15423 | 0.546 | 0.211 | 0.426 |
| 15424 | 0.522 | 0.130 | 0.364 |
| 15425 | 0.497 | 0.046 | 0.299 |
| 15431 | 0.593 | 0.258 | 0.456 |
| 15432 | 0.543 | 0.202 | 0.423 |
| 15433 | 0.530 | 0.187 | 0.414 |
| 15434 | 0.506 | 0.106 | 0.354 |
| 15435 | 0.481 | 0.022 | 0.291 |
| 15441 | 0.547 | 0.153 | 0.372 |
| 15442 | 0.497 | 0.097 | 0.344 |
| 15443 | 0.484 | 0.082 | 0.337 |
| 15444 | 0.460 | 0.001 | 0.279 |
| 15445 | 0.435 | -0.083 | 0.219 |
| 15451 | 0.479 | -0.005 | 0.245 |

| 15452 | 0.429 | -0.061 | 0.226 |
|-------|-------|--------|-------|
| 15453 | 0.416 | -0.076 | 0.221 |
| 15454 | 0.392 | -0.157 | 0.167 |
| 15455 | 0.367 | -0.241 | 0.110 |
| 15511 | 0.613 | 0.342 | 0.431 |
| 15512 | 0.563 | 0.286 | 0.418 |
| 15513 | 0.550 | 0.271 | 0.414 |
| 15514 | 0.526 | 0.190 | 0.351 |
| 15515 | 0.501 | 0.106 | 0.286 |
| 15521 | 0.549 | 0.244 | 0.404 |
| 15522 | 0.499 | 0.187 | 0.384 |
| 15523 | 0.486 | 0.173 | 0.379 |
| 15524 | 0.462 | 0.092 | 0.320 |
| 15525 | 0.437 | 0.008 | 0.260 |
| 15531 | 0.533 | 0.219 | 0.397 |
| 15532 | 0.483 | 0.163 | 0.376 |
| 15533 | 0.470 | 0.148 | 0.370 |
| 15534 | 0.446 | 0.067 | 0.313 |
| 15535 | 0.421 | -0.017 | 0.253 |
| 15541 | 0.488 | 0.114 | 0.318 |
| 15542 | 0.438 | 0.058 | 0.300 |
| 15543 | 0.425 | 0.043 | 0.295 |
| 15544 | 0.400 | -0.038 | 0.241 |
| 15545 | 0.376 | -0.122 | 0.186 |
| 15551 | 0.419 | -0.044 | 0.199 |
| 15552 | 0.369 | -0.100 | 0.186 |
| 15553 | 0.356 | -0.115 | 0.182 |
| 15554 | 0.332 | -0.196 | 0.134 |
| 15555 | 0.307 | -0.280 | 0.084 |
| 21111 | 0.813 | 0.877 | 0.880 |
| 21112 | 0.742 | 0.809 | 0.840 |
| 21113 | 0.723 | 0.791 | 0.830 |
| 21114 | 0.699 | 0.578 | 0.690 |
| 21115 | 0.674 | 0.357 | 0.544 |
| 21121 | 0.728 | 0.767 | 0.826 |
| 21122 | 0.673 | 0.708 | 0.790 |
| 21123 | 0.659 | 0.693 | 0.780 |
| 21124 | 0.635 | 0.480 | 0.648 |
| 21125 | 0.610 | 0.259 | 0.511 |
| 21131 | 0.706 | 0.739 | 0.813 |
| 21132 | 0.656 | 0.683 | 0.777 |
| 21133 | 0.643 | 0.668 | 0.768 |
| 21134 | 0.619 | 0.455 | 0.638 |
| 21135 | 0.594 | 0.234 | 0.502 |
| 21141 | 0.661 | 0.527 | 0.671 |
| 21142 | 0.611 | 0.470 | 0.641 |
| 21143 | 0.598 | 0.456 | 0.634 |
| 21144 | 0.574 | 0.296 | 0.526 |
| 21145 | 0.549 | 0.129 | 0.415 |

| 21151 | 0.592 | 0.207 | 0.457 |
|-------|-------|--------|-------|
| 21152 | 0.542 | 0.151 | 0.437 |
| 21153 | 0.529 | 0.136 | 0.432 |
| 21154 | 0.505 | 0.055 | 0.359 |
| 21155 | 0.480 | -0.029 | 0.283 |
| 21211 | 0.756 | 0.836 | 0.853 |
| 21212 | 0.702 | 0.778 | 0.816 |
| 21213 | 0.688 | 0.762 | 0.807 |
| 21214 | 0.664 | 0.549 | 0.675 |
| 21215 | 0.639 | 0.328 | 0.538 |
| 21221 | 0.688 | 0.735 | 0.803 |
| 21222 | 0.637 | 0.679 | 0.756 |
| 21223 | 0.624 | 0.664 | 0.744 |
| 21224 | 0.600 | 0.451 | 0.620 |
| 21225 | 0.575 | 0.230 | 0.491 |
| 21231 | 0.671 | 0.710 | 0.790 |
| 21232 | 0.621 | 0.654 | 0.741 |
| 21233 | 0.608 | 0.639 | 0.728 |
| 21234 | 0.584 | 0.426 | 0.606 |
| 21235 | 0.559 | 0.205 | 0.480 |
| 21241 | 0.626 | 0.498 | 0.655 |
| 21242 | 0.576 | 0.442 | 0.612 |
| 21243 | 0.563 | 0.427 | 0.601 |
| 21244 | 0.538 | 0.267 | 0.502 |
| 21245 | 0.514 | 0.100 | 0.398 |
| 21251 | 0.557 | 0.178 | 0.451 |
| 21252 | 0.507 | 0.122 | 0.418 |
| 21253 | 0.494 | 0.107 | 0.409 |
| 21254 | 0.470 | 0.026 | 0.344 |
| 21255 | 0.445 | -0.058 | 0.276 |
| 21311 | 0.742 | 0.826 | 0.846 |
| 21312 | 0.692 | 0.770 | 0.810 |
| 21313 | 0.679 | 0.755 | 0.801 |
| 21314 | 0.655 | 0.542 | 0.671 |
| 21315 | 0.630 | 0.321 | 0.536 |
| 21321 | 0.678 | 0.728 | 0.797 |
| 21322 | 0.628 | 0.671 | 0.748 |
| 21323 | 0.615 | 0.657 | 0.735 |
| 21324 | 0.591 | 0.444 | 0.613 |
| 21325 | 0.566 | 0.223 | 0.486 |
| 21331 | 0.662 | 0.703 | 0.785 |
| 21332 | 0.612 | 0.647 | 0.732 |
| 21333 | 0.599 | 0.632 | 0.719 |
| 21334 | 0.575 | 0.419 | 0.599 |
| 21335 | 0.550 | 0.198 | 0.474 |
| 21341 | 0.617 | 0.491 | 0.651 |
| 21342 | 0.567 | 0.434 | 0.605 |
| 21343 | 0.554 | 0.420 | 0.593 |
| 21344 | 0.530 | 0.260 | 0.495 |

| 21345 | 0.505 | 0.093 | 0.394 |
|-------|-------|--------|-------|
| 21351 | 0.548 | 0.171 | 0.449 |
| 21352 | 0.498 | 0.115 | 0.413 |
| 21353 | 0.485 | 0.100 | 0.404 |
| 21354 | 0.461 | 0.019 | 0.340 |
| 21355 | 0.436 | -0.065 | 0.274 |
| 21411 | 0.713 | 0.719 | 0.772 |
| 21412 | 0.663 | 0.663 | 0.741 |
| 21413 | 0.650 | 0.648 | 0.733 |
| 21414 | 0.626 | 0.478 | 0.622 |
| 21415 | 0.601 | 0.302 | 0.507 |
| 21421 | 0.649 | 0.620 | 0.728 |
| 21422 | 0.599 | 0.564 | 0.684 |
| 21423 | 0.586 | 0.549 | 0.673 |
| 21424 | 0.562 | 0.380 | 0.569 |
| 21425 | 0.537 | 0.204 | 0.462 |
| 21431 | 0.633 | 0.596 | 0.717 |
| 21432 | 0.583 | 0.540 | 0.670 |
| 21433 | 0.570 | 0.525 | 0.658 |
| 21434 | 0.546 | 0.355 | 0.556 |
| 21435 | 0.521 | 0.179 | 0.451 |
| 21441 | 0.588 | 0.419 | 0.598 |
| 21442 | 0.538 | 0.362 | 0.558 |
| 21443 | 0.525 | 0.348 | 0.547 |
| 21444 | 0.501 | 0.213 | 0.462 |
| 21445 | 0.476 | 0.074 | 0.373 |
| 21451 | 0.519 | 0.152 | 0.420 |
| 21452 | 0.469 | 0.096 | 0.389 |
| 21453 | 0.456 | 0.081 | 0.381 |
| 21454 | 0.432 | 0.000 | 0.319 |
| 21455 | 0.407 | -0.084 | 0.255 |
| 21511 | 0.653 | 0.499 | 0.620 |
| 21512 | 0.603 | 0.443 | 0.600 |
| 21513 | 0.590 | 0.428 | 0.595 |
| 21514 | 0.566 | 0.347 | 0.522 |
| 21515 | 0.541 | 0.263 | 0.446 |
| 21521 | 0.589 | 0.401 | 0.586 |
| 21522 | 0.539 | 0.344 | 0.554 |
| 21523 | 0.526 | 0.330 | 0.546 |
| 21524 | 0.502 | 0.249 | 0.480 |
| 21525 | 0.477 | 0.165 | 0.412 |
| 21531 | 0.573 | 0.376 | 0.578 |
| 21532 | 0.523 | 0.320 | 0.543 |
| 21533 | 0.510 | 0.305 | 0.534 |
| 21534 | 0.486 | 0.224 | 0.470 |
| 21535 | 0.461 | 0.140 | 0.404 |
| 21541 | 0.528 | 0.271 | 0.491 |
| 21542 | 0.478 | 0.215 | 0.462 |
| 21543 | 0.465 | 0.200 | 0.454 |

| 21544 | 0.441 | 0.119 | 0.392 |
|-------|-------|--------|-------|
| 21545 | 0.416 | 0.035 | 0.329 |
| 21551 | 0.459 | 0.113 | 0.359 |
| 21552 | 0.409 | 0.057 | 0.339 |
| 21553 | 0.396 | 0.042 | 0.334 |
| 21554 | 0.372 | -0.039 | 0.276 |
| 21555 | 0.347 | -0.123 | 0.215 |
| 22111 | 0.746 | 0.778 | 0.823 |
| 22112 | 0.692 | 0.720 | 0.786 |
| 22113 | 0.678 | 0.705 | 0.777 |
| 22114 | 0.654 | 0.492 | 0.645 |
| 22115 | 0.629 | 0.271 | 0.507 |
| 22121 | 0.678 | 0.678 | 0.772 |
| 22122 | 0.627 | 0.621 | 0.725 |
| 22123 | 0.614 | 0.606 | 0.713 |
| 22124 | 0.590 | 0.393 | 0.589 |
| 22125 | 0.565 | 0.172 | 0.461 |
| 22131 | 0.661 | 0.653 | 0.760 |
| 22132 | 0.611 | 0.596 | 0.710 |
| 22133 | 0.598 | 0.582 | 0.697 |
| 22134 | 0.574 | 0.369 | 0.575 |
| 22135 | 0.549 | 0.148 | 0.449 |
| 22141 | 0.616 | 0.440 | 0.624 |
| 22142 | 0.566 | 0.384 | 0.581 |
| 22143 | 0.553 | 0.369 | 0.570 |
| 22144 | 0.529 | 0.209 | 0.471 |
| 22145 | 0.504 | 0.043 | 0.368 |
| 22151 | 0.547 | 0.121 | 0.420 |
| 22152 | 0.497 | 0.064 | 0.387 |
| 22153 | 0.484 | 0.050 | 0.379 |
| 22154 | 0.460 | -0.031 | 0.314 |
| 22155 | 0.435 | -0.115 | 0.246 |
| 22211 | 0.707 | 0.747 | 0.799 |
| 22212 | 0.656 | 0.691 | 0.751 |
| 22213 | 0.643 | 0.676 | 0.739 |
| 22214 | 0.619 | 0.463 | 0.616 |
| 22215 | 0.594 | 0.242 | 0.487 |
| 22221 | 0.642 | 0.648 | 0.738 |
| 22222 | 0.592 | 0.592 | 0.678 |
| 22223 | 0.579 | 0.577 | 0.662 |
| 22224 | 0.555 | 0.364 | 0.547 |
| 22225 | 0.530 | 0.143 | 0.427 |
| 22231 | 0.626 | 0.624 | 0.723 |
| 22232 | 0.576 | 0.567 | 0.659 |
| 22233 | 0.563 | 0.553 | 0.643 |
| 22234 | 0.539 | 0.340 | 0.530 |
| 22235 | 0.514 | 0.119 | 0.412 |
| 22241 | 0.581 | 0.411 | 0.594 |
| 22242 | 0.531 | 0.355 | 0.537 |

| 22243 | 0.518 | 0.340 | 0.523 |
|-------|-------|--------|-------|
| 22244 | 0.494 | 0.180 | 0.432 |
| 22245 | 0.469 | 0.014 | 0.338 |
| 22251 | 0.512 | 0.092 | 0.400 |
| 22252 | 0.462 | 0.035 | 0.354 |
| 22253 | 0.449 | 0.021 | 0.342 |
| 22254 | 0.425 | -0.060 | 0.285 |
| 22255 | 0.400 | -0.144 | 0.226 |
| 22311 | 0.697 | 0.740 | 0.793 |
| 22312 | 0.647 | 0.683 | 0.743 |
| 22313 | 0.634 | 0.669 | 0.730 |
| 22314 | 0.610 | 0.456 | 0.609 |
| 22315 | 0.585 | 0.235 | 0.483 |
| 22321 | 0.633 | 0.641 | 0.729 |
| 22322 | 0.583 | 0.585 | 0.666 |
| 22323 | 0.570 | 0.570 | 0.649 |
| 22324 | 0.546 | 0.357 | 0.536 |
| 22325 | 0.521 | 0.136 | 0.419 |
| 22331 | 0.617 | 0.617 | 0.714 |
| 22332 | 0.567 | 0.560 | 0.647 |
| 22333 | 0.554 | 0.546 | 0.629 |
| 22334 | 0.530 | 0.333 | 0.518 |
| 22335 | 0.505 | 0.112 | 0.403 |
| 22341 | 0.572 | 0.404 | 0.587 |
| 22342 | 0.522 | 0.348 | 0.527 |
| 22343 | 0.509 | 0.333 | 0.511 |
| 22344 | 0.485 | 0.173 | 0.422 |
| 22345 | 0.460 | 0.007 | 0.330 |
| 22351 | 0.503 | 0.085 | 0.396 |
| 22352 | 0.453 | 0.028 | 0.346 |
| 22353 | 0.440 | 0.014 | 0.333 |
| 22354 | 0.416 | -0.067 | 0.278 |
| 22355 | 0.391 | -0.151 | 0.221 |
| 22411 | 0.668 | 0.632 | 0.724 |
| 22412 | 0.618 | 0.576 | 0.680 |
| 22413 | 0.605 | 0.561 | 0.668 |
| 22414 | 0.581 | 0.392 | 0.565 |
| 22415 | 0.556 | 0.216 | 0.459 |
| 22421 | 0.604 | 0.534 | 0.666 |
| 22422 | 0.554 | 0.477 | 0.608 |
| 22423 | 0.541 | 0.463 | 0.593 |
| 22424 | 0.517 | 0.293 | 0.498 |
| 22425 | 0.492 | 0.117 | 0.400 |
| 22431 | 0.588 | 0.509 | 0.652 |
| 22432 | 0.538 | 0.453 | 0.590 |
| 22433 | 0.525 | 0.438 | 0.574 |
| 22434 | 0.501 | 0.269 | 0.482 |
| 22435 | 0.476 | 0.093 | 0.386 |
| 22441 | 0.543 | 0.332 | 0.540 |

| 22442 | 0.493 | 0.276 | 0.485 |
|-------|-------|--------|-------|
| 22443 | 0.480 | 0.261 | 0.471 |
| 22444 | 0.456 | 0.127 | 0.394 |
| 22445 | 0.431 | -0.013 | 0.314 |
| 22451 | 0.474 | 0.066 | 0.372 |
| 22452 | 0.424 | 0.009 | 0.327 |
| 22453 | 0.411 | -0.005 | 0.316 |
| 22454 | 0.387 | -0.086 | 0.262 |
| 22455 | 0.362 | -0.170 | 0.207 |
| 22511 | 0.608 | 0.413 | 0.583 |
| 22512 | 0.558 | 0.356 | 0.550 |
| 22513 | 0.545 | 0.342 | 0.542 |
| 22514 | 0.521 | 0.261 | 0.477 |
| 22515 | 0.496 | 0.177 | 0.409 |
| 22521 | 0.544 | 0.314 | 0.537 |
| 22522 | 0.494 | 0.258 | 0.490 |
| 22523 | 0.481 | 0.243 | 0.478 |
| 22524 | 0.457 | 0.162 | 0.421 |
| 22525 | 0.432 | 0.078 | 0.362 |
| 22531 | 0.528 | 0.290 | 0.525 |
| 22532 | 0.478 | 0.233 | 0.475 |
| 22533 | 0.465 | 0.219 | 0.462 |
| 22534 | 0.441 | 0.138 | 0.407 |
| 22535 | 0.416 | 0.054 | 0.351 |
| 22541 | 0.483 | 0.185 | 0.444 |
| 22542 | 0.433 | 0.128 | 0.401 |
| 22543 | 0.420 | 0.114 | 0.390 |
| 22544 | 0.396 | 0.033 | 0.337 |
| 22545 | 0.371 | -0.051 | 0.282 |
| 22551 | 0.414 | 0.027 | 0.322 |
| 22552 | 0.364 | -0.030 | 0.289 |
| 22553 | 0.351 | -0.044 | 0.281 |
| 22554 | 0.327 | -0.125 | 0.230 |
| 22555 | 0.302 | -0.209 | 0.178 |
| 23111 | 0.732 | 0.758 | 0.811 |
| 23112 | 0.682 | 0.702 | 0.775 |
| 23113 | 0.669 | 0.687 | 0.766 |
| 23114 | 0.645 | 0.474 | 0.635 |
| 23115 | 0.620 | 0.253 | 0.500 |
| 23121 | 0.668 | 0.660 | 0.761 |
| 23122 | 0.618 | 0.603 | 0.712 |
| 23123 | 0.605 | 0.589 | 0.699 |
| 23124 | 0.581 | 0.376 | 0.577 |
| 23125 | 0.556 | 0.155 | 0.451 |
| 23131 | 0.652 | 0.635 | 0.749 |
| 23132 | 0.602 | 0.579 | 0.696 |
| 23133 | 0.589 | 0.564 | 0.683 |
| 23134 | 0.565 | 0.351 | 0.563 |
| 23135 | 0.540 | 0.130 | 0.439 |

| 23141 | 0.607 | 0.423 | 0.615 |
|-------|-------|--------|-------|
| 23142 | 0.557 | 0.366 | 0.569 |
| 23143 | 0.544 | 0.352 | 0.557 |
| 23144 | 0.520 | 0.192 | 0.460 |
| 23145 | 0.495 | 0.025 | 0.359 |
| 23151 | 0.538 | 0.103 | 0.413 |
| 23152 | 0.488 | 0.047 | 0.377 |
| 23153 | 0.475 | 0.032 | 0.368 |
| 23154 | 0.451 | -0.049 | 0.305 |
| 23155 | 0.426 | -0.133 | 0.239 |
| 23211 | 0.697 | 0.729 | 0.788 |
| 23212 | 0.647 | 0.673 | 0.738 |
| 23213 | 0.634 | 0.658 | 0.726 |
| 23214 | 0.610 | 0.445 | 0.604 |
| 23215 | 0.585 | 0.224 | 0.477 |
| 23221 | 0.633 | 0.631 | 0.725 |
| 23222 | 0.583 | 0.575 | 0.662 |
| 23223 | 0.570 | 0.560 | 0.645 |
| 23224 | 0.546 | 0.347 | 0.532 |
| 23225 | 0.521 | 0.126 | 0.414 |
| 23231 | 0.617 | 0.606 | 0.709 |
| 23232 | 0.567 | 0.550 | 0.643 |
| 23233 | 0.554 | 0.535 | 0.626 |
| 23234 | 0.530 | 0.322 | 0.514 |
| 23235 | 0.505 | 0.101 | 0.399 |
| 23241 | 0.572 | 0.394 | 0.582 |
| 23242 | 0.522 | 0.338 | 0.522 |
| 23243 | 0.509 | 0.323 | 0.507 |
| 23244 | 0.484 | 0.163 | 0.418 |
| 23245 | 0.460 | -0.004 | 0.326 |
| 23251 | 0.503 | 0.074 | 0.390 |
| 23252 | 0.453 | 0.018 | 0.341 |
| 23253 | 0.440 | 0.003 | 0.328 |
| 23254 | 0.416 | -0.078 | 0.273 |
| 23255 | 0.391 | -0.162 | 0.216 |
| 23311 | 0.688 | 0.722 | 0.782 |
| 23312 | 0.638 | 0.666 | 0.729 |
| 23313 | 0.625 | 0.651 | 0.716 |
| 23314 | 0.601 | 0.438 | 0.596 |
| 23315 | 0.576 | 0.217 | 0.472 |
| 23321 | 0.624 | 0.624 | 0.716 |
| 23322 | 0.574 | 0.567 | 0.649 |
| 23323 | 0.561 | 0.553 | 0.632 |
| 23324 | 0.537 | 0.340 | 0.521 |
| 23325 | 0.512 | 0.119 | 0.405 |
| 23331 | 0.608 | 0.599 | 0.700 |
| 23332 | 0.558 | 0.543 | 0.630 |
| 23333 | 0.545 | 0.528 | 0.611 |
| 23334 | 0.521 | 0.315 | 0.502 |

| 23335 | 0.496 | 0.094 | 0.389 |
|-------|-------|--------|-------|
| 23341 | 0.563 | 0.387 | 0.574 |
| 23342 | 0.513 | 0.330 | 0.511 |
| 23343 | 0.500 | 0.316 | 0.494 |
| 23344 | 0.476 | 0.156 | 0.408 |
| 23345 | 0.451 | -0.011 | 0.318 |
| 23351 | 0.494 | 0.067 | 0.385 |
| 23352 | 0.444 | 0.011 | 0.332 |
| 23353 | 0.431 | -0.004 | 0.319 |
| 23354 | 0.407 | -0.085 | 0.266 |
| 23355 | 0.382 | -0.169 | 0.211 |
| 23411 | 0.659 | 0.615 | 0.714 |
| 23412 | 0.609 | 0.559 | 0.667 |
| 23413 | 0.596 | 0.544 | 0.655 |
| 23414 | 0.572 | 0.374 | 0.554 |
| 23415 | 0.547 | 0.198 | 0.449 |
| 23421 | 0.595 | 0.516 | 0.654 |
| 23422 | 0.545 | 0.460 | 0.593 |
| 23423 | 0.532 | 0.445 | 0.577 |
| 23424 | 0.508 | 0.276 | 0.484 |
| 23425 | 0.483 | 0.100 | 0.388 |
| 23431 | 0.579 | 0.492 | 0.639 |
| 23432 | 0.529 | 0.436 | 0.574 |
| 23433 | 0.516 | 0.421 | 0.558 |
| 23434 | 0.492 | 0.251 | 0.467 |
| 23435 | 0.467 | 0.075 | 0.373 |
| 23441 | 0.534 | 0.315 | 0.528 |
| 23442 | 0.484 | 0.258 | 0.471 |
| 23443 | 0.471 | 0.244 | 0.456 |
| 23444 | 0.447 | 0.109 | 0.381 |
| 23445 | 0.422 | -0.030 | 0.303 |
| 23451 | 0.465 | 0.048 | 0.362 |
| 23452 | 0.415 | -0.008 | 0.315 |
| 23453 | 0.402 | -0.023 | 0.303 |
| 23454 | 0.378 | -0.104 | 0.251 |
| 23455 | 0.353 | -0.188 | 0.197 |
| 23511 | 0.599 | 0.395 | 0.576 |
| 23512 | 0.549 | 0.339 | 0.540 |
| 23513 | 0.536 | 0.324 | 0.531 |
| 23514 | 0.512 | 0.243 | 0.468 |
| 23515 | 0.487 | 0.159 | 0.402 |
| 23521 | 0.535 | 0.297 | 0.527 |
| 23522 | 0.485 | 0.240 | 0.477 |
| 23523 | 0.472 | 0.226 | 0.464 |
| 23524 | 0.448 | 0.145 | 0.409 |
| 23525 | 0.423 | 0.061 | 0.352 |
| 23531 | 0.519 | 0.272 | 0.515 |
| 23532 | 0.469 | 0.216 | 0.462 |
| 23533 | 0.456 | 0.201 | 0.448 |

| 23534 | 0.432 | 0.120 | 0.395 |
|-------|-------|--------|-------|
| 23535 | 0.407 | 0.036 | 0.340 |
| 23541 | 0.474 | 0.167 | 0.435 |
| 23542 | 0.424 | 0.111 | 0.389 |
| 23543 | 0.411 | 0.096 | 0.377 |
| 23544 | 0.387 | 0.015 | 0.325 |
| 23545 | 0.362 | -0.069 | 0.272 |
| 23551 | 0.405 | 0.009 | 0.315 |
| 23552 | 0.355 | -0.047 | 0.279 |
| 23553 | 0.342 | -0.062 | 0.270 |
| 23554 | 0.318 | -0.143 | 0.221 |
| 23555 | 0.293 | -0.227 | 0.170 |
| 24111 | 0.721 | 0.666 | 0.741 |
| 24112 | 0.671 | 0.610 | 0.709 |
| 24113 | 0.658 | 0.595 | 0.701 |
| 24114 | 0.634 | 0.414 | 0.584 |
| 24115 | 0.609 | 0.227 | 0.463 |
| 24121 | 0.657 | 0.568 | 0.695 |
| 24122 | 0.607 | 0.511 | 0.650 |
| 24123 | 0.594 | 0.497 | 0.638 |
| 24124 | 0.570 | 0.316 | 0.530 |
| 24125 | 0.545 | 0.128 | 0.418 |
| 24131 | 0.641 | 0.543 | 0.684 |
| 24132 | 0.591 | 0.487 | 0.636 |
| 24133 | 0.578 | 0.472 | 0.623 |
| 24134 | 0.554 | 0.291 | 0.517 |
| 24135 | 0.529 | 0.104 | 0.407 |
| 24141 | 0.595 | 0.357 | 0.561 |
| 24142 | 0.545 | 0.300 | 0.519 |
| 24143 | 0.532 | 0.286 | 0.508 |
| 24144 | 0.508 | 0.145 | 0.420 |
| 24145 | 0.483 | -0.002 | 0.328 |
| 24151 | 0.527 | 0.077 | 0.376 |
| 24152 | 0.477 | 0.020 | 0.344 |
| 24153 | 0.464 | 0.006 | 0.336 |
| 24154 | 0.440 | -0.076 | 0.274 |
| 24155 | 0.415 | -0.160 | 0.210 |
| 24211 | 0.685 | 0.637 | 0.722 |
| 24212 | 0.635 | 0.581 | 0.677 |
| 24213 | 0.622 | 0.566 | 0.665 |
| 24214 | 0.598 | 0.385 | 0.557 |
| 24215 | 0.573 | 0.198 | 0.444 |
| 24221 | 0.621 | 0.539 | 0.663 |
| 24222 | 0.571 | 0.482 | 0.604 |
| 24223 | 0.558 | 0.468 | 0.589 |
| 24224 | 0.534 | 0.287 | 0.489 |
| 24225 | 0.509 | 0.099 | 0.385 |
| 24231 | 0.605 | 0.514 | 0.648 |
| 24232 | 0.555 | 0.458 | 0.586 |

| 24233 | 0.542 | 0.443 | 0.570 |
|-------|-------|--------|-------|
| 24234 | 0.518 | 0.262 | 0.472 |
| 24235 | 0.493 | 0.075 | 0.371 |
| 24241 | 0.560 | 0.328 | 0.532 |
| 24242 | 0.510 | 0.272 | 0.477 |
| 24243 | 0.497 | 0.257 | 0.462 |
| 24244 | 0.473 | 0.116 | 0.382 |
| 24245 | 0.448 | -0.030 | 0.299 |
| 24251 | 0.491 | 0.048 | 0.357 |
| 24252 | 0.441 | -0.009 | 0.312 |
| 24253 | 0.428 | -0.023 | 0.301 |
| 24254 | 0.404 | -0.104 | 0.247 |
| 24255 | 0.379 | -0.188 | 0.191 |
| 24311 | 0.677 | 0.630 | 0.717 |
| 24312 | 0.627 | 0.574 | 0.669 |
| 24313 | 0.614 | 0.559 | 0.656 |
| 24314 | 0.590 | 0.378 | 0.550 |
| 24315 | 0.565 | 0.191 | 0.440 |
| 24321 | 0.613 | 0.532 | 0.655 |
| 24322 | 0.563 | 0.475 | 0.593 |
| 24323 | 0.550 | 0.461 | 0.577 |
| 24324 | 0.526 | 0.280 | 0.479 |
| 24325 | 0.501 | 0.092 | 0.377 |
| 24331 | 0.597 | 0.507 | 0.640 |
| 24332 | 0.547 | 0.451 | 0.574 |
| 24333 | 0.534 | 0.436 | 0.557 |
| 24334 | 0.510 | 0.255 | 0.461 |
| 24335 | 0.485 | 0.068 | 0.362 |
| 24341 | 0.551 | 0.321 | 0.525 |
| 24342 | 0.501 | 0.264 | 0.466 |
| 24343 | 0.488 | 0.250 | 0.451 |
| 24344 | 0.464 | 0.109 | 0.373 |
| 24345 | 0.439 | -0.038 | 0.292 |
| 24351 | 0.483 | 0.041 | 0.353 |
| 24352 | 0.433 | -0.016 | 0.305 |
| 24353 | 0.420 | -0.031 | 0.292 |
| 24354 | 0.396 | -0.112 | 0.240 |
| 24355 | 0.371 | -0.196 | 0.186 |
| 24411 | 0.647 | 0.544 | 0.659 |
| 24412 | 0.597 | 0.488 | 0.616 |
| 24413 | 0.584 | 0.473 | 0.604 |
| 24414 | 0.560 | 0.325 | 0.513 |
| 24415 | 0.535 | 0.172 | 0.418 |
| 24421 | 0.583 | 0.446 | 0.602 |
| 24422 | 0.533 | 0.389 | 0.545 |
| 24423 | 0.520 | 0.375 | 0.531 |
| 24424 | 0.496 | 0.227 | 0.447 |
| 24425 | 0.471 | 0.073 | 0.361 |
| 24431 | 0.567 | 0.421 | 0.588 |

| 24432 | 0.517 | 0.365 | 0.528 |
|-------|-------|--------|-------|
| 24433 | 0.504 | 0.350 | 0.512 |
| 24434 | 0.480 | 0.202 | 0.431 |
| 24435 | 0.455 | 0.049 | 0.347 |
| 24441 | 0.522 | 0.262 | 0.485 |
| 24442 | 0.472 | 0.205 | 0.432 |
| 24443 | 0.459 | 0.191 | 0.418 |
| 24444 | 0.435 | 0.069 | 0.349 |
| 24445 | 0.410 | -0.057 | 0.277 |
| 24451 | 0.453 | 0.022 | 0.331 |
| 24452 | 0.403 | -0.035 | 0.288 |
| 24453 | 0.390 | -0.050 | 0.277 |
| 24454 | 0.366 | -0.131 | 0.226 |
| 24455 | 0.341 | -0.215 | 0.173 |
| 24511 | 0.588 | 0.369 | 0.539 |
| 24512 | 0.538 | 0.312 | 0.507 |
| 24513 | 0.525 | 0.298 | 0.499 |
| 24514 | 0.501 | 0.217 | 0.437 |
| 24515 | 0.476 | 0.133 | 0.372 |
| 24521 | 0.524 | 0.270 | 0.494 |
| 24522 | 0.474 | 0.214 | 0.448 |
| 24523 | 0.461 | 0.199 | 0.437 |
| 24524 | 0.437 | 0.118 | 0.383 |
| 24525 | 0.412 | 0.034 | 0.327 |
| 24531 | 0.508 | 0.246 | 0.483 |
| 24532 | 0.458 | 0.189 | 0.434 |
| 24533 | 0.445 | 0.175 | 0.421 |
| 24534 | 0.421 | 0.094 | 0.369 |
| 24535 | 0.396 | 0.010 | 0.315 |
| 24541 | 0.462 | 0.140 | 0.404 |
| 24542 | 0.412 | 0.084 | 0.362 |
| 24543 | 0.399 | 0.069 | 0.351 |
| 24544 | 0.375 | -0.012 | 0.301 |
| 24545 | 0.350 | -0.096 | 0.248 |
| 24551 | 0.394 | -0.018 | 0.286 |
| 24552 | 0.344 | -0.074 | 0.254 |
| 24553 | 0.331 | -0.089 | 0.245 |
| 24554 | 0.307 | -0.170 | 0.197 |
| 24555 | 0.282 | -0.254 | 0.148 |
| 25111 | 0.684 | 0.379 | 0.523 |
| 25112 | 0.634 | 0.323 | 0.503 |
| 25113 | 0.621 | 0.308 | 0.498 |
| 25114 | 0.597 | 0.227 | 0.425 |
| 25115 | 0.572 | 0.143 | 0.349 |
| 25121 | 0.620 | 0.281 | 0.490 |
| 25122 | 0.570 | 0.224 | 0.457 |
| 25123 | 0.557 | 0.210 | 0.449 |
| 25124 | 0.533 | 0.129 | 0.383 |
| 25125 | 0.508 | 0.045 | 0.315 |

| 25131 | 0.604 | 0.256 | 0.481 |
|-------|-------|--------|-------|
| 25132 | 0.554 | 0.200 | 0.446 |
| 25133 | 0.541 | 0.185 | 0.437 |
| 25134 | 0.517 | 0.104 | 0.373 |
| 25135 | 0.492 | 0.020 | 0.307 |
| 25141 | 0.559 | 0.151 | 0.394 |
| 25142 | 0.509 | 0.095 | 0.365 |
| 25143 | 0.496 | 0.080 | 0.357 |
| 25144 | 0.472 | -0.001 | 0.295 |
| 25145 | 0.447 | -0.085 | 0.232 |
| 25151 | 0.490 | -0.007 | 0.262 |
| 25152 | 0.440 | -0.063 | 0.242 |
| 25153 | 0.427 | -0.078 | 0.237 |
| 25154 | 0.403 | -0.159 | 0.179 |
| 25155 | 0.378 | -0.243 | 0.118 |
| 25211 | 0.649 | 0.350 | 0.517 |
| 25212 | 0.599 | 0.294 | 0.484 |
| 25213 | 0.586 | 0.279 | 0.475 |
| 25214 | 0.562 | 0.198 | 0.410 |
| 25215 | 0.537 | 0.114 | 0.342 |
| 25221 | 0.585 | 0.252 | 0.470 |
| 25222 | 0.535 | 0.196 | 0.424 |
| 25223 | 0.522 | 0.181 | 0.412 |
| 25224 | 0.498 | 0.100 | 0.355 |
| 25225 | 0.473 | 0.016 | 0.296 |
| 25231 | 0.569 | 0.227 | 0.459 |
| 25232 | 0.519 | 0.171 | 0.409 |
| 25233 | 0.506 | 0.156 | 0.397 |
| 25234 | 0.482 | 0.075 | 0.342 |
| 25235 | 0.457 | -0.009 | 0.284 |
| 25241 | 0.524 | 0.122 | 0.377 |
| 25242 | 0.474 | 0.066 | 0.335 |
| 25243 | 0.461 | 0.051 | 0.324 |
| 25244 | 0.436 | -0.030 | 0.270 |
| 25245 | 0.412 | -0.114 | 0.215 |
| 25251 | 0.455 | -0.036 | 0.255 |
| 25252 | 0.405 | -0.092 | 0.223 |
| 25253 | 0.392 | -0.107 | 0.214 |
| 25254 | 0.368 | -0.188 | 0.164 |
| 25255 | 0.343 | -0.272 | 0.111 |
| 25311 | 0.640 | 0.343 | 0.515 |
| 25312 | 0.590 | 0.287 | 0.479 |
| 25313 | 0.577 | 0.272 | 0.470 |
| 25314 | 0.553 | 0.191 | 0.406 |
| 25315 | 0.528 | 0.107 | 0.340 |
| 25321 | 0.576 | 0.245 | 0.465 |
| 25322 | 0.526 | 0.188 | 0.416 |
| 25323 | 0.513 | 0.174 | 0.403 |
| 25324 | 0.489 | 0.093 | 0.348 |

| 25325 | 0.464 | 0.009 | 0.291 |
|-------|-------|--------|-------|
| 25331 | 0.560 | 0.220 | 0.453 |
| 25332 | 0.510 | 0.164 | 0.400 |
| 25333 | 0.497 | 0.149 | 0.387 |
| 25334 | 0.473 | 0.068 | 0.334 |
| 25335 | 0.448 | -0.016 | 0.279 |
| 25341 | 0.515 | 0.115 | 0.373 |
| 25342 | 0.465 | 0.059 | 0.328 |
| 25343 | 0.452 | 0.044 | 0.316 |
| 25344 | 0.428 | -0.037 | 0.264 |
| 25345 | 0.403 | -0.121 | 0.211 |
| 25351 | 0.446 | -0.043 | 0.253 |
| 25352 | 0.396 | -0.099 | 0.218 |
| 25353 | 0.383 | -0.114 | 0.209 |
| 25354 | 0.359 | -0.195 | 0.160 |
| 25355 | 0.334 | -0.279 | 0.109 |
| 25411 | 0.611 | 0.324 | 0.486 |
| 25412 | 0.561 | 0.268 | 0.455 |
| 25413 | 0.548 | 0.253 | 0.447 |
| 25414 | 0.524 | 0.172 | 0.385 |
| 25415 | 0.499 | 0.088 | 0.320 |
| 25421 | 0.547 | 0.226 | 0.441 |
| 25422 | 0.497 | 0.169 | 0.397 |
| 25423 | 0.484 | 0.155 | 0.386 |
| 25424 | 0.460 | 0.074 | 0.332 |
| 25425 | 0.435 | -0.010 | 0.276 |
| 25431 | 0.531 | 0.201 | 0.430 |
| 25432 | 0.481 | 0.145 | 0.383 |
| 25433 | 0.468 | 0.130 | 0.371 |
| 25434 | 0.444 | 0.049 | 0.319 |
| 25435 | 0.419 | -0.035 | 0.265 |
| 25441 | 0.486 | 0.096 | 0.352 |
| 25442 | 0.436 | 0.040 | 0.311 |
| 25443 | 0.423 | 0.025 | 0.301 |
| 25444 | 0.399 | -0.056 | 0.251 |
| 25445 | 0.374 | -0.140 | 0.199 |
| 25451 | 0.417 | -0.062 | 0.234 |
| 25452 | 0.367 | -0.118 | 0.203 |
| 25453 | 0.354 | -0.133 | 0.195 |
| 25454 | 0.330 | -0.214 | 0.148 |
| 25455 | 0.305 | -0.298 | 0.099 |
| 25511 | 0.551 | 0.285 | 0.425 |
| 25512 | 0.501 | 0.229 | 0.405 |
| 25513 | 0.488 | 0.214 | 0.400 |
| 25514 | 0.464 | 0.133 | 0.341 |
| 25515 | 0.439 | 0.049 | 0.280 |
| 25521 | 0.487 | 0.187 | 0.391 |
| 25522 | 0.437 | 0.130 | 0.359 |
| 25523 | 0.424 | 0.116 | 0.350 |

| 25524 | 0.400 | 0.035 | 0.299 |
|-------|-------|--------|-------|
| 25525 | 0.375 | -0.049 | 0.247 |
| 25531 | 0.471 | 0.162 | 0.383 |
| 25532 | 0.421 | 0.106 | 0.347 |
| 25533 | 0.408 | 0.091 | 0.338 |
| 25534 | 0.384 | 0.010 | 0.289 |
| 25535 | 0.359 | -0.074 | 0.238 |
| 25541 | 0.426 | 0.057 | 0.308 |
| 25542 | 0.376 | 0.001 | 0.278 |
| 25543 | 0.363 | -0.014 | 0.270 |
| 25544 | 0.339 | -0.095 | 0.223 |
| 25545 | 0.314 | -0.179 | 0.174 |
| 25551 | 0.357 | -0.101 | 0.194 |
| 25552 | 0.307 | -0.157 | 0.173 |
| 25553 | 0.294 | -0.172 | 0.168 |
| 25554 | 0.270 | -0.253 | 0.124 |
| 25555 | 0.245 | -0.337 | 0.078 |
| 31111 | 0.773 | 0.850 | 0.854 |
| 31112 | 0.723 | 0.794 | 0.833 |
| 31113 | 0.710 | 0.779 | 0.827 |
| 31114 | 0.686 | 0.566 | 0.688 |
| 31115 | 0.661 | 0.345 | 0.543 |
| 31121 | 0.709 | 0.752 | 0.819 |
| 31122 | 0.659 | 0.695 | 0.783 |
| 31123 | 0.646 | 0.681 | 0.774 |
| 31124 | 0.622 | 0.468 | 0.643 |
| 31125 | 0.597 | 0.247 | 0.508 |
| 31131 | 0.693 | 0.727 | 0.810 |
| 31132 | 0.643 | 0.671 | 0.771 |
| 31133 | 0.630 | 0.656 | 0.761 |
| 31134 | 0.606 | 0.443 | 0.632 |
| 31135 | 0.581 | 0.222 | 0.499 |
| 31141 | 0.648 | 0.515 | 0.669 |
| 31142 | 0.598 | 0.458 | 0.637 |
| 31143 | 0.585 | 0.444 | 0.628 |
| 31144 | 0.560 | 0.283 | 0.522 |
| 31145 | 0.536 | 0.117 | 0.412 |
| 31151 | 0.579 | 0.195 | 0.456 |
| 31152 | 0.529 | 0.139 | 0.435 |
| 31153 | 0.516 | 0.124 | 0.429 |
| 31154 | 0.492 | 0.043 | 0.357 |
| 31155 | 0.467 | -0.041 | 0.282 |
| 31211 | 0.738 | 0.821 | 0.845 |
| 31212 | 0.688 | 0.765 | 0.810 |
| 31213 | 0.675 | 0.750 | 0.801 |
| 31214 | 0.651 | 0.537 | 0.670 |
| 31215 | 0.626 | 0.316 | 0.535 |
| 31221 | 0.674 | 0.723 | 0.796 |
| 31222 | 0.624 | 0.666 | 0.748 |

| 31223 | 0.611 | 0.652 | 0.735 |
|-------|-------|--------|-------|
| 31224 | 0.587 | 0.439 | 0.613 |
| 31225 | 0.562 | 0.218 | 0.486 |
| 31231 | 0.658 | 0.698 | 0.784 |
| 31232 | 0.608 | 0.642 | 0.732 |
| 31233 | 0.595 | 0.627 | 0.719 |
| 31234 | 0.571 | 0.414 | 0.598 |
| 31235 | 0.546 | 0.193 | 0.473 |
| 31241 | 0.612 | 0.486 | 0.650 |
| 31242 | 0.562 | 0.429 | 0.604 |
| 31243 | 0.549 | 0.415 | 0.593 |
| 31244 | 0.525 | 0.254 | 0.495 |
| 31245 | 0.500 | 0.088 | 0.393 |
| 31251 | 0.544 | 0.166 | 0.448 |
| 31252 | 0.494 | 0.110 | 0.413 |
| 31253 | 0.481 | 0.095 | 0.403 |
| 31254 | 0.457 | 0.014 | 0.340 |
| 31255 | 0.432 | -0.070 | 0.273 |
| 31311 | 0.729 | 0.814 | 0.843 |
| 31312 | 0.679 | 0.758 | 0.804 |
| 31313 | 0.666 | 0.743 | 0.794 |
| 31314 | 0.642 | 0.530 | 0.666 |
| 31315 | 0.617 | 0.309 | 0.533 |
| 31321 | 0.665 | 0.716 | 0.791 |
| 31322 | 0.615 | 0.659 | 0.739 |
| 31323 | 0.602 | 0.645 | 0.725 |
| 31324 | 0.578 | 0.432 | 0.605 |
| 31325 | 0.553 | 0.211 | 0.480 |
| 31331 | 0.649 | 0.691 | 0.778 |
| 31332 | 0.599 | 0.635 | 0.723 |
| 31333 | 0.586 | 0.620 | 0.708 |
| 31334 | 0.562 | 0.407 | 0.590 |
| 31335 | 0.537 | 0.186 | 0.467 |
| 31341 | 0.604 | 0.479 | 0.645 |
| 31342 | 0.554 | 0.422 | 0.597 |
| 31343 | 0.541 | 0.408 | 0.584 |
| 31344 | 0.516 | 0.247 | 0.488 |
| 31345 | 0.492 | 0.081 | 0.389 |
| 31351 | 0.535 | 0.159 | 0.446 |
| 31352 | 0.485 | 0.103 | 0.407 |
| 31353 | 0.472 | 0.088 | 0.397 |
| 31354 | 0.448 | 0.007 | 0.335 |
| 31355 | 0.423 | -0.077 | 0.271 |
| 31411 | 0.700 | 0.707 | 0.769 |
| 31412 | 0.650 | 0.650 | 0.736 |
| 31413 | 0.637 | 0.636 | 0.728 |
| 31414 | 0.613 | 0.466 | 0.618 |
| 31415 | 0.588 | 0.290 | 0.504 |
| 31421 | 0.636 | 0.608 | 0.723 |

| 31422 | 0.586 | 0.552 | 0.676 |
|----------------|----------------|----------------|----------------|
| 31423 | 0.573 | 0.537 | 0.664 |
| 31424 | 0.549 | 0.368 | 0.563 |
| 31425 | 0.524 | 0.191 | 0.457 |
| 31431 | 0.620 | 0.584 | 0.711 |
| 31432 | 0.570 | 0.527 | 0.662 |
| 31433 | 0.557 | 0.513 | 0.649 |
| 31434 | 0.533 | 0.343 | 0.549 |
| 31435 | 0.508 | 0.167 | 0.445 |
| 31441 | 0.574 | 0.406 | 0.594 |
| 31442 | 0.524 | 0.350 | 0.551 |
| 31443 | 0.511 | 0.335 | 0.539 |
| 31444 | 0.487 | 0.201 | 0.455 |
| 31445 | 0.462 | 0.062 | 0.368 |
| 31451 | 0.506 | 0.140 | 0.417 |
| 31452 | 0.456 | 0.084 | 0.384 |
| 31453 | 0.443 | 0.069 | 0.375 |
| 31454 | 0.419 | -0.012 | 0.315 |
| 31455 | 0.394 | -0.096 | 0.252 |
| 31511 | 0.640 | 0.487 | 0.619 |
| 31512 | 0.590 | 0.431 | 0.598 |
| 31513 | 0.577 | 0.416 | 0.592 |
| 31514 | 0.553 | 0.335 | 0.520 |
| 31515 | 0.528 | 0.251 | 0.445 |
| 31521 | 0.576 | 0.389 | 0.584 |
| 31522 | 0.526 | 0.332 | 0.549 |
| 31523 | 0.513 | 0.318 | 0.540 |
| 31524 | 0.489 | 0.237 | 0.476 |
| 31525 | 0.464 | 0.153 | 0.410 |
| 31531 | 0.560 | 0.364 | 0.575 |
| 31532 | 0.510 | 0.308 | 0.537 |
| 31533 | 0.497 | 0.293 | 0.527 |
| 31534 | 0.473 | 0.212 | 0.465 |
| 31535 | 0.448 | 0.128 | 0.401 |
| 31541 | 0.515 | 0.259 | 0.488 |
| 31542 | 0.465 | 0.203 | 0.457 |
| 31543 | 0.452 | 0.188 | 0.449 |
| 31544 | 0.427 | 0.107 | 0.389 |
| 31545 | 0.403 | 0.023 | 0.326 |
| 31551 | 0.446 | 0.101 | 0.358 |
| 31552 | 0.396 | 0.045 | 0.337 |
| 31553 | 0.383 | 0.030 | 0.331 |
| 31554 | 0.359 | -0.051 | 0.274 |
| 31555 | 0.334 | -0.135 | 0.214 |
| 32111 | 0.728 | 0.763 | 0.816 |
| 32112 | 0.678 | 0.707 | 0.780 |
| 32113 | 0.665 | 0.692 | 0.770 |
| 32114<br>32115 | 0.641<br>0.616 | 0.479<br>0.258 | 0.640<br>0.505 |
| 32115 | 0.010 | 0.258 | 0.505 |

| 32121 | 0.664 | 0.665 | 0.766 |
|-------|-------|--------|-------|
| 32122 | 0.614 | 0.609 | 0.716 |
| 32123 | 0.601 | 0.594 | 0.704 |
| 32124 | 0.577 | 0.381 | 0.582 |
| 32125 | 0.552 | 0.160 | 0.455 |
| 32131 | 0.648 | 0.640 | 0.753 |
| 32132 | 0.598 | 0.584 | 0.701 |
| 32133 | 0.585 | 0.569 | 0.687 |
| 32134 | 0.561 | 0.356 | 0.567 |
| 32135 | 0.536 | 0.135 | 0.443 |
| 32141 | 0.603 | 0.428 | 0.619 |
| 32142 | 0.553 | 0.372 | 0.573 |
| 32143 | 0.540 | 0.357 | 0.561 |
| 32144 | 0.516 | 0.197 | 0.464 |
| 32145 | 0.491 | 0.030 | 0.364 |
| 32151 | 0.534 | 0.108 | 0.418 |
| 32152 | 0.484 | 0.052 | 0.382 |
| 32153 | 0.471 | 0.037 | 0.372 |
| 32154 | 0.447 | -0.044 | 0.309 |
| 32155 | 0.422 | -0.128 | 0.244 |
| 32211 | 0.693 | 0.735 | 0.792 |
| 32212 | 0.643 | 0.678 | 0.743 |
| 32213 | 0.630 | 0.664 | 0.730 |
| 32214 | 0.606 | 0.451 | 0.608 |
| 32215 | 0.581 | 0.230 | 0.482 |
| 32221 | 0.629 | 0.636 | 0.729 |
| 32222 | 0.579 | 0.580 | 0.666 |
| 32223 | 0.566 | 0.565 | 0.650 |
| 32224 | 0.542 | 0.352 | 0.536 |
| 32225 | 0.517 | 0.131 | 0.419 |
| 32231 | 0.613 | 0.612 | 0.714 |
| 32232 | 0.563 | 0.555 | 0.647 |
| 32233 | 0.550 | 0.541 | 0.630 |
| 32234 | 0.526 | 0.328 | 0.518 |
| 32235 | 0.501 | 0.107 | 0.403 |
| 32241 | 0.567 | 0.399 | 0.586 |
| 32242 | 0.517 | 0.343 | 0.527 |
| 32243 | 0.504 | 0.328 | 0.511 |
| 32244 | 0.480 | 0.168 | 0.422 |
| 32245 | 0.455 | 0.002 | 0.330 |
| 32251 | 0.499 | 0.080 | 0.395 |
| 32252 | 0.449 | 0.023 | 0.346 |
| 32253 | 0.436 | 0.009 | 0.333 |
| 32254 | 0.412 | -0.072 | 0.278 |
| 32255 | 0.387 | -0.157 | 0.221 |
| 32311 | 0.684 | 0.727 | 0.786 |
| 32312 | 0.634 | 0.671 | 0.734 |
| 32313 | 0.621 | 0.656 | 0.720 |
| 32314 | 0.597 | 0.443 | 0.600 |

| 32315 | 0.572 | 0.222 | 0.476 |
|-------|-------|--------|-------|
| 32321 | 0.620 | 0.629 | 0.720 |
| 32322 | 0.570 | 0.573 | 0.654 |
| 32323 | 0.557 | 0.558 | 0.636 |
| 32324 | 0.533 | 0.345 | 0.525 |
| 32325 | 0.508 | 0.124 | 0.410 |
| 32331 | 0.604 | 0.604 | 0.704 |
| 32332 | 0.554 | 0.548 | 0.634 |
| 32333 | 0.541 | 0.533 | 0.616 |
| 32334 | 0.517 | 0.320 | 0.506 |
| 32335 | 0.492 | 0.099 | 0.393 |
| 32341 | 0.559 | 0.392 | 0.578 |
| 32342 | 0.509 | 0.336 | 0.515 |
| 32343 | 0.496 | 0.321 | 0.499 |
| 32344 | 0.472 | 0.161 | 0.412 |
| 32345 | 0.447 | -0.006 | 0.322 |
| 32351 | 0.490 | 0.072 | 0.389 |
| 32352 | 0.440 | 0.016 | 0.337 |
| 32353 | 0.427 | 0.001 | 0.323 |
| 32354 | 0.403 | -0.080 | 0.270 |
| 32355 | 0.378 | -0.164 | 0.215 |
| 32411 | 0.655 | 0.620 | 0.719 |
| 32412 | 0.605 | 0.564 | 0.672 |
| 32413 | 0.592 | 0.549 | 0.659 |
| 32414 | 0.568 | 0.379 | 0.558 |
| 32415 | 0.543 | 0.203 | 0.454 |
| 32421 | 0.591 | 0.522 | 0.658 |
| 32422 | 0.541 | 0.465 | 0.597 |
| 32423 | 0.528 | 0.451 | 0.581 |
| 32424 | 0.504 | 0.281 | 0.489 |
| 32425 | 0.479 | 0.105 | 0.392 |
| 32431 | 0.575 | 0.497 | 0.643 |
| 32432 | 0.525 | 0.441 | 0.579 |
| 32433 | 0.512 | 0.426 | 0.562 |
| 32434 | 0.488 | 0.256 | 0.471 |
| 32435 | 0.463 | 0.080 | 0.377 |
| 32441 | 0.529 | 0.320 | 0.533 |
| 32442 | 0.479 | 0.263 | 0.475 |
| 32443 | 0.466 | 0.249 | 0.460 |
| 32444 | 0.442 | 0.115 | 0.385 |
| 32445 | 0.417 | -0.025 | 0.307 |
| 32451 | 0.461 | 0.053 | 0.367 |
| 32452 | 0.411 | -0.003 | 0.319 |
| 32453 | 0.398 | -0.018 | 0.307 |
| 32454 | 0.374 | -0.099 | 0.255 |
| 32455 | 0.349 | -0.183 | 0.202 |
| 32511 | 0.595 | 0.400 | 0.581 |
| 32512 | 0.545 | 0.344 | 0.545 |
| 32513 | 0.532 | 0.329 | 0.535 |

| 32514 | 0.508 | 0.248 | 0.472 |
|----------------|----------------|-----------------|----------------|
| 32515 | 0.483 | 0.164 | 0.407 |
| 32521 | 0.531 | 0.302 | 0.531 |
| 32522 | 0.481 | 0.246 | 0.482 |
| 32523 | 0.468 | 0.231 | 0.469 |
| 32524 | 0.444 | 0.150 | 0.414 |
| 32525 | 0.419 | 0.066 | 0.357 |
| 32531 | 0.515 | 0.277 | 0.519 |
| 32532 | 0.465 | 0.221 | 0.466 |
| 32533 | 0.452 | 0.206 | 0.452 |
| 32534 | 0.428 | 0.125 | 0.399 |
| 32535 | 0.403 | 0.041 | 0.344 |
| 32541 | 0.470 | 0.172 | 0.440 |
| 32542 | 0.420 | 0.116 | 0.393 |
| 32543 | 0.407 | 0.101 | 0.381 |
| 32544 | 0.383 | 0.020 | 0.330 |
| 32545 | 0.358 | -0.064 | 0.277 |
| 32551 | 0.401 | 0.014 | 0.320 |
| 32552 | 0.351 | -0.042 | 0.284 |
| 32553 | 0.338 | -0.057 | 0.274 |
| 32554 | 0.314 | -0.138 | 0.226 |
| 32555 | 0.289 | -0.222 | 0.175 |
| 33111 | 0.719 | 0.746 | 0.808 |
| 33112 | 0.669 | 0.690 | 0.769 |
| 33113 | 0.656 | 0.675 | 0.759 |
| 33114 | 0.632 | 0.462 | 0.630 |
| 33115 | 0.607 | 0.241 | 0.497 |
| 33121 | 0.655 | 0.648 | 0.755 |
| 33122 | 0.605 | 0.591 | 0.703 |
| 33123 | 0.592 | 0.577 | 0.689 |
| 33124 | 0.568 | 0.364 | 0.569 |
| 33125 | 0.543 | 0.143 | 0.445 |
| 33131 | 0.639 | 0.623 | 0.742 |
| 33132 | 0.589 | 0.567 | 0.687 |
| 33133 | 0.576 | 0.552 | 0.672 |
| 33134 | 0.552 | 0.339 | 0.554 |
| 33135 | 0.527 | 0.118 | 0.432 |
| 33141 | 0.594 | 0.411 | 0.609 |
| 33142 | 0.544 | 0.354 | 0.561 |
| 33143 | 0.531 | 0.340 | 0.548 |
| 33144 | 0.506 | 0.179 | 0.453 |
| 33145 | 0.482 | 0.013 | 0.354 |
| 33151 | 0.525 | 0.091 | 0.410 |
| 33152 | 0.475 | 0.035 | 0.371 |
| 33153 | 0.462 | 0.020 | 0.361 |
| 33154 | 0.438 | -0.061 | 0.300 |
| 33155<br>33211 | 0.413 | -0.145<br>0.717 | 0.236 |
| 33211 | 0.684<br>0.634 | 0.717<br>0.661 | 0.782<br>0.729 |
| 33212 | 0.034 | 0.001 | 0.729 |

| 33213 | 0.621 | 0.646 | 0.716 |
|-------|-------|--------|-------|
| 33214 | 0.597 | 0.433 | 0.596 |
| 33215 | 0.572 | 0.212 | 0.471 |
| 33221 | 0.620 | 0.619 | 0.716 |
| 33222 | 0.570 | 0.562 | 0.650 |
| 33223 | 0.557 | 0.548 | 0.633 |
| 33224 | 0.533 | 0.335 | 0.521 |
| 33225 | 0.508 | 0.114 | 0.405 |
| 33231 | 0.604 | 0.594 | 0.700 |
| 33232 | 0.554 | 0.538 | 0.630 |
| 33233 | 0.541 | 0.523 | 0.612 |
| 33234 | 0.517 | 0.310 | 0.502 |
| 33235 | 0.492 | 0.089 | 0.389 |
| 33241 | 0.558 | 0.382 | 0.574 |
| 33242 | 0.508 | 0.325 | 0.511 |
| 33243 | 0.495 | 0.311 | 0.495 |
| 33244 | 0.471 | 0.150 | 0.408 |
| 33245 | 0.446 | -0.016 | 0.317 |
| 33251 | 0.490 | 0.062 | 0.384 |
| 33252 | 0.440 | 0.006 | 0.332 |
| 33253 | 0.427 | -0.009 | 0.319 |
| 33254 | 0.403 | -0.090 | 0.265 |
| 33255 | 0.378 | -0.174 | 0.210 |
| 33311 | 0.675 | 0.710 | 0.775 |
| 33312 | 0.625 | 0.654 | 0.720 |
| 33313 | 0.612 | 0.639 | 0.705 |
| 33314 | 0.588 | 0.426 | 0.587 |
| 33315 | 0.563 | 0.205 | 0.465 |
| 33321 | 0.611 | 0.612 | 0.706 |
| 33322 | 0.561 | 0.555 | 0.637 |
| 33323 | 0.548 | 0.541 | 0.619 |
| 33324 | 0.524 | 0.328 | 0.509 |
| 33325 | 0.499 | 0.107 | 0.395 |
| 33331 | 0.595 | 0.587 | 0.689 |
| 33332 | 0.545 | 0.531 | 0.616 |
| 33333 | 0.532 | 0.516 | 0.597 |
| 33334 | 0.508 | 0.303 | 0.490 |
| 33335 | 0.483 | 0.082 | 0.378 |
| 33341 | 0.550 | 0.375 | 0.565 |
| 33342 | 0.500 | 0.318 | 0.499 |
| 33343 | 0.487 | 0.304 | 0.482 |
| 33344 | 0.462 | 0.143 | 0.397 |
| 33345 | 0.438 | -0.023 | 0.309 |
| 33351 | 0.481 | 0.055 | 0.378 |
| 33352 | 0.431 | -0.001 | 0.323 |
| 33353 | 0.418 | -0.016 | 0.308 |
| 33354 | 0.394 | -0.097 | 0.257 |
| 33355 | 0.369 | -0.181 | 0.204 |
| 33411 | 0.646 | 0.603 | 0.709 |

| 33412 | 0.596 | 0.546 | 0.659 |
|-------|-------|--------|-------|
| 33413 | 0.583 | 0.532 | 0.646 |
| 33414 | 0.559 | 0.362 | 0.546 |
| 33415 | 0.534 | 0.186 | 0.443 |
| 33421 | 0.582 | 0.504 | 0.645 |
| 33422 | 0.532 | 0.448 | 0.581 |
| 33423 | 0.519 | 0.433 | 0.565 |
| 33424 | 0.495 | 0.264 | 0.474 |
| 33425 | 0.470 | 0.087 | 0.379 |
| 33431 | 0.566 | 0.480 | 0.630 |
| 33432 | 0.516 | 0.423 | 0.562 |
| 33433 | 0.503 | 0.409 | 0.545 |
| 33434 | 0.479 | 0.239 | 0.456 |
| 33435 | 0.454 | 0.063 | 0.363 |
| 33441 | 0.520 | 0.302 | 0.520 |
| 33442 | 0.470 | 0.246 | 0.460 |
| 33443 | 0.457 | 0.231 | 0.444 |
| 33444 | 0.433 | 0.097 | 0.371 |
| 33445 | 0.408 | -0.042 | 0.295 |
| 33451 | 0.452 | 0.036 | 0.356 |
| 33452 | 0.402 | -0.020 | 0.306 |
| 33453 | 0.389 | -0.035 | 0.293 |
| 33454 | 0.365 | -0.116 | 0.244 |
| 33455 | 0.340 | -0.200 | 0.192 |
| 33511 | 0.586 | 0.383 | 0.573 |
| 33512 | 0.536 | 0.327 | 0.534 |
| 33513 | 0.523 | 0.312 | 0.524 |
| 33514 | 0.499 | 0.231 | 0.463 |
| 33515 | 0.474 | 0.147 | 0.399 |
| 33521 | 0.522 | 0.285 | 0.521 |
| 33522 | 0.472 | 0.228 | 0.468 |
| 33523 | 0.459 | 0.214 | 0.454 |
| 33524 | 0.435 | 0.133 | 0.401 |
| 33525 | 0.410 | 0.049 | 0.346 |
| 33531 | 0.506 | 0.260 | 0.508 |
| 33532 | 0.456 | 0.204 | 0.452 |
| 33533 | 0.443 | 0.189 | 0.437 |
| 33534 | 0.419 | 0.108 | 0.386 |
| 33535 | 0.394 | 0.024 | 0.333 |
| 33541 | 0.461 | 0.155 | 0.430 |
| 33542 | 0.411 | 0.099 | 0.380 |
| 33543 | 0.398 | 0.084 | 0.368 |
| 33544 | 0.373 | 0.003 | 0.318 |
| 33545 | 0.349 | -0.081 | 0.267 |
| 33551 | 0.392 | -0.003 | 0.312 |
| 33552 | 0.342 | -0.059 | 0.273 |
| 33553 | 0.329 | -0.074 | 0.263 |
| 33554 | 0.305 | -0.155 | 0.216 |
| 33555 | 0.280 | -0.239 | 0.167 |

| 34111 | 0.707 | 0.654 | 0.739 |
|-------|-------|--------|-------|
| 34112 | 0.657 | 0.598 | 0.704 |
| 34113 | 0.644 | 0.583 | 0.695 |
| 34114 | 0.620 | 0.402 | 0.580 |
| 34115 | 0.595 | 0.214 | 0.461 |
| 34121 | 0.643 | 0.555 | 0.690 |
| 34122 | 0.593 | 0.499 | 0.642 |
| 34123 | 0.580 | 0.484 | 0.629 |
| 34124 | 0.556 | 0.304 | 0.523 |
| 34125 | 0.531 | 0.116 | 0.413 |
| 34131 | 0.627 | 0.531 | 0.678 |
| 34132 | 0.577 | 0.475 | 0.627 |
| 34133 | 0.564 | 0.460 | 0.613 |
| 34134 | 0.540 | 0.279 | 0.509 |
| 34135 | 0.515 | 0.091 | 0.401 |
| 34141 | 0.582 | 0.345 | 0.556 |
| 34142 | 0.532 | 0.288 | 0.512 |
| 34143 | 0.519 | 0.274 | 0.500 |
| 34144 | 0.495 | 0.133 | 0.413 |
| 34145 | 0.470 | -0.014 | 0.324 |
| 34151 | 0.513 | 0.064 | 0.374 |
| 34152 | 0.463 | 0.008 | 0.339 |
| 34153 | 0.450 | -0.007 | 0.330 |
| 34154 | 0.426 | -0.088 | 0.270 |
| 34155 | 0.401 | -0.172 | 0.207 |
| 34211 | 0.672 | 0.625 | 0.717 |
| 34212 | 0.622 | 0.569 | 0.668 |
| 34213 | 0.609 | 0.554 | 0.656 |
| 34214 | 0.585 | 0.373 | 0.550 |
| 34215 | 0.560 | 0.185 | 0.439 |
| 34221 | 0.608 | 0.527 | 0.655 |
| 34222 | 0.558 | 0.470 | 0.593 |
| 34223 | 0.545 | 0.456 | 0.577 |
| 34224 | 0.521 | 0.275 | 0.479 |
| 34225 | 0.496 | 0.087 | 0.377 |
| 34231 | 0.592 | 0.502 | 0.639 |
| 34232 | 0.542 | 0.446 | 0.574 |
| 34233 | 0.529 | 0.431 | 0.557 |
| 34234 | 0.505 | 0.250 | 0.461 |
| 34235 | 0.480 | 0.062 | 0.362 |
| 34241 | 0.547 | 0.316 | 0.525 |
| 34242 | 0.497 | 0.259 | 0.466 |
| 34243 | 0.484 | 0.245 | 0.451 |
| 34244 | 0.460 | 0.104 | 0.373 |
| 34245 | 0.435 | -0.043 | 0.291 |
| 34251 | 0.478 | 0.035 | 0.352 |
| 34252 | 0.428 | -0.021 | 0.304 |
| 34253 | 0.415 | -0.036 | 0.292 |
| 34254 | 0.391 | -0.117 | 0.240 |

| 34255 | 0.366 | -0.201 | 0.186 |
|-------|-------|--------|-------|
| 34311 | 0.663 | 0.618 | 0.711 |
| 34312 | 0.613 | 0.562 | 0.660 |
| 34313 | 0.600 | 0.547 | 0.646 |
| 34314 | 0.576 | 0.366 | 0.542 |
| 34315 | 0.551 | 0.178 | 0.434 |
| 34321 | 0.599 | 0.519 | 0.646 |
| 34322 | 0.549 | 0.463 | 0.581 |
| 34323 | 0.536 | 0.448 | 0.564 |
| 34324 | 0.512 | 0.268 | 0.468 |
| 34325 | 0.487 | 0.080 | 0.369 |
| 34331 | 0.583 | 0.495 | 0.630 |
| 34332 | 0.533 | 0.439 | 0.561 |
| 34333 | 0.520 | 0.424 | 0.543 |
| 34334 | 0.496 | 0.243 | 0.450 |
| 34335 | 0.471 | 0.055 | 0.352 |
| 34341 | 0.538 | 0.309 | 0.517 |
| 34342 | 0.488 | 0.252 | 0.455 |
| 34343 | 0.475 | 0.238 | 0.439 |
| 34344 | 0.451 | 0.097 | 0.363 |
| 34345 | 0.426 | -0.050 | 0.284 |
| 34351 | 0.469 | 0.028 | 0.347 |
| 34352 | 0.419 | -0.028 | 0.296 |
| 34353 | 0.406 | -0.043 | 0.282 |
| 34354 | 0.382 | -0.124 | 0.232 |
| 34355 | 0.357 | -0.208 | 0.180 |
| 34411 | 0.634 | 0.532 | 0.654 |
| 34412 | 0.584 | 0.476 | 0.608 |
| 34413 | 0.571 | 0.461 | 0.596 |
| 34414 | 0.547 | 0.313 | 0.506 |
| 34415 | 0.522 | 0.159 | 0.413 |
| 34421 | 0.570 | 0.433 | 0.594 |
| 34422 | 0.520 | 0.377 | 0.535 |
| 34423 | 0.507 | 0.362 | 0.519 |
| 34424 | 0.483 | 0.214 | 0.438 |
| 34425 | 0.458 | 0.061 | 0.353 |
| 34431 | 0.554 | 0.409 | 0.580 |
| 34432 | 0.504 | 0.353 | 0.516 |
| 34433 | 0.491 | 0.338 | 0.500 |
| 34434 | 0.467 | 0.190 | 0.421 |
| 34435 | 0.442 | 0.036 | 0.338 |
| 34441 | 0.509 | 0.249 | 0.478 |
| 34442 | 0.459 | 0.193 | 0.422 |
| 34443 | 0.446 | 0.178 | 0.407 |
| 34444 | 0.422 | 0.057 | 0.340 |
| 34445 | 0.397 | -0.069 | 0.270 |
| 34451 | 0.440 | 0.009 | 0.326 |
| 34452 | 0.390 | -0.047 | 0.280 |
| 34453 | 0.377 | -0.062 | 0.268 |
| 2 | | | |

| 34454 | 0.353 | -0.143 | 0.219 |
|-------|-------|--------|-------|
| 34455 | 0.328 | -0.227 | 0.169 |
| 34511 | 0.574 | 0.356 | 0.537 |
| 34512 | 0.524 | 0.300 | 0.502 |
| 34513 | 0.511 | 0.285 | 0.493 |
| 34514 | 0.487 | 0.204 | 0.433 |
| 34515 | 0.462 | 0.120 | 0.370 |
| 34521 | 0.510 | 0.258 | 0.489 |
| 34522 | 0.460 | 0.201 | 0.440 |
| 34523 | 0.447 | 0.187 | 0.428 |
| 34524 | 0.423 | 0.106 | 0.375 |
| 34525 | 0.398 | 0.022 | 0.321 |
| 34531 | 0.494 | 0.233 | 0.477 |
| 34532 | 0.444 | 0.177 | 0.425 |
| 34533 | 0.431 | 0.162 | 0.411 |
| 34534 | 0.407 | 0.081 | 0.361 |
| 34535 | 0.382 | -0.003 | 0.309 |
| 34541 | 0.449 | 0.128 | 0.400 |
| 34542 | 0.399 | 0.072 | 0.354 |
| 34543 | 0.386 | 0.057 | 0.343 |
| 34544 | 0.362 | -0.024 | 0.294 |
| 34545 | 0.337 | -0.108 | 0.244 |
| 34551 | 0.380 | -0.030 | 0.283 |
| 34552 | 0.330 | -0.086 | 0.248 |
| 34553 | 0.317 | -0.101 | 0.239 |
| 34554 | 0.293 | -0.182 | 0.193 |
| 34555 | 0.268 | -0.266 | 0.145 |
| 35111 | 0.671 | 0.367 | 0.522 |
| 35112 | 0.621 | 0.311 | 0.501 |
| 35113 | 0.608 | 0.296 | 0.495 |
| 35114 | 0.584 | 0.215 | 0.423 |
| 35115 | 0.559 | 0.131 | 0.348 |
| 35121 | 0.607 | 0.269 | 0.487 |
| 35122 | 0.557 | 0.212 | 0.452 |
| 35123 | 0.544 | 0.198 | 0.443 |
| 35124 | 0.520 | 0.117 | 0.379 |
| 35125 | 0.495 | 0.033 | 0.313 |
| 35131 | 0.591 | 0.244 | 0.478 |
| 35132 | 0.541 | 0.188 | 0.440 |
| 35133 | 0.528 | 0.173 | 0.430 |
| 35134 | 0.504 | 0.092 | 0.368 |
| 35135 | 0.479 | 0.008 | 0.304 |
| 35141 | 0.546 | 0.139 | 0.391 |
| 35142 | 0.496 | 0.083 | 0.360 |
| 35143 | 0.483 | 0.068 | 0.352 |
| 35144 | 0.458 | -0.013 | 0.292 |
| 35145 | 0.434 | -0.097 | 0.229 |
| 35151 | 0.477 | -0.019 | 0.261 |
| 35152 | 0.427 | -0.075 | 0.240 |

| 35153 | 0.414 | -0.090 | 0.234 |
|-------|-------|--------|-------|
| 35154 | 0.390 | -0.171 | 0.177 |
| 35155 | 0.365 | -0.255 | 0.117 |
| 35211 | 0.636 | 0.338 | 0.514 |
| 35212 | 0.586 | 0.282 | 0.479 |
| 35213 | 0.573 | 0.267 | 0.469 |
| 35214 | 0.549 | 0.186 | 0.406 |
| 35215 | 0.524 | 0.102 | 0.339 |
| 35221 | 0.572 | 0.240 | 0.465 |
| 35222 | 0.522 | 0.183 | 0.416 |
| 35223 | 0.509 | 0.169 | 0.403 |
| 35224 | 0.485 | 0.088 | 0.348 |
| 35225 | 0.460 | 0.004 | 0.290 |
| 35231 | 0.556 | 0.215 | 0.452 |
| 35232 | 0.506 | 0.159 | 0.400 |
| 35233 | 0.493 | 0.144 | 0.387 |
| 35234 | 0.469 | 0.063 | 0.334 |
| 35235 | 0.444 | -0.021 | 0.278 |
| 35241 | 0.510 | 0.110 | 0.372 |
| 35242 | 0.460 | 0.054 | 0.327 |
| 35243 | 0.447 | 0.039 | 0.315 |
| 35244 | 0.423 | -0.042 | 0.264 |
| 35245 | 0.398 | -0.126 | 0.210 |
| 35251 | 0.442 | -0.048 | 0.252 |
| 35252 | 0.392 | -0.104 | 0.217 |
| 35253 | 0.379 | -0.119 | 0.208 |
| 35254 | 0.355 | -0.200 | 0.159 |
| 35255 | 0.330 | -0.284 | 0.108 |
| 35311 | 0.627 | 0.331 | 0.512 |
| 35312 | 0.577 | 0.275 | 0.473 |
| 35313 | 0.564 | 0.260 | 0.463 |
| 35314 | 0.540 | 0.179 | 0.401 |
| 35315 | 0.515 | 0.095 | 0.337 |
| 35321 | 0.563 | 0.233 | 0.459 |
| 35322 | 0.513 | 0.176 | 0.407 |
| 35323 | 0.500 | 0.162 | 0.393 |
| 35324 | 0.476 | 0.081 | 0.340 |
| 35325 | 0.451 | -0.004 | 0.285 |
| 35331 | 0.547 | 0.208 | 0.446 |
| 35332 | 0.497 | 0.152 | 0.391 |
| 35333 | 0.484 | 0.137 | 0.376 |
| 35334 | 0.460 | 0.056 | 0.325 |
| 35335 | 0.435 | -0.028 | 0.272 |
| 35341 | 0.502 | 0.103 | 0.368 |
| 35342 | 0.452 | 0.047 | 0.319 |
| 35343 | 0.439 | 0.032 | 0.307 |
| 35344 | 0.414 | -0.049 | 0.257 |
| 35345 | 0.390 | -0.133 | 0.206 |
| 35351 | 0.433 | -0.055 | 0.250 |

| 35352 | 0.383 | -0.111 | 0.212 |
|-------|-------|--------|-------|
| 35353 | 0.370 | -0.126 | 0.202 |
| 35354 | 0.346 | -0.207 | 0.155 |
| 35355 | 0.321 | -0.291 | 0.106 |
| 35411 | 0.598 | 0.312 | 0.483 |
| 35412 | 0.548 | 0.256 | 0.450 |
| 35413 | 0.535 | 0.241 | 0.441 |
| 35414 | 0.511 | 0.160 | 0.381 |
| 35415 | 0.486 | 0.076 | 0.318 |
| 35421 | 0.534 | 0.213 | 0.436 |
| 35422 | 0.484 | 0.157 | 0.389 |
| 35423 | 0.471 | 0.142 | 0.377 |
| 35424 | 0.447 | 0.061 | 0.325 |
| 35425 | 0.422 | -0.023 | 0.271 |
| 35431 | 0.518 | 0.189 | 0.424 |
| 35432 | 0.468 | 0.133 | 0.374 |
| 35433 | 0.455 | 0.118 | 0.361 |
| 35434 | 0.431 | 0.037 | 0.312 |
| 35435 | 0.406 | -0.047 | 0.260 |
| 35441 | 0.472 | 0.084 | 0.347 |
| 35442 | 0.422 | 0.028 | 0.304 |
| 35443 | 0.409 | 0.013 | 0.293 |
| 35444 | 0.385 | -0.068 | 0.245 |
| 35445 | 0.360 | -0.152 | 0.195 |
| 35451 | 0.404 | -0.074 | 0.231 |
| 35452 | 0.354 | -0.130 | 0.198 |
| 35453 | 0.341 | -0.145 | 0.190 |
| 35454 | 0.317 | -0.226 | 0.144 |
| 35455 | 0.292 | -0.310 | 0.097 |
| 35511 | 0.538 | 0.273 | 0.424 |
| 35512 | 0.488 | 0.217 | 0.403 |
| 35513 | 0.475 | 0.202 | 0.397 |
| 35514 | 0.451 | 0.121 | 0.339 |
| 35515 | 0.426 | 0.037 | 0.279 |
| 35521 | 0.474 | 0.175 | 0.389 |
| 35522 | 0.424 | 0.118 | 0.353 |
| 35523 | 0.411 | 0.104 | 0.344 |
| 35524 | 0.387 | 0.023 | 0.295 |
| 35525 | 0.362 | -0.062 | 0.244 |
| 35531 | 0.458 | 0.150 | 0.380 |
| 35532 | 0.408 | 0.094 | 0.341 |
| 35533 | 0.395 | 0.079 | 0.331 |
| 35534 | 0.371 | -0.002 | 0.284 |
| 35535 | 0.346 | -0.086 | 0.235 |
| 35541 | 0.413 | 0.045 | 0.305 |
| 35542 | 0.363 | -0.011 | 0.273 |
| 35543 | 0.350 | -0.026 | 0.265 |
| 35544 | 0.325 | -0.107 | 0.219 |
| 35545 | 0.301 | -0.191 | 0.172 |

| 35551 | 0.344 | -0.113 | 0.193 |
|-------|-------|--------|-------|
| 35552 | 0.294 | -0.169 | 0.171 |
| 35553 | 0.281 | -0.184 | 0.165 |
| 35554 | 0.257 | -0.265 | 0.122 |
| 35555 | 0.232 | -0.349 | 0.077 |
| 41111 | 0.748 | 0.813 | 0.824 |
| 41112 | 0.698 | 0.757 | 0.804 |
| 41113 | 0.685 | 0.742 | 0.798 |
| 41114 | 0.661 | 0.539 | 0.663 |
| 41115 | 0.636 | 0.327 | 0.523 |
| 41121 | 0.684 | 0.714 | 0.790 |
| 41122 | 0.634 | 0.658 | 0.755 |
| 41123 | 0.621 | 0.643 | 0.747 |
| 41124 | 0.597 | 0.440 | 0.620 |
| 41125 | 0.572 | 0.229 | 0.489 |
| 41131 | 0.668 | 0.690 | 0.781 |
| 41132 | 0.618 | 0.634 | 0.744 |
| 41133 | 0.605 | 0.619 | 0.734 |
| 41134 | 0.581 | 0.416 | 0.609 |
| 41135 | 0.556 | 0.204 | 0.480 |
| 41141 | 0.623 | 0.485 | 0.643 |
| 41142 | 0.573 | 0.429 | 0.612 |
| 41143 | 0.560 | 0.414 | 0.604 |
| 41144 | 0.536 | 0.260 | 0.501 |
| 41145 | 0.511 | 0.099 | 0.394 |
| 41151 | 0.554 | 0.177 | 0.436 |
| 41152 | 0.504 | 0.121 | 0.415 |
| 41153 | 0.491 | 0.106 | 0.410 |
| 41154 | 0.467 | 0.025 | 0.339 |
| 41155 | 0.442 | -0.059 | 0.264 |
| 41211 | 0.713 | 0.784 | 0.816 |
| 41212 | 0.663 | 0.728 | 0.782 |
| 41213 | 0.650 | 0.713 | 0.773 |
| 41214 | 0.626 | 0.510 | 0.647 |
| 41215 | 0.601 | 0.299 | 0.516 |
| 41221 | 0.649 | 0.686 | 0.769 |
| 41222 | 0.599 | 0.629 | 0.721 |
| 41223 | 0.586 | 0.615 | 0.708 |
| 41224 | 0.562 | 0.411 | 0.590 |
| 41225 | 0.537 | 0.200 | 0.468 |
| 41231 | 0.633 | 0.661 | 0.757 |
| 41232 | 0.583 | 0.605 | 0.706 |
| 41233 | 0.570 | 0.590 | 0.692 |
| 41234 | 0.546 | 0.387 | 0.576 |
| 41235 | 0.521 | 0.176 | 0.456 |
| 41241 | 0.587 | 0.456 | 0.626 |
| 41242 | 0.537 | 0.400 | 0.581 |
| 41243 | 0.524 | 0.385 | 0.570 |
| 41244 | 0.500 | 0.231 | 0.475 |

| 41245 | 0.475 | 0.070 | 0.376 |
|-------|-------|--------|-------|
| 41251 | 0.519 | 0.149 | 0.429 |
| 41252 | 0.469 | 0.092 | 0.394 |
| 41253 | 0.456 | 0.078 | 0.386 |
| 41254 | 0.432 | -0.004 | 0.322 |
| 41255 | 0.407 | -0.088 | 0.256 |
| 41311 | 0.704 | 0.777 | 0.814 |
| 41312 | 0.654 | 0.721 | 0.777 |
| 41313 | 0.641 | 0.706 | 0.767 |
| 41314 | 0.617 | 0.503 | 0.643 |
| 41315 | 0.592 | 0.291 | 0.514 |
| 41321 | 0.640 | 0.678 | 0.763 |
| 41322 | 0.590 | 0.622 | 0.712 |
| 41323 | 0.577 | 0.607 | 0.699 |
| 41324 | 0.553 | 0.404 | 0.583 |
| 41325 | 0.528 | 0.193 | 0.462 |
| 41331 | 0.624 | 0.654 | 0.751 |
| 41332 | 0.574 | 0.598 | 0.696 |
| 41333 | 0.561 | 0.583 | 0.682 |
| 41334 | 0.537 | 0.380 | 0.568 |
| 41335 | 0.512 | 0.168 | 0.450 |
| 41341 | 0.579 | 0.449 | 0.621 |
| 41342 | 0.529 | 0.393 | 0.574 |
| 41343 | 0.516 | 0.378 | 0.561 |
| 41344 | 0.492 | 0.224 | 0.468 |
| 41345 | 0.467 | 0.063 | 0.371 |
| 41351 | 0.510 | 0.141 | 0.427 |
| 41352 | 0.460 | 0.085 | 0.389 |
| 41353 | 0.447 | 0.070 | 0.380 |
| 41354 | 0.423 | -0.011 | 0.318 |
| 41355 | 0.398 | -0.095 | 0.254 |
| 41411 | 0.675 | 0.676 | 0.744 |
| 41412 | 0.625 | 0.620 | 0.711 |
| 41413 | 0.612 | 0.605 | 0.703 |
| 41414 | 0.588 | 0.442 | 0.596 |
| 41415 | 0.563 | 0.272 | 0.485 |
| 41421 | 0.611 | 0.577 | 0.698 |
| 41422 | 0.561 | 0.521 | 0.653 |
| 41423 | 0.548 | 0.506 | 0.641 |
| 41424 | 0.524 | 0.343 | 0.542 |
| 41425 | 0.499 | 0.174 | 0.439 |
| 41431 | 0.595 | 0.553 | 0.687 |
| 41432 | 0.545 | 0.497 | 0.638 |
| 41433 | 0.532 | 0.482 | 0.625 |
| 41434 | 0.508 | 0.319 | 0.529 |
| 41435 | 0.483 | 0.149 | 0.428 |
| 41441 | 0.550 | 0.381 | 0.572 |
| 41442 | 0.500 | 0.325 | 0.530 |
| 41443 | 0.487 | 0.310 | 0.519 |

| 41444 | 0.462 | 0.180 | 0.437 |
|-------|-------|--------|-------|
| 41445 | 0.438 | 0.044 | 0.351 |
| 41451 | 0.481 | 0.122 | 0.398 |
| 41452 | 0.431 | 0.066 | 0.366 |
| 41453 | 0.418 | 0.051 | 0.358 |
| 41454 | 0.394 | -0.030 | 0.298 |
| 41455 | 0.369 | -0.114 | 0.236 |
| 41511 | 0.615 | 0.469 | 0.599 |
| 41512 | 0.565 | 0.413 | 0.578 |
| 41513 | 0.552 | 0.398 | 0.573 |
| 41514 | 0.528 | 0.317 | 0.501 |
| 41515 | 0.503 | 0.233 | 0.427 |
| 41521 | 0.551 | 0.371 | 0.565 |
| 41522 | 0.501 | 0.315 | 0.531 |
| 41523 | 0.488 | 0.300 | 0.522 |
| 41524 | 0.464 | 0.219 | 0.459 |
| 41525 | 0.439 | 0.135 | 0.393 |
| 41531 | 0.535 | 0.346 | 0.556 |
| 41532 | 0.485 | 0.290 | 0.519 |
| 41533 | 0.472 | 0.275 | 0.509 |
| 41534 | 0.448 | 0.194 | 0.448 |
| 41535 | 0.423 | 0.110 | 0.384 |
| 41541 | 0.490 | 0.241 | 0.470 |
| 41542 | 0.440 | 0.185 | 0.439 |
| 41543 | 0.427 | 0.170 | 0.431 |
| 41544 | 0.403 | 0.089 | 0.372 |
| 41545 | 0.378 | 0.005 | 0.310 |
| 41551 | 0.421 | 0.083 | 0.340 |
| 41552 | 0.371 | 0.027 | 0.320 |
| 41553 | 0.358 | 0.012 | 0.314 |
| 41554 | 0.334 | -0.069 | 0.257 |
| 41555 | 0.309 | -0.153 | 0.198 |
| 42111 | 0.703 | 0.726 | 0.787 |
| 42112 | 0.653 | 0.670 | 0.752 |
| 42113 | 0.640 | 0.655 | 0.743 |
| 42114 | 0.616 | 0.452 | 0.617 |
| 42115 | 0.591 | 0.241 | 0.486 |
| 42121 | 0.639 | 0.628 | 0.738 |
| 42122 | 0.589 | 0.572 | 0.690 |
| 42123 | 0.576 | 0.557 | 0.677 |
| 42124 | 0.552 | 0.353 | 0.560 |
| 42125 | 0.527 | 0.142 | 0.437 |
| 42131 | 0.623 | 0.603 | 0.726 |
| 42132 | 0.573 | 0.547 | 0.674 |
| 42133 | 0.560 | 0.532 | 0.661 |
| 42134 | 0.536 | 0.329 | 0.545 |
| 42135 | 0.511 | 0.118 | 0.425 |
| 42141 | 0.578 | 0.399 | 0.595 |
| 42142 | 0.528 | 0.342 | 0.550 |
| 42143 | 0.515 | 0.328 | 0.539 |
|----------------|----------------|----------------|----------------|
| 42144 | 0.491 | 0.173 | 0.444 |
| 42145 | 0.466 | 0.013 | 0.346 |
| 42151 | 0.509 | 0.091 | 0.399 |
| 42152 | 0.459 | 0.034 | 0.364 |
| 42153 | 0.446 | 0.020 | 0.355 |
| 42154 | 0.422 | -0.061 | 0.292 |
| 42155 | 0.397 | -0.145 | 0.227 |
| 42211<br>42212 | 0.668 | 0.698 | 0.764 |
| | 0.618 | 0.641<br>0.627 | 0.716<br>0.704 |
| 42213<br>42214 | 0.605<br>0.581 | 0.627 | 0.704 |
| 42214 | 0.556 | 0.423 | 0.366 |
| | 0.556 | 0.212 | 0.404 |
| 42221<br>42222 | 0.554 | 0.599 | 0.703 |
| 42222 | | | 0.624 |
| 42223 | 0.541<br>0.517 | 0.528<br>0.325 | 0.624 |
| 42224 | 0.517 | 0.323 | 0.515 |
| 42223 | 0.492 | 0.113 | 0.402 |
| 42231 | 0.538 | 0.518 | 0.622 |
| 42232 | 0.525 | 0.518 | 0.605 |
| 42234 | 0.525 | 0.304 | 0.603 |
| 42235 | 0.301 | 0.089 | 0.496 |
| 42241 | 0.543 | 0.009 | 0.563 |
| 42242 | 0.493 | 0.313 | 0.505 |
| 42243 | 0.480 | 0.299 | 0.490 |
| 42244 | 0.455 | 0.144 | 0.403 |
| 42245 | 0.431 | -0.016 | 0.314 |
| 42251 | 0.474 | 0.062 | 0.377 |
| 42252 | 0.424 | 0.006 | 0.329 |
| 42253 | 0.411 | -0.009 | 0.316 |
| 42254 | 0.387 | -0.090 | 0.262 |
| 42255 | 0.362 | -0.174 | 0.205 |
| 42311 | 0.659 | 0.690 | 0.759 |
| 42312 | 0.609 | 0.634 | 0.707 |
| 42313 | 0.596 | 0.619 | 0.694 |
| 42314 | 0.572 | 0.416 | 0.578 |
| 42315 | 0.547 | 0.205 | 0.459 |
| 42321 | 0.595 | 0.592 | 0.694 |
| 42322 | 0.545 | 0.536 | 0.629 |
| 42323 | 0.532 | 0.521 | 0.612 |
| 42324 | 0.508 | 0.317 | 0.504 |
| 42325 | 0.483 | 0.106 | 0.393 |
| 42331 | 0.579 | 0.567 | 0.678 |
| 42332 | 0.529 | 0.511 | 0.609 |
| 42333 | 0.516 | 0.496 | 0.591 |
| 42334 | 0.492 | 0.293 | 0.486 |
| 42335 | 0.467 | 0.082 | 0.377 |
| 42341 | 0.534 | 0.363 | 0.555 |

| 42342 | 0.484 | 0.306 | 0.494 |
|-------|-------|--------|-------|
| 42343 | 0.471 | 0.292 | 0.477 |
| 42344 | 0.447 | 0.137 | 0.393 |
| 42345 | 0.422 | -0.023 | 0.306 |
| 42351 | 0.465 | 0.055 | 0.372 |
| 42352 | 0.415 | -0.002 | 0.320 |
| 42353 | 0.402 | -0.016 | 0.307 |
| 42354 | 0.378 | -0.097 | 0.254 |
| 42355 | 0.353 | -0.181 | 0.200 |
| 42411 | 0.630 | 0.589 | 0.694 |
| 42412 | 0.580 | 0.533 | 0.648 |
| 42413 | 0.567 | 0.518 | 0.636 |
| 42414 | 0.543 | 0.355 | 0.538 |
| 42415 | 0.518 | 0.186 | 0.436 |
| 42421 | 0.566 | 0.491 | 0.635 |
| 42422 | 0.516 | 0.434 | 0.575 |
| 42423 | 0.503 | 0.420 | 0.559 |
| 42424 | 0.479 | 0.257 | 0.469 |
| 42425 | 0.454 | 0.087 | 0.376 |
| 42431 | 0.550 | 0.466 | 0.620 |
| 42432 | 0.500 | 0.410 | 0.557 |
| 42433 | 0.487 | 0.395 | 0.540 |
| 42434 | 0.463 | 0.232 | 0.452 |
| 42435 | 0.438 | 0.063 | 0.361 |
| 42441 | 0.505 | 0.294 | 0.512 |
| 42442 | 0.455 | 0.238 | 0.455 |
| 42443 | 0.442 | 0.223 | 0.441 |
| 42444 | 0.418 | 0.093 | 0.367 |
| 42445 | 0.393 | -0.042 | 0.291 |
| 42451 | 0.436 | 0.036 | 0.349 |
| 42452 | 0.386 | -0.021 | 0.303 |
| 42453 | 0.373 | -0.035 | 0.291 |
| 42454 | 0.349 | -0.116 | 0.240 |
| 42455 | 0.324 | -0.200 | 0.187 |
| 42511 | 0.570 | 0.383 | 0.562 |
| 42512 | 0.520 | 0.326 | 0.527 |
| 42513 | 0.507 | 0.312 | 0.518 |
| 42514 | 0.483 | 0.231 | 0.455 |
| 42515 | 0.458 | 0.147 | 0.390 |
| 42521 | 0.506 | 0.284 | 0.513 |
| 42522 | 0.456 | 0.228 | 0.465 |
| 42523 | 0.443 | 0.213 | 0.452 |
| 42524 | 0.419 | 0.132 | 0.398 |
| 42525 | 0.394 | 0.048 | 0.341 |
| 42531 | 0.490 | 0.260 | 0.501 |
| 42532 | 0.440 | 0.203 | 0.449 |
| 42533 | 0.427 | 0.189 | 0.436 |
| 42534 | 0.403 | 0.108 | 0.383 |
| 42535 | 0.378 | 0.024 | 0.329 |

| 42541 | 0.445 | 0.155 | 0.422 |
|-------|-------|--------|-------|
| 42542 | 0.395 | 0.098 | 0.377 |
| 42543 | 0.382 | 0.084 | 0.365 |
| 42544 | 0.358 | 0.003 | 0.314 |
| 42545 | 0.333 | -0.081 | 0.261 |
| 42551 | 0.376 | -0.003 | 0.303 |
| 42552 | 0.326 | -0.060 | 0.268 |
| 42553 | 0.313 | -0.074 | 0.259 |
| 42554 | 0.289 | -0.155 | 0.210 |
| 42555 | 0.264 | -0.239 | 0.160 |
| 43111 | 0.694 | 0.709 | 0.779 |
| 43112 | 0.644 | 0.653 | 0.741 |
| 43113 | 0.631 | 0.638 | 0.732 |
| 43114 | 0.607 | 0.435 | 0.607 |
| 43115 | 0.582 | 0.223 | 0.478 |
| 43121 | 0.630 | 0.610 | 0.728 |
| 43122 | 0.580 | 0.554 | 0.677 |
| 43123 | 0.567 | 0.539 | 0.663 |
| 43124 | 0.543 | 0.336 | 0.547 |
| 43125 | 0.518 | 0.125 | 0.427 |
| 43131 | 0.614 | 0.586 | 0.715 |
| 43132 | 0.564 | 0.530 | 0.660 |
| 43133 | 0.551 | 0.515 | 0.646 |
| 43134 | 0.527 | 0.312 | 0.533 |
| 43135 | 0.502 | 0.100 | 0.414 |
| 43141 | 0.569 | 0.381 | 0.585 |
| 43142 | 0.519 | 0.325 | 0.538 |
| 43143 | 0.506 | 0.310 | 0.525 |
| 43144 | 0.482 | 0.156 | 0.433 |
| 43145 | 0.457 | -0.005 | 0.336 |
| 43151 | 0.500 | 0.073 | 0.391 |
| 43152 | 0.450 | 0.017 | 0.353 |
| 43153 | 0.437 | 0.002 | 0.344 |
| 43154 | 0.413 | -0.079 | 0.282 |
| 43155 | 0.388 | -0.163 | 0.219 |
| 43211 | 0.659 | 0.680 | 0.754 |
| 43212 | 0.609 | 0.624 | 0.703 |
| 43213 | 0.596 | 0.609 | 0.690 |
| 43214 | 0.572 | 0.406 | 0.574 |
| 43215 | 0.547 | 0.195 | 0.454 |
| 43221 | 0.595 | 0.582 | 0.689 |
| 43222 | 0.545 | 0.525 | 0.625 |
| 43223 | 0.532 | 0.511 | 0.608 |
| 43224 | 0.508 | 0.307 | 0.500 |
| 43225 | 0.483 | 0.096 | 0.389 |
| 43231 | 0.579 | 0.557 | 0.673 |
| 43232 | 0.529 | 0.501 | 0.605 |
| 43233 | 0.516 | 0.486 | 0.587 |
| 43234 | 0.492 | 0.283 | 0.482 |

| 43235 | 0.467 | 0.072 | 0.372 |
|-------|-------|--------|-------|
| 43241 | 0.533 | 0.352 | 0.551 |
| 43242 | 0.483 | 0.296 | 0.489 |
| 43243 | 0.470 | 0.281 | 0.473 |
| 43244 | 0.446 | 0.127 | 0.389 |
| 43245 | 0.421 | -0.034 | 0.301 |
| 43251 | 0.465 | 0.045 | 0.367 |
| 43252 | 0.415 | -0.012 | 0.316 |
| 43253 | 0.402 | -0.027 | 0.302 |
| 43254 | 0.378 | -0.108 | 0.249 |
| 43255 | 0.353 | -0.192 | 0.195 |
| 43311 | 0.650 | 0.673 | 0.748 |
| 43312 | 0.600 | 0.617 | 0.693 |
| 43313 | 0.587 | 0.602 | 0.679 |
| 43314 | 0.563 | 0.399 | 0.566 |
| 43315 | 0.538 | 0.187 | 0.448 |
| 43321 | 0.586 | 0.574 | 0.680 |
| 43322 | 0.536 | 0.518 | 0.612 |
| 43323 | 0.523 | 0.503 | 0.594 |
| 43324 | 0.499 | 0.300 | 0.488 |
| 43325 | 0.474 | 0.089 | 0.379 |
| 43331 | 0.570 | 0.550 | 0.663 |
| 43332 | 0.520 | 0.494 | 0.591 |
| 43333 | 0.507 | 0.479 | 0.573 |
| 43334 | 0.483 | 0.276 | 0.469 |
| 43335 | 0.458 | 0.064 | 0.362 |
| 43341 | 0.525 | 0.345 | 0.542 |
| 43342 | 0.475 | 0.289 | 0.477 |
| 43343 | 0.462 | 0.274 | 0.461 |
| 43344 | 0.438 | 0.120 | 0.378 |
| 43345 | 0.413 | -0.041 | 0.293 |
| 43351 | 0.456 | 0.037 | 0.361 |
| 43352 | 0.406 | -0.019 | 0.306 |
| 43353 | 0.393 | -0.034 | 0.292 |
| 43354 | 0.369 | -0.115 | 0.241 |
| 43355 | 0.344 | -0.199 | 0.189 |
| 43411 | 0.621 | 0.572 | 0.684 |
| 43412 | 0.571 | 0.516 | 0.635 |
| 43413 | 0.558 | 0.501 | 0.623 |
| 43414 | 0.534 | 0.338 | 0.526 |
| 43415 | 0.509 | 0.168 | 0.426 |
| 43421 | 0.557 | 0.473 | 0.622 |
| 43422 | 0.507 | 0.417 | 0.559 |
| 43423 | 0.494 | 0.402 | 0.543 |
| 43424 | 0.470 | 0.239 | 0.455 |
| 43425 | 0.445 | 0.070 | 0.363 |
| 43431 | 0.541 | 0.449 | 0.606 |
| 43432 | 0.491 | 0.393 | 0.540 |
| 43433 | 0.478 | 0.378 | 0.523 |

| 43434 | 0.454 | 0.215 | 0.437 |
|-------|-------|----------|-------|
| 43435 | 0.429 | 0.045 | 0.347 |
| 43441 | 0.496 | 0.277 | 0.500 |
| 43442 | 0.446 | 0.221 | 0.440 |
| 43443 | 0.433 | 0.206 | 0.425 |
| 43444 | 0.408 | 0.076 | 0.353 |
| 43445 | 0.384 | -0.060 | 0.279 |
| 43451 | 0.427 | 0.018 | 0.339 |
| 43452 | 0.377 | -0.038 | 0.290 |
| 43453 | 0.364 | -0.053 | 0.277 |
| 43454 | 0.340 | -0.134 | 0.228 |
| 43455 | 0.315 | -0.218 | 0.177 |
| 43511 | 0.561 | 0.365 | 0.554 |
| 43512 | 0.511 | 0.309 | 0.516 |
| 43513 | 0.498 | 0.294 | 0.507 |
| 43514 | 0.474 | 0.213 | 0.445 |
| 43515 | 0.449 | 0.129 | 0.382 |
| 43521 | 0.497 | 0.267 | 0.503 |
| 43522 | 0.447 | 0.211 | 0.452 |
| 43523 | 0.434 | 0.196 | 0.438 |
| 43524 | 0.410 | 0.115 | 0.385 |
| 43525 | 0.385 | 0.031 | 0.330 |
| 43531 | 0.481 | 0.242 | 0.490 |
| 43532 | 0.431 | 0.186 | 0.435 |
| 43533 | 0.418 | 0.171 | 0.421 |
| 43534 | 0.394 | 0.090 | 0.370 |
| 43535 | 0.369 | 0.006 | 0.318 |
| 43541 | 0.436 | 0.137 | 0.412 |
| 43542 | 0.386 | 0.081 | 0.364 |
| 43543 | 0.373 | 0.066 | 0.352 |
| 43544 | 0.349 | -0.015 | 0.303 |
| 43545 | 0.324 | -0.099 | 0.252 |
| 43551 | 0.367 | -0.021 | 0.295 |
| 43552 | 0.317 | -0.077 | 0.257 |
| 43553 | 0.304 | -0.092 | 0.248 |
| 43554 | 0.280 | -0.173 | 0.201 |
| 43555 | 0.255 | -0.257 | 0.152 |
| 44111 | 0.683 | 0.622 | 0.712 |
| 44112 | 0.633 | 0.565 | 0.678 |
| 44113 | 0.620 | 0.551 | 0.669 |
| 44114 | 0.596 | 0.377 | 0.558 |
| 44115 | 0.571 | 0.197 | 0.442 |
| 44121 | 0.619 | 0.523 | 0.664 |
| 44122 | 0.569 | 0.467 | 0.618 |
| 44123 | 0.556 | 0.452 | 0.605 |
| 44124 | 0.532 | 0.278 | 0.502 |
| 44125 | 0.507 | 0.098 | 0.395 |
| 44131 | 0.603 | 0.499 | 0.653 |
| 44132 | 0.553 | 0.442 | 0.602 |
| | 2.220 | <b>-</b> | |

| 44133 | 0.540 | 0.428 | 0.589 |
|----------------|----------------|----------------|----------------|
| 44134 | 0.516 | 0.254 | 0.488 |
| 44135 | 0.491 | 0.074 | 0.384 |
| 44141 | 0.557 | 0.318 | 0.534 |
| 44142 | 0.507 | 0.262 | 0.490 |
| 44143 | 0.494 | 0.247 | 0.479 |
| 44144 | 0.470 | 0.110 | 0.394 |
| 44145 | 0.445 | -0.032 | 0.306 |
| 44151 | 0.489 | 0.047 | 0.355 |
| 44152 | 0.439 | -0.010 | 0.322 |
| 44153 | 0.426 | -0.024 | 0.313 |
| 44154 | 0.402 | -0.105 | 0.253 |
| 44155 | 0.377 | -0.189 | 0.190 |
| 44211 | 0.647 | 0.593 | 0.691 |
| 44212 | 0.597 | 0.536 | 0.644 |
| 44213 | 0.584 | 0.522 | 0.632 |
| 44214 | 0.560 | 0.348 | 0.529 |
| 44215 | 0.535 | 0.168 | 0.422 |
| 44221 | 0.583 | 0.494 | 0.630 |
| 44222 | 0.533 | 0.438 | 0.570 |
| 44223 | 0.520 | 0.423 | 0.554 |
| 44224 | 0.496 | 0.249 | 0.459 |
| 44225 | 0.471 | 0.069 | 0.361 |
| 44231 | 0.567 | 0.470 | 0.615 |
| 44232 | 0.517 | 0.413 | 0.551 |
| 44233 | 0.504 | 0.399 | 0.535 |
| 44234 | 0.480 | 0.225 | 0.442 |
| 44235 | 0.455 | 0.045 | 0.346 |
| 44241 | 0.522 | 0.289 | 0.503 |
| 44242 | 0.472 | 0.233 | 0.446 |
| 44243 | 0.459 | 0.218 | 0.431 |
| 44244 | 0.435 | 0.082 | 0.355 |
| 44245 | 0.410 | -0.060 | 0.276 |
| 44251 | 0.453 | 0.018 | 0.335 |
| 44252 | 0.403 | -0.039 | 0.288 |
| 44253 | 0.390 | -0.053 | 0.276 |
| 44254 | 0.366 | -0.134 | 0.224 |
| 44255 | 0.341 | -0.218 | 0.170 |
| 44311<br>44312 | 0.639 | 0.586 | 0.686 |
| | 0.589 | 0.529 | 0.636 |
| 44313 | 0.576 | 0.515 | 0.622 |
| 44314 | 0.552 | 0.341 | 0.521 |
| 44315 | 0.527 | 0.161 | 0.417 |
| 44321 | 0.575 | 0.487 | 0.622 |
| 44322 | 0.525 | 0.431 | 0.558 |
| 44323 | 0.512 | 0.416 | 0.541 |
| 44324<br>44325 | 0.488 | 0.242 | 0.449 |
| 44325 | 0.463<br>0.559 | 0.062<br>0.463 | 0.352<br>0.606 |
| 44331 | 0.559 | 0.403 | 0.000 |

| 44332 | 0.509 | 0.406 | 0.539 |
|-------|-------|--------|-------|
| 44333 | 0.496 | 0.392 | 0.521 |
| 44334 | 0.472 | 0.218 | 0.430 |
| 44335 | 0.447 | 0.038 | 0.336 |
| 44341 | 0.513 | 0.282 | 0.496 |
| 44342 | 0.463 | 0.226 | 0.435 |
| 44343 | 0.450 | 0.211 | 0.419 |
| 44344 | 0.426 | 0.074 | 0.345 |
| 44345 | 0.401 | -0.068 | 0.268 |
| 44351 | 0.445 | 0.011 | 0.330 |
| 44352 | 0.395 | -0.046 | 0.279 |
| 44353 | 0.382 | -0.060 | 0.266 |
| 44354 | 0.358 | -0.141 | 0.217 |
| 44355 | 0.333 | -0.225 | 0.165 |
| 44411 | 0.609 | 0.504 | 0.631 |
| 44412 | 0.559 | 0.448 | 0.586 |
| 44413 | 0.546 | 0.433 | 0.574 |
| 44414 | 0.522 | 0.290 | 0.487 |
| 44415 | 0.497 | 0.142 | 0.396 |
| 44421 | 0.545 | 0.406 | 0.572 |
| 44422 | 0.495 | 0.350 | 0.514 |
| 44423 | 0.482 | 0.335 | 0.499 |
| 44424 | 0.458 | 0.192 | 0.419 |
| 44425 | 0.433 | 0.043 | 0.337 |
| 44431 | 0.529 | 0.381 | 0.558 |
| 44432 | 0.479 | 0.325 | 0.496 |
| 44433 | 0.466 | 0.310 | 0.480 |
| 44434 | 0.442 | 0.167 | 0.403 |
| 44435 | 0.417 | 0.019 | 0.322 |
| 44441 | 0.484 | 0.226 | 0.458 |
| 44442 | 0.434 | 0.169 | 0.403 |
| 44443 | 0.421 | 0.155 | 0.389 |
| 44444 | 0.397 | 0.036 | 0.323 |
| 44445 | 0.372 | -0.087 | 0.255 |
| 44451 | 0.415 | -0.009 | 0.309 |
| 44452 | 0.365 | -0.065 | 0.264 |
| 44453 | 0.352 | -0.080 | 0.252 |
| 44454 | 0.328 | -0.160 | 0.204 |
| 44455 | 0.303 | -0.245 | 0.154 |
| 44511 | 0.550 | 0.339 | 0.518 |
| 44512 | 0.500 | 0.282 | 0.485 |
| 44513 | 0.487 | 0.268 | 0.476 |
| 44514 | 0.463 | 0.187 | 0.416 |
| 44515 | 0.438 | 0.103 | 0.353 |
| 44521 | 0.486 | 0.240 | 0.471 |
| 44522 | 0.436 | 0.184 | 0.424 |
| 44523 | 0.423 | 0.169 | 0.411 |
| 44524 | 0.399 | 0.088 | 0.360 |
| 44525 | 0.374 | 0.004 | 0.306 |

| 44531 | 0.470 | 0.216 | 0.460 |
|-------|-------|--------|-------|
| 44532 | 0.420 | 0.159 | 0.409 |
| 44533 | 0.407 | 0.145 | 0.395 |
| 44534 | 0.383 | 0.064 | 0.346 |
| 44535 | 0.358 | -0.020 | 0.294 |
| 44541 | 0.424 | 0.111 | 0.382 |
| 44542 | 0.374 | 0.054 | 0.338 |
| 44543 | 0.361 | 0.040 | 0.327 |
| 44544 | 0.337 | -0.041 | 0.279 |
| 44545 | 0.312 | -0.126 | 0.229 |
| 44551 | 0.356 | -0.047 | 0.266 |
| 44552 | 0.306 | -0.104 | 0.233 |
| 44553 | 0.293 | -0.118 | 0.224 |
| 44554 | 0.269 | -0.199 | 0.178 |
| 44555 | 0.244 | -0.283 | 0.131 |
| 45111 | 0.646 | 0.349 | 0.502 |
| 45112 | 0.596 | 0.293 | 0.481 |
| 45113 | 0.583 | 0.278 | 0.476 |
| 45114 | 0.559 | 0.197 | 0.404 |
| 45115 | 0.534 | 0.113 | 0.330 |
| 45121 | 0.582 | 0.251 | 0.468 |
| 45122 | 0.532 | 0.195 | 0.434 |
| 45123 | 0.519 | 0.180 | 0.425 |
| 45124 | 0.495 | 0.099 | 0.362 |
| 45125 | 0.470 | 0.015 | 0.296 |
| 45131 | 0.566 | 0.226 | 0.459 |
| 45132 | 0.516 | 0.170 | 0.422 |
| 45133 | 0.503 | 0.155 | 0.412 |
| 45134 | 0.479 | 0.074 | 0.351 |
| 45135 | 0.454 | -0.010 | 0.287 |
| 45141 | 0.521 | 0.121 | 0.373 |
| 45142 | 0.471 | 0.065 | 0.342 |
| 45143 | 0.458 | 0.050 | 0.334 |
| 45144 | 0.434 | -0.031 | 0.275 |
| 45145 | 0.409 | -0.115 | 0.213 |
| 45151 | 0.452 | -0.037 | 0.243 |
| 45152 | 0.402 | -0.093 | 0.223 |
| 45153 | 0.389 | -0.108 | 0.217 |
| 45154 | 0.365 | -0.189 | 0.160 |
| 45155 | 0.340 | -0.273 | 0.101 |
| 45211 | 0.611 | 0.321 | 0.495 |
| 45212 | 0.561 | 0.264 | 0.460 |
| 45213 | 0.548 | 0.250 | 0.452 |
| 45214 | 0.524 | 0.169 | 0.388 |
| 45215 | 0.499 | 0.085 | 0.322 |
| 45221 | 0.547 | 0.222 | 0.447 |
| 45222 | 0.497 | 0.166 | 0.399 |
| 45223 | 0.484 | 0.151 | 0.387 |
| 45224 | 0.460 | 0.070 | 0.332 |

| 45225 | 0.435 | -0.014 | 0.274 |
|-------|-------|--------|-------|
| 45231 | 0.531 | 0.198 | 0.435 |
| 45232 | 0.481 | 0.141 | 0.384 |
| 45233 | 0.468 | 0.127 | 0.370 |
| 45234 | 0.444 | 0.046 | 0.318 |
| 45235 | 0.419 | -0.039 | 0.263 |
| 45241 | 0.485 | 0.092 | 0.355 |
| 45242 | 0.435 | 0.036 | 0.311 |
| 45243 | 0.422 | 0.021 | 0.299 |
| 45244 | 0.398 | -0.060 | 0.248 |
| 45245 | 0.373 | -0.144 | 0.195 |
| 45251 | 0.417 | -0.066 | 0.235 |
| 45252 | 0.367 | -0.122 | 0.201 |
| 45253 | 0.354 | -0.137 | 0.193 |
| 45254 | 0.330 | -0.218 | 0.144 |
| 45255 | 0.305 | -0.302 | 0.093 |
| 45311 | 0.602 | 0.313 | 0.493 |
| 45312 | 0.552 | 0.257 | 0.455 |
| 45313 | 0.539 | 0.242 | 0.446 |
| 45314 | 0.515 | 0.161 | 0.384 |
| 45315 | 0.490 | 0.077 | 0.320 |
| 45321 | 0.538 | 0.215 | 0.441 |
| 45322 | 0.488 | 0.159 | 0.390 |
| 45323 | 0.475 | 0.144 | 0.377 |
| 45324 | 0.451 | 0.063 | 0.324 |
| 45325 | 0.426 | -0.021 | 0.269 |
| 45331 | 0.522 | 0.190 | 0.429 |
| 45332 | 0.472 | 0.134 | 0.374 |
| 45333 | 0.459 | 0.119 | 0.360 |
| 45334 | 0.435 | 0.038 | 0.309 |
| 45335 | 0.410 | -0.046 | 0.257 |
| 45341 | 0.477 | 0.085 | 0.350 |
| 45342 | 0.427 | 0.029 | 0.303 |
| 45343 | 0.414 | 0.014 | 0.291 |
| 45344 | 0.390 | -0.067 | 0.242 |
| 45345 | 0.365 | -0.151 | 0.191 |
| 45351 | 0.408 | -0.073 | 0.233 |
| 45352 | 0.358 | -0.129 | 0.196 |
| 45353 | 0.345 | -0.144 | 0.187 |
| 45354 | 0.321 | -0.225 | 0.140 |
| 45355 | 0.296 | -0.309 | 0.091 |
| 45411 | 0.573 | 0.294 | 0.464 |
| 45412 | 0.523 | 0.238 | 0.432 |
| 45413 | 0.510 | 0.223 | 0.424 |
| 45414 | 0.486 | 0.142 | 0.364 |
| 45415 | 0.461 | 0.058 | 0.302 |
| 45421 | 0.509 | 0.196 | 0.418 |
| 45422 | 0.459 | 0.139 | 0.373 |
| 45423 | 0.446 | 0.125 | 0.361 |

| 45424 | 0.422 | 0.044 | 0.310 |
|----------------|----------------|------------------|----------------|
| 45425 | 0.397 | -0.040 | 0.256 |
| 45431 | 0.493 | 0.171 | 0.407 |
| 45432 | 0.443 | 0.115 | 0.358 |
| 45433 | 0.430 | 0.100 | 0.345 |
| 45434 | 0.406 | 0.019 | 0.296 |
| 45435 | 0.381 | -0.065 | 0.245 |
| 45441 | 0.448 | 0.066 | 0.330 |
| 45442 | 0.398 | 0.010 | 0.288 |
| 45443 | 0.385 | -0.005 | 0.277 |
| 45444 | 0.360 | -0.086 | 0.229 |
| 45445 | 0.336 | -0.170 | 0.180 |
| 45451 | 0.379 | -0.092 | 0.215 |
| 45452 | 0.329 | -0.148 | 0.183 |
| 45453 | 0.316 | -0.163 | 0.175 |
| 45454 | 0.292 | -0.244 | 0.129 |
| 45455 | 0.267 | -0.328 | 0.082 |
| 45511 | 0.513 | 0.255 | 0.406 |
| 45512 | 0.463 | 0.199 | 0.386 |
| 45513 | 0.450 | 0.184 | 0.380 |
| 45514 | 0.426 | 0.103 | 0.323 |
| 45515 | 0.401 | 0.019 | 0.263 |
| 45521 | 0.449 | 0.157 | 0.372 |
| 45522 | 0.399 | 0.101 | 0.337 |
| 45523 | 0.386 | 0.086 | 0.328 |
| 45524 | 0.362 | 0.005 | 0.280 |
| 45525 | 0.337 | -0.079 | 0.229 |
| 45531 | 0.433 | 0.132 | 0.363 |
| 45532 | 0.383 | 0.076 | 0.325 |
| 45533 | 0.370 | 0.061 | 0.316 |
| 45534 | 0.346 | -0.020 | 0.269 |
| 45535 | 0.321 | -0.104 | 0.220 |
| 45541 | 0.388 | 0.027 | 0.289 |
| 45542 | 0.338 | -0.029 | 0.258 |
| 45543 | 0.325 | -0.044 | 0.250 |
| 45544 | 0.301 | -0.125 | 0.205 |
| 45545 | 0.276 | -0.209 | 0.158 |
| 45551<br>45552 | 0.319<br>0.269 | -0.131<br>-0.187 | 0.177<br>0.156 |
| 45552 | 0.259 | | 0.150 |
| 45554 | | -0.202 | 0.130 |
| | 0.232 | -0.283 | 0.100 |
| 45555<br>51111 | 0.207<br>0.430 | -0.367<br>0.336 | 0.064 |
| 51111 | 0.430 | 0.336 | 0.442 |
| 51112 | 0.367 | 0.265 | 0.429 |
| 51113 | 0.367 | 0.265 | 0.426 |
| 51114 | 0.343 | 0.104 | 0.349 |
| 51113 | 0.366 | 0.100 | 0.200 |
| 51121 | 0.316 | 0.236 | 0.416 |
| 01122 | 0.510 | 0.101 | 0.580 |

| = | | | |
|----------------|----------------|----------------|----------------|
| 51123 | 0.303 | 0.167 | 0.391 |
| 51124 | 0.279 | 0.086 | 0.318 |
| 51125 | 0.254 | 0.002 | 0.242 |
| 51131 | 0.350 | 0.213 | 0.409 |
| 51132 | 0.300 | 0.157 | 0.388 |
| 51133 | 0.287 | 0.142 | 0.382 |
| 51134 | 0.263 | 0.061 | 0.310 |
| 51135 | 0.238 | -0.023 | 0.235 |
| 51141 | 0.305 | 0.108 | 0.318 |
| 51142 | 0.255 | 0.052 | 0.300 |
| 51143 | 0.242 | 0.037 | 0.295 |
| 51144 | 0.217 | -0.044 | 0.227 |
| 51145 | 0.193 | -0.128 | 0.156 |
| 51151 | 0.236 | -0.050 | 0.181 |
| 51152 | 0.186 | -0.106 | 0.168 |
| 51153 | 0.173 | -0.121 | 0.165 |
| 51154 | 0.149 | -0.202 | 0.102 |
| 51155 | 0.124 | -0.286 | 0.037 |
| 51211 | 0.395 | 0.307 | 0.442 |
| 51212 | 0.345 | 0.251 | 0.422 |
| 51213 | 0.332 | 0.236 | 0.417 |
| 51214 | 0.308 | 0.155 | 0.344 |
| 51215 | 0.283 | 0.071 | 0.268 |
| 51221 | 0.331 | 0.209 | 0.409 |
| 51222 | 0.281 | 0.152 | 0.377 |
| 51223 | 0.268 | 0.138 | 0.368 |
| 51224 | 0.244 | 0.057 | 0.303 |
| 51225 | 0.219 | -0.027 | 0.235 |
| 51231 | 0.315 | 0.184 | 0.400 |
| 51232 | 0.265 | 0.128 | 0.365 |
| 51233 | 0.252 | 0.113 | 0.356 |
| 51234 | 0.228<br>0.203 | 0.032 | 0.293 |
| 51235 | | -0.052 | 0.226 |
| 51241<br>51242 | 0.269 | 0.079<br>0.023 | 0.313 |
| 51242 | 0.219<br>0.206 | 0.023 | 0.284<br>0.276 |
| 51243 | 0.200 | -0.073 | 0.276 |
| 51244 | 0.152 | -0.073 | 0.213 |
| 51245 | 0.137 | -0.157 | 0.130 |
| 51251 | 0.201 | -0.079 | 0.161 |
| 51252 | 0.131 | -0.150 | 0.156 |
| 51253 | 0.138 | -0.130 | 0.130 |
| 51254 | 0.089 | -0.231 | 0.036 |
| 51255 | 0.089 | 0.300 | 0.442 |
| 51311 | 0.336 | 0.300 | 0.442 |
| 51312 | 0.323 | 0.229 | 0.421 |
| 51314 | 0.323 | 0.148 | 0.343 |
| 51315 | 0.274 | 0.064 | 0.268 |
| 51321 | 0.322 | 0.202 | 0.407 |
| 31021 | U.ULL | 0.202 | 0.401 |

| 51322 | 0.272 | 0.145 | 0.372 |
|-------|-------|--------|-------|
| 51323 | 0.259 | 0.131 | 0.363 |
| 51324 | 0.235 | 0.050 | 0.299 |
| 51325 | 0.210 | -0.035 | 0.233 |
| 51331 | 0.306 | 0.177 | 0.398 |
| 51332 | 0.256 | 0.121 | 0.360 |
| 51333 | 0.243 | 0.106 | 0.350 |
| 51334 | 0.219 | 0.025 | 0.288 |
| 51335 | 0.194 | -0.059 | 0.224 |
| 51341 | 0.261 | 0.072 | 0.311 |
| 51342 | 0.211 | 0.016 | 0.280 |
| 51343 | 0.198 | 0.001 | 0.272 |
| 51344 | 0.173 | -0.080 | 0.211 |
| 51345 | 0.149 | -0.164 | 0.149 |
| 51351 | 0.192 | -0.086 | 0.181 |
| 51352 | 0.142 | -0.142 | 0.160 |
| 51353 | 0.129 | -0.157 | 0.154 |
| 51354 | 0.105 | -0.238 | 0.096 |
| 51355 | 0.080 | -0.322 | 0.036 |
| 51411 | 0.357 | 0.281 | 0.410 |
| 51412 | 0.307 | 0.225 | 0.391 |
| 51413 | 0.294 | 0.210 | 0.386 |
| 51414 | 0.270 | 0.129 | 0.317 |
| 51415 | 0.245 | 0.045 | 0.245 |
| 51421 | 0.293 | 0.182 | 0.378 |
| 51422 | 0.243 | 0.126 | 0.347 |
| 51423 | 0.230 | 0.111 | 0.340 |
| 51424 | 0.206 | 0.030 | 0.277 |
| 51425 | 0.181 | -0.054 | 0.213 |
| 51431 | 0.277 | 0.158 | 0.369 |
| 51432 | 0.227 | 0.102 | 0.337 |
| 51433 | 0.214 | 0.087 | 0.328 |
| 51434 | 0.190 | 0.006 | 0.268 |
| 51435 | 0.165 | -0.078 | 0.205 |
| 51441 | 0.231 | 0.053 | 0.285 |
| 51442 | 0.181 | -0.003 | 0.258 |
| 51443 | 0.168 | -0.018 | 0.251 |
| 51444 | 0.144 | -0.099 | 0.193 |
| 51445 | 0.119 | -0.183 | 0.132 |
| 51451 | 0.163 | -0.105 | 0.158 |
| 51452 | 0.113 | -0.161 | 0.140 |
| 51453 | 0.100 | -0.176 | 0.135 |
| 51454 | 0.076 | -0.257 | 0.080 |
| 51455 | 0.051 | -0.341 | 0.023 |
| 51511 | 0.297 | 0.242 | 0.344 |
| 51512 | 0.247 | 0.186 | 0.331 |
| 51513 | 0.234 | 0.171 | 0.327 |
| 51514 | 0.210 | 0.090 | 0.264 |
| 51515 | 0.185 | 0.006 | 0.199 |

| 51521 | 0.233 | 0.144 | 0.318 |
|-------|--------|--------|--------|
| 51522 | 0.183 | 0.087 | 0.297 |
| 51523 | 0.170 | 0.073 | 0.292 |
| 51524 | 0.146 | -0.009 | 0.233 |
| 51525 | 0.121 | -0.093 | 0.173 |
| 51531 | 0.217 | 0.119 | 0.311 |
| 51532 | 0.167 | 0.063 | 0.289 |
| 51533 | 0.154 | 0.048 | 0.283 |
| 51534 | 0.130 | -0.033 | 0.226 |
| 51535 | 0.105 | -0.117 | 0.166 |
| 51541 | 0.172 | 0.014 | 0.232 |
| 51542 | 0.122 | -0.042 | 0.213 |
| 51543 | 0.109 | -0.057 | 0.208 |
| 51544 | 0.084 | -0.138 | 0.154 |
| 51545 | 0.060 | -0.222 | 0.099 |
| 51551 | 0.103 | -0.144 | 0.112 |
| 51552 | 0.053 | -0.200 | 0.099 |
| 51553 | 0.040 | -0.215 | 0.096 |
| 51554 | 0.016 | -0.296 | 0.047 |
| 51555 | -0.009 | -0.380 | -0.003 |
| 52111 | 0.385 | 0.249 | 0.413 |
| 52112 | 0.335 | 0.193 | 0.392 |
| 52113 | 0.322 | 0.178 | 0.387 |
| 52114 | 0.298 | 0.097 | 0.314 |
| 52115 | 0.273 | 0.013 | 0.238 |
| 52121 | 0.321 | 0.151 | 0.379 |
| 52122 | 0.271 | 0.095 | 0.346 |
| 52123 | 0.258 | 0.080 | 0.338 |
| 52124 | 0.234 | -0.001 | 0.272 |
| 52125 | 0.209 | -0.085 | 0.204 |
| 52131 | 0.305 | 0.126 | 0.371 |
| 52132 | 0.255 | 0.070 | 0.335 |
| 52133 | 0.242 | 0.055 | 0.325 |
| 52134 | 0.218 | -0.026 | 0.262 |
| 52135 | 0.193 | -0.110 | 0.196 |
| 52141 | 0.260 | 0.021 | 0.283 |
| 52142 | 0.210 | -0.035 | 0.253 |
| 52143 | 0.197 | -0.050 | 0.246 |
| 52144 | 0.173 | -0.131 | 0.184 |
| 52145 | 0.148 | -0.215 | 0.120 |
| 52151 | 0.191 | -0.137 | 0.151 |
| 52152 | 0.141 | -0.193 | 0.131 |
| 52153 | 0.128 | -0.208 | 0.126 |
| 52154 | 0.104 | -0.289 | 0.068 |
| 52155 | 0.079 | -0.373 | 0.007 |
| 52211 | 0.350 | 0.221 | 0.406 |
| 52212 | 0.300 | 0.164 | 0.373 |
| 52213 | 0.287 | 0.150 | 0.364 |
| 52214 | 0.263 | 0.069 | 0.299 |

| 52215 | 0.238 | -0.016 | 0.231 |
|-------|-------|--------|--------|
| 52221 | 0.286 | 0.122 | 0.359 |
| 52222 | 0.236 | 0.066 | 0.313 |
| 52223 | 0.223 | 0.051 | 0.301 |
| 52224 | 0.199 | -0.030 | 0.244 |
| 52225 | 0.174 | -0.114 | 0.185 |
| 52231 | 0.270 | 0.098 | 0.347 |
| 52232 | 0.220 | 0.041 | 0.298 |
| 52233 | 0.207 | 0.027 | 0.285 |
| 52234 | 0.183 | -0.054 | 0.230 |
| 52235 | 0.158 | -0.139 | 0.173 |
| 52241 | 0.224 | -0.008 | 0.266 |
| 52242 | 0.174 | -0.064 | 0.223 |
| 52243 | 0.161 | -0.079 | 0.212 |
| 52244 | 0.137 | -0.160 | 0.159 |
| 52245 | 0.112 | -0.244 | 0.104 |
| 52251 | 0.156 | -0.166 | 0.144 |
| 52252 | 0.106 | -0.222 | 0.112 |
| 52253 | 0.093 | -0.237 | 0.103 |
| 52254 | 0.069 | -0.317 | 0.052 |
| 52255 | 0.044 | -0.402 | -0.001 |
| 52311 | 0.341 | 0.213 | 0.404 |
| 52312 | 0.291 | 0.157 | 0.368 |
| 52313 | 0.278 | 0.142 | 0.358 |
| 52314 | 0.254 | 0.061 | 0.295 |
| 52315 | 0.229 | -0.023 | 0.230 |
| 52321 | 0.277 | 0.115 | 0.354 |
| 52322 | 0.227 | 0.059 | 0.305 |
| 52323 | 0.214 | 0.044 | 0.292 |
| 52324 | 0.190 | -0.037 | 0.237 |
| 52325 | 0.165 | -0.121 | 0.180 |
| 52331 | 0.261 | 0.090 | 0.341 |
| 52332 | 0.211 | 0.034 | 0.289 |
| 52333 | 0.198 | 0.019 | 0.275 |
| 52334 | 0.174 | -0.062 | 0.222 |
| 52335 | 0.149 | -0.146 | 0.167 |
| 52341 | 0.216 | -0.015 | 0.262 |
| 52342 | 0.166 | -0.071 | 0.216 |
| 52343 | 0.153 | -0.086 | 0.204 |
| 52344 | 0.129 | -0.167 | 0.153 |
| 52345 | 0.104 | -0.251 | 0.100 |
| 52351 | 0.147 | -0.173 | 0.143 |
| 52352 | 0.097 | -0.229 | 0.107 |
| 52353 | 0.084 | -0.244 | 0.097 |
| 52354 | 0.060 | -0.325 | 0.049 |
| 52355 | 0.035 | -0.409 | -0.002 |
| 52411 | 0.312 | 0.194 | 0.374 |
| 52412 | 0.262 | 0.138 | 0.344 |
| 52413 | 0.249 | 0.123 | 0.336 |

| 52414 | 0.225 | 0.042 | 0.274 |
|-------|--------|--------|--------|
| 52415 | 0.200 | -0.042 | 0.210 |
| 52421 | 0.248 | 0.096 | 0.330 |
| 52422 | 0.198 | 0.040 | 0.286 |
| 52423 | 0.185 | 0.025 | 0.275 |
| 52424 | 0.161 | -0.056 | 0.221 |
| 52425 | 0.136 | -0.140 | 0.165 |
| 52431 | 0.232 | 0.071 | 0.319 |
| 52432 | 0.182 | 0.015 | 0.272 |
| 52433 | 0.169 | 0.000 | 0.259 |
| 52434 | 0.145 | -0.081 | 0.208 |
| 52435 | 0.120 | -0.165 | 0.154 |
| 52441 | 0.186 | -0.034 | 0.240 |
| 52442 | 0.136 | -0.090 | 0.200 |
| 52443 | 0.123 | -0.105 | 0.189 |
| 52444 | 0.099 | -0.186 | 0.140 |
| 52445 | 0.074 | -0.270 | 0.088 |
| 52451 | 0.118 | -0.192 | 0.123 |
| 52452 | 0.068 | -0.248 | 0.092 |
| 52453 | 0.055 | -0.263 | 0.084 |
| 52454 | 0.031 | -0.344 | 0.037 |
| 52455 | 0.006 | -0.428 | -0.012 |
| 52511 | 0.252 | 0.155 | 0.314 |
| 52512 | 0.202 | 0.099 | 0.294 |
| 52513 | 0.189 | 0.084 | 0.289 |
| 52514 | 0.165 | 0.003 | 0.230 |
| 52515 | 0.140 | -0.081 | 0.170 |
| 52521 | 0.188 | 0.057 | 0.280 |
| 52522 | 0.138 | 0.001 | 0.248 |
| 52523 | 0.125 | -0.014 | 0.239 |
| 52524 | 0.101 | -0.095 | 0.189 |
| 52525 | 0.076 | -0.179 | 0.136 |
| 52531 | 0.172 | 0.032 | 0.272 |
| 52532 | 0.122 | -0.024 | 0.236 |
| 52533 | 0.109 | -0.039 | 0.227 |
| 52534 | 0.085 | -0.120 | 0.178 |
| 52535 | 0.060 | -0.204 | 0.128 |
| 52541 | 0.127 | -0.073 | 0.196 |
| 52542 | 0.077 | -0.129 | 0.167 |
| 52543 | 0.064 | -0.144 | 0.159 |
| 52544 | 0.040 | -0.225 | 0.112 |
| 52545 | 0.015 | -0.309 | 0.064 |
| 52551 | 0.058 | -0.231 | 0.083 |
| 52552 | 0.008 | -0.287 | 0.062 |
| 52553 | -0.005 | -0.302 | 0.057 |
| 52554 | -0.029 | -0.383 | 0.013 |
| 52555 | -0.054 | -0.467 | -0.032 |
| 53111 | 0.376 | 0.232 | 0.407 |
| 53112 | 0.326 | 0.176 | 0.385 |

| 53113 | 0.313 | 0.161 | 0.379 |
|-------|-------|--------|--------|
| 53114 | 0.289 | 0.080 | 0.307 |
| 53115 | 0.264 | -0.004 | 0.232 |
| 53121 | 0.312 | 0.134 | 0.372 |
| 53122 | 0.262 | 0.077 | 0.336 |
| 53123 | 0.249 | 0.063 | 0.327 |
| 53124 | 0.225 | -0.019 | 0.263 |
| 53125 | 0.200 | -0.103 | 0.197 |
| 53131 | 0.296 | 0.109 | 0.363 |
| 53132 | 0.246 | 0.053 | 0.324 |
| 53133 | 0.233 | 0.038 | 0.314 |
| 53134 | 0.209 | -0.043 | 0.252 |
| 53135 | 0.184 | -0.127 | 0.188 |
| 53141 | 0.251 | 0.004 | 0.276 |
| 53142 | 0.201 | -0.052 | 0.244 |
| 53143 | 0.188 | -0.067 | 0.236 |
| 53144 | 0.163 | -0.148 | 0.176 |
| 53145 | 0.139 | -0.232 | 0.113 |
| 53151 | 0.182 | -0.154 | 0.145 |
| 53152 | 0.132 | -0.210 | 0.124 |
| 53153 | 0.119 | -0.225 | 0.118 |
| 53154 | 0.095 | -0.306 | 0.061 |
| 53155 | 0.070 | -0.390 | 0.001 |
| 53211 | 0.341 | 0.203 | 0.398 |
| 53212 | 0.291 | 0.147 | 0.363 |
| 53213 | 0.278 | 0.132 | 0.353 |
| 53214 | 0.254 | 0.051 | 0.290 |
| 53215 | 0.229 | -0.033 | 0.224 |
| 53221 | 0.277 | 0.105 | 0.349 |
| 53222 | 0.227 | 0.048 | 0.300 |
| 53223 | 0.214 | 0.034 | 0.287 |
| 53224 | 0.190 | -0.047 | 0.232 |
| 53225 | 0.165 | -0.131 | 0.175 |
| 53231 | 0.261 | 0.080 | 0.337 |
| 53232 | 0.211 | 0.024 | 0.284 |
| 53233 | 0.198 | 0.009 | 0.271 |
| 53234 | 0.174 | -0.072 | 0.218 |
| 53235 | 0.149 | -0.156 | 0.162 |
| 53241 | 0.215 | -0.025 | 0.257 |
| 53242 | 0.165 | -0.081 | 0.211 |
| 53243 | 0.152 | -0.096 | 0.199 |
| 53244 | 0.128 | -0.177 | 0.148 |
| 53245 | 0.103 | -0.261 | 0.094 |
| 53251 | 0.147 | -0.183 | 0.137 |
| 53252 | 0.097 | -0.239 | 0.102 |
| 53253 | 0.084 | -0.254 | 0.092 |
| 53254 | 0.060 | -0.335 | 0.043 |
| 53255 | 0.035 | -0.419 | -0.008 |
| 53311 | 0.332 | 0.196 | 0.396 |

| 53312 | 0.282 | 0.140 | 0.357 |
|-------|--------|----------------|--------|
| 53313 | 0.269 | 0.125 | 0.347 |
| 53314 | 0.245 | 0.044 | 0.286 |
| 53315 | 0.220 | -0.040 | 0.222 |
| 53321 | 0.268 | 0.098 | 0.343 |
| 53322 | 0.218 | 0.041 | 0.291 |
| 53323 | 0.205 | 0.027 | 0.277 |
| 53324 | 0.181 | -0.055 | 0.224 |
| 53325 | 0.156 | -0.139 | 0.169 |
| 53331 | 0.252 | 0.073 | 0.330 |
| 53332 | 0.202 | 0.017 | 0.275 |
| 53333 | 0.189 | 0.002 | 0.260 |
| 53334 | 0.165 | -0.079 | 0.209 |
| 53335 | 0.140 | -0.163 | 0.156 |
| 53341 | 0.207 | -0.032 | 0.252 |
| 53342 | 0.157 | -0.088 | 0.203 |
| 53343 | 0.144 | -0.103 | 0.191 |
| 53344 | 0.119 | -0.184 | 0.141 |
| 53345 | 0.095 | -0.268 | 0.090 |
| 53351 | 0.138 | -0.190 | 0.135 |
| 53352 | 0.088 | -0.246 | 0.096 |
| 53353 | 0.075 | -0.261 | 0.086 |
| 53354 | 0.051 | -0.342 | 0.039 |
| 53355 | 0.026 | -0.426 | -0.010 |
| 53411 | 0.303 | 0.177 | 0.367 |
| 53412 | 0.253 | 0.121 | 0.334 |
| 53413 | 0.240 | 0.106 | 0.325 |
| 53414 | 0.216 | 0.025 | 0.265 |
| 53415 | 0.191 | -0.059 | 0.203 |
| 53421 | 0.239 | 0.078 | 0.320 |
| 53422 | 0.189 | 0.022 | 0.274 |
| 53423 | 0.176 | 0.007 | 0.261 |
| 53424 | 0.152 | -0.074 | 0.210 |
| 53425 | 0.127 | -0.158 | 0.156 |
| 53431 | 0.223 | 0.054 | 0.308 |
| 53432 | 0.173 | -0.002 | 0.259 |
| 53433 | 0.160 | -0.017 | 0.246 |
| 53434 | 0.136 | -0.098 | 0.196 |
| 53435 | 0.111 | -0.182 | 0.144 |
| 53441 | 0.177 | -0.051 | 0.232 |
| 53442 | 0.127 | -0.107 | 0.188 |
| 53443 | 0.114 | -0.122 | 0.177 |
| 53444 | 0.090 | -0.203 | 0.129 |
| 53445 | 0.065 | -0.287 | 0.079 |
| 53451 | 0.109 | -0.209 | 0.116 |
| 53452 | 0.059 | -0.265 | 0.083 |
| 53453 | 0.046 | -0.280 | 0.074 |
| 53454 | 0.022 | -0.361 | 0.028 |
| 53455 | -0.003 | <b>-0</b> .445 | -0.019 |

| 53511 | 0.243 | 0.138 | 0.308 |
|-------|--------|--------|--------|
| 53512 | 0.193 | 0.082 | 0.287 |
| 53513 | 0.180 | 0.067 | 0.281 |
| 53514 | 0.156 | -0.014 | 0.224 |
| 53515 | 0.131 | -0.098 | 0.164 |
| 53521 | 0.179 | 0.040 | 0.273 |
| 53522 | 0.129 | -0.017 | 0.238 |
| 53523 | 0.116 | -0.032 | 0.229 |
| 53524 | 0.092 | -0.113 | 0.180 |
| 53525 | 0.067 | -0.197 | 0.129 |
| 53531 | 0.163 | 0.015 | 0.264 |
| 53532 | 0.113 | -0.041 | 0.226 |
| 53533 | 0.100 | -0.056 | 0.216 |
| 53534 | 0.076 | -0.137 | 0.169 |
| 53535 | 0.051 | -0.221 | 0.120 |
| 53541 | 0.118 | -0.090 | 0.189 |
| 53542 | 0.068 | -0.146 | 0.158 |
| 53543 | 0.055 | -0.161 | 0.149 |
| 53544 | 0.030 | -0.242 | 0.104 |
| 53545 | 0.006 | -0.326 | 0.057 |
| 53551 | 0.049 | -0.248 | 0.077 |
| 53552 | -0.001 | -0.304 | 0.055 |
| 53553 | -0.014 | -0.319 | 0.049 |
| 53554 | -0.038 | -0.400 | 0.006 |
| 53555 | -0.063 | -0.484 | -0.038 |
| 54111 | 0.364 | 0.205 | 0.368 |
| 54112 | 0.314 | 0.149 | 0.348 |
| 54113 | 0.301 | 0.134 | 0.343 |
| 54114 | 0.277 | 0.053 | 0.273 |
| 54115 | 0.252 | -0.031 | 0.200 |
| 54121 | 0.300 | 0.107 | 0.335 |
| 54122 | 0.250 | 0.050 | 0.303 |
| 54123 | 0.237 | 0.036 | 0.295 |
| 54124 | 0.213 | -0.045 | 0.232 |
| 54125 | 0.188 | -0.129 | 0.167 |
| 54131 | 0.284 | 0.082 | 0.327 |
| 54132 | 0.234 | 0.026 | 0.292 |
| 54133 | 0.221 | 0.011 | 0.283 |
| 54134 | 0.197 | -0.070 | 0.222 |
| 54135 | 0.172 | -0.154 | 0.159 |
| 54141 | 0.239 | -0.023 | 0.242 |
| 54142 | 0.189 | -0.079 | 0.213 |
| 54143 | 0.176 | -0.094 | 0.206 |
| 54144 | 0.152 | -0.175 | 0.147 |
| 54145 | 0.127 | -0.259 | 0.086 |
| 54151 | 0.170 | -0.181 | 0.114 |
| 54152 | 0.120 | -0.237 | 0.094 |
| 54153 | 0.107 | -0.252 | 0.089 |
| 54154 | 0.083 | -0.333 | 0.034 |

| 54155 | 0.058 | -0.417 | -0.024 |
|-------|-------|--------|--------|
| 54211 | 0.329 | 0.176 | 0.361 |
| 54212 | 0.279 | 0.120 | 0.330 |
| 54213 | 0.266 | 0.105 | 0.321 |
| 54214 | 0.242 | 0.024 | 0.259 |
| 54215 | 0.217 | -0.060 | 0.194 |
| 54221 | 0.265 | 0.078 | 0.316 |
| 54222 | 0.215 | 0.022 | 0.271 |
| 54223 | 0.202 | 0.007 | 0.259 |
| 54224 | 0.178 | -0.074 | 0.205 |
| 54225 | 0.153 | -0.158 | 0.149 |
| 54231 | 0.249 | 0.053 | 0.305 |
| 54232 | 0.199 | -0.003 | 0.256 |
| 54233 | 0.186 | -0.018 | 0.244 |
| 54234 | 0.162 | -0.099 | 0.192 |
| 54235 | 0.137 | -0.183 | 0.138 |
| 54241 | 0.204 | -0.052 | 0.226 |
| 54242 | 0.154 | -0.108 | 0.184 |
| 54243 | 0.141 | -0.123 | 0.173 |
| 54244 | 0.117 | -0.204 | 0.123 |
| 54245 | 0.092 | -0.288 | 0.071 |
| 54251 | 0.135 | -0.210 | 0.107 |
| 54252 | 0.085 | -0.266 | 0.076 |
| 54253 | 0.072 | -0.281 | 0.068 |
| 54254 | 0.048 | -0.362 | 0.020 |
| 54255 | 0.023 | -0.446 | -0.030 |
| 54311 | 0.320 | 0.169 | 0.360 |
| 54312 | 0.270 | 0.113 | 0.325 |
| 54313 | 0.257 | 0.098 | 0.316 |
| 54314 | 0.233 | 0.017 | 0.256 |
| 54315 | 0.208 | -0.067 | 0.193 |
| 54321 | 0.256 | 0.071 | 0.311 |
| 54322 | 0.206 | 0.014 | 0.263 |
| 54323 | 0.193 | 0.000 | 0.251 |
| 54324 | 0.169 | -0.081 | 0.198 |
| 54325 | 0.144 | -0.165 | 0.144 |
| 54331 | 0.240 | 0.046 | 0.299 |
| 54332 | 0.190 | -0.010 | 0.248 |
| 54333 | 0.177 | -0.025 | 0.234 |
| 54334 | 0.153 | -0.106 | 0.184 |
| 54335 | 0.128 | -0.190 | 0.132 |
| 54341 | 0.195 | -0.059 | 0.222 |
| 54342 | 0.145 | -0.115 | 0.177 |
| 54343 | 0.132 | -0.130 | 0.166 |
| 54344 | 0.108 | -0.211 | 0.117 |
| 54345 | 0.083 | -0.295 | 0.067 |
| 54351 | 0.126 | -0.217 | 0.106 |
| 54352 | 0.076 | -0.273 | 0.071 |
| 54353 | 0.063 | -0.288 | 0.062 |
| 3.000 | 0.000 | 0.200 | U.UUL |

| 54354 | 0.039 | -0.369 | 0.016 |
|-------|--------|--------|--------|
| 54355 | 0.014 | -0.453 | -0.032 |
| 54411 | 0.291 | 0.150 | 0.332 |
| 54412 | 0.241 | 0.094 | 0.303 |
| 54413 | 0.228 | 0.079 | 0.295 |
| 54414 | 0.204 | -0.002 | 0.236 |
| 54415 | 0.179 | -0.086 | 0.175 |
| 54421 | 0.227 | 0.052 | 0.289 |
| 54422 | 0.177 | -0.005 | 0.246 |
| 54423 | 0.164 | -0.019 | 0.235 |
| 54424 | 0.140 | -0.100 | 0.185 |
| 54425 | 0.115 | -0.184 | 0.132 |
| 54431 | 0.211 | 0.027 | 0.278 |
| 54432 | 0.161 | -0.029 | 0.232 |
| 54433 | 0.148 | -0.044 | 0.220 |
| 54434 | 0.124 | -0.125 | 0.172 |
| 54435 | 0.099 | -0.209 | 0.121 |
| 54441 | 0.166 | -0.078 | 0.202 |
| 54442 | 0.116 | -0.134 | 0.163 |
| 54443 | 0.103 | -0.149 | 0.153 |
| 54444 | 0.079 | -0.230 | 0.106 |
| 54445 | 0.054 | -0.314 | 0.057 |
| 54451 | 0.097 | -0.236 | 0.088 |
| 54452 | 0.047 | -0.292 | 0.059 |
| 54453 | 0.034 | -0.307 | 0.051 |
| 54454 | 0.010 | -0.388 | 0.006 |
| 54455 | -0.015 | -0.472 | -0.040 |
| 54511 | 0.231 | 0.111 | 0.276 |
| 54512 | 0.181 | 0.055 | 0.257 |
| 54513 | 0.168 | 0.040 | 0.252 |
| 54514 | 0.144 | -0.041 | 0.197 |
| 54515 | 0.119 | -0.125 | 0.140 |
| 54521 | 0.167 | 0.013 | 0.243 |
| 54522 | 0.117 | -0.044 | 0.212 |
| 54523 | 0.104 | -0.058 | 0.204 |
| 54524 | 0.080 | -0.139 | 0.156 |
| 54525 | 0.055 | -0.223 | 0.106 |
| 54531 | 0.151 | -0.012 | 0.235 |
| 54532 | 0.101 | -0.068 | 0.201 |
| 54533 | 0.088 | -0.083 | 0.192 |
| 54534 | 0.064 | -0.164 | 0.146 |
| 54535 | 0.039 | -0.248 | 0.098 |
| 54541 | 0.106 | -0.117 | 0.162 |
| 54542 | 0.056 | -0.173 | 0.134 |
| 54543 | 0.043 | -0.188 | 0.126 |
| 54544 | 0.019 | -0.269 | 0.082 |
| 54545 | -0.006 | -0.353 | 0.037 |
| 54551 | 0.037 | -0.275 | 0.053 |
| 54552 | -0.013 | -0.331 | 0.033 |

| 54553 | -0.026 | -0.346 | 0.027 |
|-------|--------|--------|--------|
| 54554 | -0.050 | -0.427 | -0.013 |
| 54555 | -0.075 | -0.511 | -0.055 |
| 55111 | 0.328 | 0.122 | 0.247 |
| 55112 | 0.278 | 0.066 | 0.234 |
| 55113 | 0.265 | 0.051 | 0.230 |
| 55114 | 0.241 | -0.030 | 0.167 |
| 55115 | 0.216 | -0.114 | 0.102 |
| 55121 | 0.264 | 0.024 | 0.221 |
| 55122 | 0.214 | -0.033 | 0.200 |
| 55123 | 0.201 | -0.048 | 0.195 |
| 55124 | 0.177 | -0.129 | 0.136 |
| 55125 | 0.152 | -0.213 | 0.076 |
| 55131 | 0.248 | -0.001 | 0.214 |
| 55132 | 0.198 | -0.057 | 0.192 |
| 55133 | 0.185 | -0.072 | 0.186 |
| 55134 | 0.161 | -0.153 | 0.129 |
| 55135 | 0.136 | -0.237 | 0.069 |
| 55141 | 0.203 | -0.106 | 0.135 |
| 55142 | 0.153 | -0.162 | 0.116 |
| 55143 | 0.140 | -0.177 | 0.111 |
| 55144 | 0.115 | -0.258 | 0.057 |
| 55145 | 0.091 | -0.342 | 0.002 |
| 55151 | 0.134 | -0.264 | 0.016 |
| 55152 | 0.084 | -0.320 | 0.003 |
| 55153 | 0.071 | -0.335 | -0.001 |
| 55154 | 0.047 | -0.416 | -0.050 |
| 55155 | 0.022 | -0.500 | -0.100 |
| 55211 | 0.293 | 0.093 | 0.247 |
| 55212 | 0.243 | 0.037 | 0.227 |
| 55213 | 0.230 | 0.022 | 0.222 |
| 55214 | 0.206 | -0.059 | 0.163 |
| 55215 | 0.181 | -0.143 | 0.102 |
| 55221 | 0.229 | -0.005 | 0.214 |
| 55222 | 0.179 | -0.062 | 0.181 |
| 55223 | 0.166 | -0.076 | 0.173 |
| 55224 | 0.142 | -0.157 | 0.122 |
| 55225 | 0.117 | -0.241 | 0.069 |
| 55231 | 0.213 | -0.030 | 0.205 |
| 55232 | 0.163 | -0.086 | 0.170 |
| 55233 | 0.150 | -0.101 | 0.160 |
| 55234 | 0.126 | -0.182 | 0.111 |
| 55235 | 0.101 | -0.266 | 0.060 |
| 55241 | 0.167 | -0.135 | 0.129 |
| 55242 | 0.117 | -0.191 | 0.100 |
| 55243 | 0.104 | -0.206 | 0.092 |
| 55244 | 0.080 | -0.287 | 0.045 |
| 55245 | 0.055 | -0.371 | -0.004 |
| 55251 | 0.099 | -0.293 | 0.015 |

| 55252 | 0.049 | -0.349 | -0.005 |
|-------|--------|----------------|--------|
| 55253 | 0.036 | -0.364 | -0.010 |
| 55254 | 0.012 | -0.445 | -0.054 |
| 55255 | -0.013 | -0.529 | -0.100 |
| 55311 | 0.284 | 0.086 | 0.247 |
| 55312 | 0.234 | 0.030 | 0.226 |
| 55313 | 0.221 | 0.015 | 0.220 |
| 55314 | 0.197 | -0.066 | 0.162 |
| 55315 | 0.172 | <b>-0</b> .150 | 0.102 |
| 55321 | 0.220 | -0.013 | 0.212 |
| 55322 | 0.170 | -0.069 | 0.176 |
| 55323 | 0.157 | -0.084 | 0.167 |
| 55324 | 0.133 | -0.165 | 0.118 |
| 55325 | 0.108 | -0.249 | 0.067 |
| 55331 | 0.204 | -0.037 | 0.203 |
| 55332 | 0.154 | -0.093 | 0.164 |
| 55333 | 0.141 | -0.108 | 0.154 |
| 55334 | 0.117 | -0.189 | 0.107 |
| 55335 | 0.092 | -0.273 | 0.058 |
| 55341 | 0.159 | -0.142 | 0.128 |
| 55342 | 0.109 | -0.198 | 0.096 |
| 55343 | 0.096 | -0.213 | 0.088 |
| 55344 | 0.071 | -0.294 | 0.042 |
| 55345 | 0.047 | -0.378 | -0.005 |
| 55351 | 0.090 | -0.300 | 0.015 |
| 55352 | 0.040 | -0.356 | -0.006 |
| 55353 | 0.027 | -0.371 | -0.012 |
| 55354 | 0.003 | <b>-0</b> .452 | -0.055 |
| 55355 | -0.022 | -0.536 | -0.100 |
| 55411 | 0.255 | 0.067 | 0.224 |
| 55412 | 0.205 | 0.011 | 0.206 |
| 55413 | 0.192 | -0.004 | 0.201 |
| 55414 | 0.168 | -0.085 | 0.146 |
| 55415 | 0.143 | -0.169 | 0.089 |
| 55421 | 0.191 | -0.032 | 0.192 |
| 55422 | 0.141 | -0.088 | 0.162 |
| 55423 | 0.128 | -0.103 | 0.154 |
| 55424 | 0.104 | -0.184 | 0.106 |
| 55425 | 0.079 | -0.268 | 0.057 |
| 55431 | 0.175 | -0.056 | 0.184 |
| 55432 | 0.125 | -0.112 | 0.151 |
| 55433 | 0.112 | -0.127 | 0.142 |
| 55434 | 0.088 | -0.208 | 0.096 |
| 55435 | 0.063 | -0.292 | 0.049 |
| 55441 | 0.129 | -0.161 | 0.111 |
| 55442 | 0.079 | -0.217 | 0.084 |
| 55443 | 0.066 | -0.232 | 0.077 |
| 55444 | 0.042 | -0.313 | 0.033 |
| 55445 | 0.017 | -0.397 | -0.012 |

| 55451 | 0.061 | -0.319 | 0.002 |
|-------|--------|----------------|--------|
| 55452 | 0.011 | -0.375 | -0.016 |
| 55453 | -0.002 | -0.390 | -0.021 |
| 55454 | -0.026 | -0.471 | -0.061 |
| 55455 | -0.051 | -0.555 | -0.103 |
| 55511 | 0.195 | 0.028 | 0.178 |
| 55512 | 0.145 | -0.028 | 0.165 |
| 55513 | 0.132 | -0.043 | 0.162 |
| 55514 | 0.108 | -0.124 | 0.113 |
| 55515 | 0.083 | -0.208 | 0.063 |
| 55521 | 0.131 | -0.071 | 0.152 |
| 55522 | 0.081 | -0.127 | 0.132 |
| 55523 | 0.068 | -0.142 | 0.127 |
| 55524 | 0.044 | -0.223 | 0.083 |
| 55525 | 0.019 | -0.307 | 0.037 |
| 55531 | 0.115 | -0.095 | 0.145 |
| 55532 | 0.065 | -0.151 | 0.124 |
| 55533 | 0.052 | <b>-0</b> .166 | 0.118 |
| 55534 | 0.028 | -0.247 | 0.075 |
| 55535 | 0.003 | -0.331 | 0.030 |
| 55541 | 0.070 | -0.200 | 0.078 |
| 55542 | 0.020 | -0.256 | 0.060 |
| 55543 | 0.007 | -0.271 | 0.055 |
| 55544 | -0.018 | -0.352 | 0.015 |
| 55545 | -0.043 | -0.436 | -0.026 |
| 55551 | 0.001 | -0.358 | -0.024 |
| 55552 | -0.049 | -0.414 | -0.037 |
| 55553 | -0.062 | -0.429 | -0.040 |
| 55554 | -0.086 | -0.510 | -0.074 |
| 55555 | -0.111 | -0.594 | -0.109 |

## 11.6 Appendix 6: Lab Reference Ranges

For some lab parameters, operational site ( PPD ) confirmed that lab ranges are missing. Hence corresponding text book ranges will be used in database. Details of those ranges are as follows:

| FormName | AnalyteName | LabLow | LabHigh | LabUnits | Reference |
|---|---|---|---|---|---|
| Urinalysis | Urine<br>Specific<br>Gravity | 1.005 | 1.030 | | Laboratory and<br>Diagnostic Tests, 8 th<br>ED. Frances Talaska<br>Fishbach, Marshall<br>Barnett Dunning,<br>Lippincott Williams &<br>Wilkins - Wolter<br>Kluwer, Inc. Page 201 |
| Urinalysis | Urine pH | 4.6 | 8.0 | | Laboratory and Diagnostic Tests, 8 th ED. Frances Talaska Fishbach, Marshall Barnett Dunning, Lippincott Williams & Wilkins - Wolter Kluwer, Inc. Page 202 |
| Coagulation - Liver Abnormality Assessment | Prothrombin<br>Time Intl.<br>Normalized<br>Ratio | 0.93 | 1.13 | | Hematology clinical<br>principles and<br>applications. 3rd ED.<br>Bernadette F Rodak;<br>George A Fritsma;<br>Kathryn Doig. St.<br>Louis,<br>Mo Saunders Elsevier<br>2007 |

## Document Approval Signature(s)

This document has been signed electronically in compliance with IQVIA and IQVIA Companies' electronic signature policies and procedures. This page is a manifestation of the electronic signatures, which may be confirmed within the IQVIA and IQVIA Companies' source system in accordance with IQVIA and IQVIA Companies' records retention policies.

Note: the Title field in the signature block has been intentionally left blank.

UserName: PPD

Title:

Date: Tuesday, 28 January 2020, 01:56 AM Eastern Time

Meaning: I Approve the Document

UserName: PPD

Title:

Date: Tuesday, 28 January 2020, 02:00 AM Eastern Time

Meaning: I Approve the Document

\_\_\_\_\_